CLINICAL TRIAL: NCT01272999
Title: POSTMARKETING OBSERVATIONAL STUDY OF THE IMPACT OF PREVNAR 13 (PNEUMOCOCCAL 13-VALENT CONJUGATE VACCINE) ON OTITIS MEDIA IN CHILDREN
Brief Title: Impact of Prevnar 13 on Ear Infections in Children
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 6096A1-4024; B1851040 (Other: Alias Study Number); 2014-001174-34 (EudraCT Number)
Record Dates: First submitted 2010-12-08; First posted 2011-01-10 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2020-10

CONDITIONS: Acute Otitis Media; Mastoiditis
Keywords: Acute otitis media; Prevnar 13; Streptococcus pneumoniae
MeSH Terms: conditions — Otitis Media; Mastoiditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Microbiology samples (middle ear fluid) taken by treating physicians in standard course of care for ear infections.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Otitis media cases
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Non interventional

SUMMARY:
Prevnar (7 valent pneumococcal conjugate vaccine [7vPnC]) has been shown to be effective against ear infections in children. Prevnar 13 is a new vaccine that is similar to Prevnar. It is expected that the effectiveness of Prevnar 13 against ear infections in children will be similar to that observed following Prevnar. Pfizer has committed to conduct a postmarketing study of the impact of Prevnar 13 in reducing ear infections among children.

ELIGIBILITY:
Inclusion Criteria:

* Case eligibility should be based on microbiologic data and should be reviewed and documented by an appropriately qualified member of the investigator's study team before cases are included in the study database.
* S pneumoniae identified from middle ear fluid or mastoiditis sample.
* Specimen obtained from children aged up to 18 years.

Exclusion Criteria:

* As this is an observational, laboratory based database study, there are no exclusion criteria

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children aged 6 weeks to 18 years
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2010-05-21 (Actual); Primary Completion 2013-12-19 (Actual); Study Completion 2013-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles - University of Southern California School of Medicine, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Children's Memorial Hospital- Feinberg School Medicine, Northwestern University, Chicago, Illinois
  - Brenner Children's Hospital - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Nationwide Children's Hospital - Ohio State University of Medicine and Public Health, Columbus, Ohio
  - Children's Hospital of Pittsburgh - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-4024&StudyName=Impact%20of%20Prevnar%2013%20on%20Ear%20Infections%20in%20Children

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a 3-year prospective laboratory-based surveillance study wherein the results of the samples obtained were summarized separately for each year. In this study, no more than 1 sample was obtained from a participant and no more than 1 serotype was isolated from any sample.
Groups:
- MEF Population: Participants with Streptococcus pneumoniae (S pneumoniae) isolates from middle ear fluid (MEF) sample without regard to whether or not they received routinely recommended vaccination of 13-valent pneumococcal conjugate vaccine (13vPnC, Prevnar 13) according to the Advisory Committee on Immunization Practices (ACIP)-recommended schedule during a surveillance period starting from December 20, 2010 through December 31, 2013.
- Mastoid Population: Participants with S pneumoniae isolates from mastoid sample without regard to whether or not they received routinely recommended vaccination of 13-valent pneumococcal conjugate vaccine (13vPnC, Prevnar 13) according to the Advisory Committee on Immunization Practices (ACIP)-recommended schedule during a surveillance period starting from December 20, 2010 through December 31, 2013.
Period: Overall Study
Arm/Group | MEF Population | Mastoid Population
Started | 357 | 34
Completed | 357 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants from whom microbiologic specimen of S pneumoniae isolates from MEF or mastoiditis sample were obtained during surveillance period.
Groups:
- Total: Total of all reporting groups
Arm/Group | MEF Population | Mastoid Population | Total
Number analyzed (Participants) | 357 | 34 | 391
Age, Continuous [Mean (Standard Deviation); unit: months] | 28.7 (26.0) | 35.5 (47.2) | 29.3 (28.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 144 | 18 | 162
  Male | 209 | 16 | 225
  Not collected | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Streptococcus Pneumoniae Serotype Isolates From Middle Ear Fluid (MEF) Sample at Surveillance Year 1
Description: The distribution of S pneumoniae serotypes isolated from MEF samples from children in the target population for vaccination over the surveillance year 1 were presented. The percentage of isolates of S pneumoniae serotypes included in Prevnar 13 (3, 7F, 19A, 19F) and not included in Prevnar 13 (6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38) along with total (both included and not included), clumps and missing or non-viable were computed along with exact 2-sided 95 percent (%) confidence interval (CI) based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this outcome measure (OM).
Time Frame: Surveillance Year 1
Population: MEF population included all participants who have at least 1 S pneumoniae isolate from MEF samples. N (number of participants analyzed) includes total number of participants in MEF population, however actual 'N' for this OM is unknown as this data were not calculated as per planned analysis.
Measure: Number (95% Confidence Interval); unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 135
percentage of isolates
  Serotype included in Prevnar 13:3 | 5.9 [2.6 to 11.3]
  Serotype included in Prevnar 13:7F | 0.7 [0.0 to 4.1]
  Serotype included in Prevnar 13:19A | 31.9 [24.1 to 40.4]
  Serotype included in Prevnar 13:19F | 2.2 [0.5 to 6.4]
  Total Serotype included in Prevnar 13 | 40.7 [32.4 to 49.5]
  Serotype not included in Prevnar 13:6C | 6.7 [3.1 to 12.3]
  Serotype not included in Prevnar 13:7C | 1.5 [0.2 to 5.2]
  Serotype not included in Prevnar 13:9N | 2.2 [0.5 to 6.4]
  Serotype not included in Prevnar 13:10 | 3.7 [1.2 to 8.4]
  Serotype not included in Prevnar 13:11 | 3.7 [1.2 to 8.4]
  Serotype not included in Prevnar 13:12 | 0.7 [0.0 to 4.1]
  Serotype not included in Prevnar 13:12F | 0.0 [0.0 to 2.7]
  Serotype not included in Prevnar 13:13 | 0.7 [0.0 to 4.1]
  Serotype not included in Prevnar 13:15A | 3.7 [1.2 to 8.4]
  Serotype not included in Prevnar 13:15B | 4.4 [1.6 to 9.4]
  Serotype not included in Prevnar 13:15C | 3.7 [1.2 to 8.4]
  Serotype not included in Prevnar 13:15F | 0.0 [0.0 to 2.7]
  Serotype not included in Prevnar 13:16 | 1.5 [0.2 to 5.2]
  Serotype not included in Prevnar 13:17 | 0.0 [0.0 to 2.7]
  Serotype not included in Prevnar 13:20 | 0.0 [0.0 to 2.7]
  Serotype not included in Prevnar 13:21 | 3.0 [0.8 to 7.4]
  Serotype not included in Prevnar 13:22F | 1.5 [0.2 to 5.2]
  Serotype not included in Prevnar 13:23A | 3.7 [1.2 to 8.4]
  Serotype not included in Prevnar 13:23B | 2.2 [0.5 to 6.4]
  Serotype not included in Prevnar 13:31 | 2.2 [0.5 to 6.4]
  Serotype not included in Prevnar 13:33A | 0.7 [0.0 to 4.1]
  Serotype not included in Prevnar 13:33F | 3.0 [0.8 to 7.4]
  Serotype not included in Prevnar 13:34 | 0.0 [0.0 to 2.7]
  Serotype not included in Prevnar 13:35B | 6.7 [3.1 to 12.3]
  Serotype not included in Prevnar 13:35F | 0.0 [0.0 to 2.7]
  Serotype not included in Prevnar 13:38 | 0.7 [0.0 to 4.1]
  Total Serotype not included in Prevnar 13 | 56.3 [47.5 to 64.8]
  Serotype clumps | 1.5 [0.2 to 5.2]
  Serotype Missing/non-viable | 1.5 [0.2 to 5.2]

2. Primary Outcome: Percentage of Streptococcus Pneumoniae Serotype Isolates From Middle Ear Fluid (MEF) Sample at Surveillance Year 2
Description: The distribution of S pneumoniae serotypes isolated from MEF samples from children in the target population for vaccination over the surveillance year 2 were presented. The percentage of isolates of S pneumoniae serotypes included in Prevnar 13 (3, 7F, 19A, 19F) and not included in Prevnar 13 (6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38) along with total (both included and not included), clumps and missing or non-viable were computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 111
percentage of isolates
  Serotype included in Prevnar 13:3 | 6.3 [2.6 to 12.6]
  Serotype included in Prevnar 13:7F | 0.0 [0.0 to 3.3]
  Serotype included in Prevnar 13:19A | 23.4 [15.9 to 32.4]
  Serotype included in Prevnar 13:19F | 1.8 [0.2 to 6.4]
  Total Serotype included in Prevnar 13 | 31.5 [23.0 to 41.0]
  Serotype not included in Prevnar 13:6C | 4.5 [1.5 to 10.2]
  Serotype not included in Prevnar 13:7C | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:9N | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:10 | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:11 | 7.2 [3.2 to 13.7]
  Serotype not included in Prevnar 13:12 | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:12F | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:13 | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:15A | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:15B | 4.5 [1.5 to 10.2]
  Serotype not included in Prevnar 13:15C | 2.7 [0.6 to 7.7]
  Serotype not included in Prevnar 13:15F | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:16 | 2.7 [0.6 to 7.7]
  Serotype not included in Prevnar 13:17 | 1.8 [0.2 to 6.4]
  Serotype not included in Prevnar 13:20 | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:21 | 9.0 [4.4 to 15.9]
  Serotype not included in Prevnar 13:22F | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:23A | 4.5 [1.5 to 10.2]
  Serotype not included in Prevnar 13:23B | 7.2 [3.2 to 13.7]
  Serotype not included in Prevnar 13:31 | 1.8 [0.2 to 6.4]
  Serotype not included in Prevnar 13:33A | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:33F | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:34 | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:35B | 13.5 [7.8 to 21.3]
  Serotype not included in Prevnar 13:35F | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:38 | 0.9 [0.0 to 4.9]
  Total Serotype not included in Prevnar 13 | 66.7 [57.1 to 75.3]
  Serotype clumps | 0.9 [0.0 to 4.9]
  Serotype Missing/non-viable | 0.9 [0.0 to 4.9]

3. Primary Outcome: Percentage of Streptococcus Pneumoniae Serotype Isolates From Middle Ear Fluid (MEF) Sample at Surveillance Year 3
Description: The distribution of S pneumoniae serotypes isolated from MEF samples from children in the target population for vaccination over the surveillance year 3 were presented. The percentage of isolates of S pneumoniae serotypes included in Prevnar 13 (3, 7F, 19A, 19F) and not included in Prevnar 13 (6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38) along with total (both included and not included), clumps and missing or non-viable were computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 111
percentage of isolates
  Serotype included in Prevnar 13:3 | 7.2 [3.2 to 13.7]
  Serotype included in Prevnar 13:7F | 0.0 [0.0 to 3.3]
  Serotype included in Prevnar 13:19A | 9.9 [5.1 to 17.0]
  Serotype included in Prevnar 13:19F | 6.3 [2.6 to 12.6]
  Total Serotype included in Prevnar 13 | 23.4 [15.9 to 32.4]
  Serotype not included in Prevnar 13:6C | 1.8 [0.2 to 6.4]
  Serotype not included in Prevnar 13:7C | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:9N | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:10 | 2.7 [0.6 to 7.7]
  Serotype not included in Prevnar 13:11 | 3.6 [1.0 to 9.0]
  Serotype not included in Prevnar 13:12 | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:12F | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:13 | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:15A | 6.3 [2.6 to 12.6]
  Serotype not included in Prevnar 13:15B | 5.4 [2.0 to 11.4]
  Serotype not included in Prevnar 13:15C | 5.4 [2.0 to 11.4]
  Serotype not included in Prevnar 13:15F | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:16 | 5.4 [2.0 to 11.4]
  Serotype not included in Prevnar 13:17 | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:20 | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:21 | 5.4 [2.0 to 11.4]
  Serotype not included in Prevnar 13:22F | 2.7 [0.6 to 7.7]
  Serotype not included in Prevnar 13:23A | 2.7 [0.6 to 7.7]
  Serotype not included in Prevnar 13:23B | 8.1 [3.8 to 14.8]
  Serotype not included in Prevnar 13:31 | 4.5 [1.5 to 10.2]
  Serotype not included in Prevnar 13:33A | 0.0 [0.0 to 3.3]
  Serotype not included in Prevnar 13:33F | 1.8 [0.2 to 6.4]
  Serotype not included in Prevnar 13:34 | 0.9 [0.0 to 4.9]
  Serotype not included in Prevnar 13:35B | 10.8 [5.7 to 18.1]
  Serotype not included in Prevnar 13:35F | 1.8 [0.2 to 6.4]
  Serotype not included in Prevnar 13:38 | 1.8 [0.2 to 6.4]
  Total Serotype not included in Prevnar 13 | 74.8 [65.6 to 82.5]
  Serotype clumps | 0.0 [0.0 to 3.3]
  Serotype Missing/non-viable | 1.8 [0.2 to 6.4]

4. Primary Outcome: Percentage of Streptococcus Pneumoniae Serotype Isolates From Mastoiditis Sample at Surveillance Year 1
Description: The distribution of S pneumoniae serotypes isolated from mastoiditis samples from children in the target population for vaccination over the surveillance year 1 were presented. The percentage of isolates of S pneumoniae serotypes included in Prevnar 13 (1, 3, 7F, 14, 19A, 19F) and not included in Prevnar 13 (6C, 12, 15A, 15B, 15F, 21, 22F, 23A, 33F, 35B, 38) along with total (both included and not included in Prevnar 13 ), clumps and missing or non-viable were computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1
Population: Mastoid population included all participants who have at least 1 S pneumoniae isolate from mastoid samples. N (number of participants analyzed) includes total number of participants in mastoid population, however actual 'N' for this OM is unknown as this data were not calculated as per planned analysis.
Measure: Number (95% Confidence Interval); unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
Number analyzed (Isolates) | 18
percentage of isolates
  Serotype included in Prevnar 13:1 | 0.0 [0.0 to 18.5]
  Serotype included in Prevnar 13:3 | 0.0 [0.0 to 18.5]
  Serotype included in Prevnar 13:7F | 0.0 [0.0 to 18.5]
  Serotype included in Prevnar 13:14 | 0.0 [0.0 to 18.5]
  Serotype included in Prevnar 13:19A | 38.9 [17.3 to 64.3]
  Serotype included in Prevnar 13:19F | 11.1 [1.4 to 34.7]
  Total Serotype included in Prevnar 13 | 50.0 [26.0 to 74.0]
  Serotype not included in Prevnar 13:6C | 5.6 [0.1 to 27.3]
  Serotype not included in Prevnar 13:12 | 5.6 [0.1 to 27.3]
  Serotype not included in Prevnar 13:15A | 5.6 [0.1 to 27.3]
  Serotype not included in Prevnar 13:15B | 5.6 [0.1 to 27.3]
  Serotype not included in Prevnar 13:15F | 0.0 [0.0 to 18.5]
  Serotype not included in Prevnar 13:21 | 0.0 [0.0 to 18.5]
  Serotype not included in Prevnar 13:22F | 11.1 [1.4 to 34.7]
  Serotype not included in Prevnar 13:23A | 5.6 [0.1 to 27.3]
  Serotype not included in Prevnar 13:33F | 0.0 [0.0 to 18.5]
  Serotype not included in Prevnar 13:35B | 5.6 [0.1 to 27.3]
  Serotype not included in Prevnar 13:38 | 5.6 [0.1 to 27.3]
  Total Serotype not included in Prevnar 13 | 50.0 [26.0 to 74.0]
  Serotype missing/non-viable | 0.0 [0.0 to 18.5]

5. Primary Outcome: Percentage of Streptococcus Pneumoniae Serotype Isolates From Mastoiditis Sample at Surveillance Year 2
Description: The distribution of S pneumoniae serotypes isolated from mastoiditis samples from children in the target population for vaccination over the surveillance year 2 were presented. The percentage of isolates of S pneumoniae serotypes included in Prevnar 13 (1, 3, 7F, 14, 19A, 19F) and not included in Prevnar 13 (6C, 12, 15A, 15B, 15F, 21, 22F, 23A, 33F, 35B, 38) along with total (both included and not included in Prevnar 13 ), clumps and missing or non-viable were computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 2
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
Number analyzed (Isolates) | 7
percentage of isolates
  Serotype included in Prevnar 13:1 | 0.0 [0.0 to 41.0]
  Serotype included in Prevnar 13:3 | 28.6 [3.7 to 71.0]
  Serotype included in Prevnar 13:7F | 0.0 [0.0 to 41.0]
  Serotype included in Prevnar 13:14 | 0.0 [0.0 to 41.0]
  Serotype included in Prevnar 13:19A | 71.4 [29.0 to 96.3]
  Serotype included in Prevnar 13:19F | 0.0 [0.0 to 41.0]
  Total Serotype included in Prevnar 13 | 100.0 [59.0 to 100.0]
  Serotype not included in Prevnar 13:6C | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:12 | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:15A | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:15B | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:15F | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:21 | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:22F | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:23A | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:33F | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:35B | 0.0 [0.0 to 41.0]
  Serotype not included in Prevnar 13:38 | 0.0 [0.0 to 41.0]
  Total Serotype not included in Prevnar 13 | 0.0 [0.0 to 41.0]
  Serotype missing/non-viable | 0.0 [0.0 to 41.0]

6. Primary Outcome: Percentage of Streptococcus Pneumoniae Serotype Isolates From Mastoiditis Sample at Surveillance Year 3
Description: The distribution of S pneumoniae serotypes isolated from mastoiditis samples from children in the target population for vaccination over the surveillance year 3 were presented. The percentage of isolates of S pneumoniae serotypes included in Prevnar 13 (1, 3, 7F, 14, 19A, 19F) and not included in Prevnar 13 (6C, 12, 15A, 15B, 15F, 21, 22F, 23A, 33F, 35B, 38) along with total (both included and not included in Prevnar 13 ), clumps and missing or non-viable were computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
Number analyzed (Isolates) | 9
percentage of isolates
  Serotype included in Prevnar 13:1 | 0.0 [0.0 to 33.6]
  Serotype included in Prevnar 13:3 | 44.4 [13.7 to 78.8]
  Serotype included in Prevnar 13:7F | 0.0 [0.0 to 33.6]
  Serotype included in Prevnar 13:14 | 0.0 [0.0 to 33.6]
  Serotype included in Prevnar 13:19A | 11.1 [0.3 to 48.2]
  Serotype included in Prevnar 13:19F | 11.1 [0.3 to 48.2]
  Total Serotype included in Prevnar 13 | 66.7 [29.9 to 92.5]
  Serotype not included in Prevnar 13:6C | 0.0 [0.0 to 33.6]
  Serotype not included in Prevnar 13:12 | 0.0 [0.0 to 33.6]
  Serotype not included in Prevnar 13:15A | 0.0 [0.0 to 33.6]
  Serotype not included in Prevnar 13:15B | 0.0 [0.0 to 33.6]
  Serotype not included in Prevnar 13:15F | 0.0 [0.0 to 33.6]
  Serotype not included in Prevnar 13:21 | 0.0 [0.0 to 33.6]
  Serotype not included in Prevnar 13:22F | 11.1 [0.3 to 48.2]
  Serotype not included in Prevnar 13:23A | 0.0 [0.0 to 33.6]
  Serotype not included in Prevnar 13:33F | 22.2 [2.8 to 60.0]
  Serotype not included in Prevnar 13:35B | 0.0 [0.0 to 33.6]
  Serotype not included in Prevnar 13:38 | 0.0 [0.0 to 33.6]
  Total Serotype not included in Prevnar 13 | 33.3 [7.5 to 70.1]
  Serotype missing/non-viable | 0.0 [0.0 to 33.6]

7. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Amoxicillin: Middle Ear Fluid (MEF) Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for amoxicillin from MEF samples was categorized as resistant, susceptible or intermediate based on minimum inhibitory concentration (MIC) for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 19 A, 19 F, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38, clumps and missing or non-viable, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: MEF population. N (number of participants analyzed) includes total number of participants in MEF population, however actual 'N' for this OM is unknown as this data were not calculated as per planned analysis and number analyzed = number of isolates for the given serotype at specified time point.
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 135
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 135
  Serotype 3 at Year 1:S | 3.0
  Serotype 6C at Year 1:S: number analyzed (Participants) | 135
  Serotype 6C at Year 1:S | 3.0
  Serotype 7C at Year 1:S: number analyzed (Participants) | 135
  Serotype 7C at Year 1:S | 0.0
  Serotype 9N at Year 1:S: number analyzed (Participants) | 135
  Serotype 9N at Year 1:S | 0.7
  Serotype 10 at Year 1:S: number analyzed (Participants) | 135
  Serotype 10 at Year 1:S | 1.5
  Serotype 11 at Year 1:S: number analyzed (Participants) | 135
  Serotype 11 at Year 1:S | 1.5
  Serotype 12 at Year 1:S: number analyzed (Participants) | 135
  Serotype 12 at Year 1:S | 0.0
  Serotype 12F at Year 1:S: number analyzed (Participants) | 135
  Serotype 12F at Year 1:S | 0.0
  Serotype 13 at Year 1:S: number analyzed (Participants) | 135
  Serotype 13 at Year 1:S | 0.0
  Serotype 15A at Year 1:S: number analyzed (Participants) | 135
  Serotype 15A at Year 1:S | 1.5
  Serotype 15B at Year 1:S: number analyzed (Participants) | 135
  Serotype 15B at Year 1:S | 0.7
  Serotype 15C at Year 1:S: number analyzed (Participants) | 135
  Serotype 15C at Year 1:S | 3.0
  Serotype 15F at Year 1:S: number analyzed (Participants) | 135
  Serotype 15F at Year 1:S | 0.0
  Serotype 16 at Year 1:S: number analyzed (Participants) | 135
  Serotype 16 at Year 1:S | 0.0
  Serotype 17 at Year 1:S: number analyzed (Participants) | 135
  Serotype 17 at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 135
  Serotype 19A at Year 1:S | 3.0
  Serotype 19F at Year 1:S: number analyzed (Participants) | 135
  Serotype 19F at Year 1:S | 0.7
  Serotype 20 at Year 1:S: number analyzed (Participants) | 135
  Serotype 20 at Year 1:S | 0.0
  Serotype 21 at Year 1:S: number analyzed (Participants) | 135
  Serotype 21 at Year 1:S | 1.5
  Serotype 22F at Year 1:S: number analyzed (Participants) | 135
  Serotype 22F at Year 1:S | 0.0
  Serotype 23A at Year 1:S: number analyzed (Participants) | 135
  Serotype 23A at Year 1:S | 1.5
  Serotype 23B at Year 1:S: number analyzed (Participants) | 135
  Serotype 23B at Year 1:S | 0.7
  Serotype 31 at Year 1:S: number analyzed (Participants) | 135
  Serotype 31 at Year 1:S | 0.0
  Serotype 33A at Year 1:S: number analyzed (Participants) | 135
  Serotype 33A at Year 1:S | 0.7
  Serotype 33F at Year 1:S: number analyzed (Participants) | 135
  Serotype 33F at Year 1:S | 0.0
  Serotype 34 at Year 1:S: number analyzed (Participants) | 135
  Serotype 34 at Year 1:S | 0.0
  Serotype 35B at Year 1:S: number analyzed (Participants) | 135
  Serotype 35B at Year 1:S | 3.0
  Serotype 35F at Year 1:S: number analyzed (Participants) | 135
  Serotype 35F at Year 1:S | 0.0
  Serotype 38 at Year 1:S: number analyzed (Participants) | 135
  Serotype 38 at Year 1:S | 0.0
  Serotype clumps at Year 1:S: number analyzed (Participants) | 135
  Serotype clumps at Year 1:S | 0.0
  Serotype Missing/non-viable at Year 1:S: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:S | 0.0
  Serotype 3 at Year 2:S: number analyzed (Participants) | 111
  Serotype 3 at Year 2:S | 1.8
  Serotype 6C at Year 2:S: number analyzed (Participants) | 111
  Serotype 6C at Year 2:S | 0.9
  Serotype 7C at Year 2:S: number analyzed (Participants) | 111
  Serotype 7C at Year 2:S | 0.0
  Serotype 9N at Year 2:S: number analyzed (Participants) | 111
  Serotype 9N at Year 2:S | 0.0
  Serotype 10 at Year 2:S: number analyzed (Participants) | 111
  Serotype 10 at Year 2:S | 0.9
  Serotype 11 at Year 2:S: number analyzed (Participants) | 111
  Serotype 11 at Year 2:S | 2.7
  Serotype 12 at Year 2:S: number analyzed (Participants) | 111
  Serotype 12 at Year 2:S | 0.0
  Serotype 12F at Year 2:S: number analyzed (Participants) | 111
  Serotype 12F at Year 2:S | 0.9
  Serotype 13 at Year 2:S: number analyzed (Participants) | 111
  Serotype 13 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 111
  Serotype 15A at Year 2:S | 0.9
  Serotype 15B at Year 2:S: number analyzed (Participants) | 111
  Serotype 15B at Year 2:S | 0.0
  Serotype 15C at Year 2:S: number analyzed (Participants) | 111
  Serotype 15C at Year 2:S | 2.7
  Serotype 15F at Year 2:S: number analyzed (Participants) | 111
  Serotype 15F at Year 2:S | 0.0
  Serotype 16 at Year 2:S: number analyzed (Participants) | 111
  Serotype 16 at Year 2:S | 0.9
  Serotype 17 at Year 2:S: number analyzed (Participants) | 111
  Serotype 17 at Year 2:S | 1.8
  Serotype 19A at Year 2:S: number analyzed (Participants) | 111
  Serotype 19A at Year 2:S | 1.8
  Serotype 19F at Year 2:S: number analyzed (Participants) | 111
  Serotype 19F at Year 2:S | 0.9
  Serotype 20 at Year 2:S: number analyzed (Participants) | 111
  Serotype 20 at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 111
  Serotype 21 at Year 2:S | 2.7
  Serotype 22F at Year 2:S: number analyzed (Participants) | 111
  Serotype 22F at Year 2:S | 0.0
  Serotype 23A at Year 2:S: number analyzed (Participants) | 111
  Serotype 23A at Year 2:S | 2.7
  Serotype 23B at Year 2:S: number analyzed (Participants) | 111
  Serotype 23B at Year 2:S | 2.7
  Serotype 31 at Year 2:S: number analyzed (Participants) | 111
  Serotype 31 at Year 2:S | 1.8
  Serotype 33A at Year 2:S: number analyzed (Participants) | 111
  Serotype 33A at Year 2:S | 0.0
  Serotype 33F at Year 2:S: number analyzed (Participants) | 111
  Serotype 33F at Year 2:S | 0.0
  Serotype 34 at Year 2:S: number analyzed (Participants) | 111
  Serotype 34 at Year 2:S | 0.9
  Serotype 35B at Year 2:S: number analyzed (Participants) | 111
  Serotype 35B at Year 2:S | 4.5
  Serotype 35F at Year 2:S: number analyzed (Participants) | 111
  Serotype 35F at Year 2:S | 0.9
  Serotype 38 at Year 2:S: number analyzed (Participants) | 111
  Serotype 38 at Year 2:S | 0.9
  Serotype clumps at Year 2:S: number analyzed (Participants) | 111
  Serotype clumps at Year 2:S | 0.0
  Serotype Missing/non-viable at Year 2:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:S | 0.9
  Serotype 3 at Year 3:S: number analyzed (Participants) | 111
  Serotype 3 at Year 3:S | 3.6
  Serotype 6C at Year 3:S: number analyzed (Participants) | 111
  Serotype 6C at Year 3:S | 0.0
  Serotype 7C at Year 3:S: number analyzed (Participants) | 111
  Serotype 7C at Year 3:S | 0.0
  Serotype 9N at Year 3:S: number analyzed (Participants) | 111
  Serotype 9N at Year 3:S | 0.9
  Serotype 10 at Year 3:S: number analyzed (Participants) | 111
  Serotype 10 at Year 3:S | 1.8
  Serotype 11 at Year 3:S: number analyzed (Participants) | 111
  Serotype 11 at Year 3:S | 1.8
  Serotype 12 at Year 3:S: number analyzed (Participants) | 111
  Serotype 12 at Year 3:S | 0.0
  Serotype 12F at Year 3:S: number analyzed (Participants) | 111
  Serotype 12F at Year 3:S | 0.0
  Serotype 13 at Year 3:S: number analyzed (Participants) | 111
  Serotype 13 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 111
  Serotype 15A at Year 3:S | 2.7
  Serotype 15B at Year 3:S: number analyzed (Participants) | 111
  Serotype 15B at Year 3:S | 3.6
  Serotype 15C at Year 3:S: number analyzed (Participants) | 111
  Serotype 15C at Year 3:S | 0.9
  Serotype 15F at Year 3:S: number analyzed (Participants) | 111
  Serotype 15F at Year 3:S | 0.0
  Serotype 16 at Year 3:S: number analyzed (Participants) | 111
  Serotype 16 at Year 3:S | 3.6
  Serotype 17 at Year 3:S: number analyzed (Participants) | 111
  Serotype 17 at Year 3:S | 0.9
  Serotype 19A at Year 3:S: number analyzed (Participants) | 111
  Serotype 19A at Year 3:S | 0.0
  Serotype 19F at Year 3:S: number analyzed (Participants) | 111
  Serotype 19F at Year 3:S | 1.8
  Serotype 20 at Year 3:S: number analyzed (Participants) | 111
  Serotype 20 at Year 3:S | 0.9
  Serotype 21 at Year 3:S: number analyzed (Participants) | 111
  Serotype 21 at Year 3:S | 1.8
  Serotype 22F at Year 3:S: number analyzed (Participants) | 111
  Serotype 22F at Year 3:S | 0.0
  Serotype 23A at Year 3:S: number analyzed (Participants) | 111
  Serotype 23A at Year 3:S | 2.7
  Serotype 23B at Year 3:S: number analyzed (Participants) | 111
  Serotype 23B at Year 3:S | 6.3
  Serotype 31 at Year 3:S: number analyzed (Participants) | 111
  Serotype 31 at Year 3:S | 1.8
  Serotype 33A at Year 3:S: number analyzed (Participants) | 111
  Serotype 33A at Year 3:S | 0.0
  Serotype 33F at Year 3:S: number analyzed (Participants) | 111
  Serotype 33F at Year 3:S | 0.0
  Serotype 34 at Year 3:S: number analyzed (Participants) | 111
  Serotype 34 at Year 3:S | 0.0
  Serotype 35B at Year 3:S: number analyzed (Participants) | 111
  Serotype 35B at Year 3:S | 5.4
  Serotype 35F at Year 3:S: number analyzed (Participants) | 111
  Serotype 35F at Year 3:S | 0.0
  Serotype 38 at Year 3:S: number analyzed (Participants) | 111
  Serotype 38 at Year 3:S | 0.9
  Serotype clumps at Year 3:S: number analyzed (Participants) | 111
  Serotype clumps at Year 3:S | 0.0
  Serotype Missing/non-viable at Year 3:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:S | 0.0
  Serotype 3 at Year 1:I: number analyzed (Participants) | 135
  Serotype 3 at Year 1:I | 0.0
  Serotype 6C at Year 1:I: number analyzed (Participants) | 135
  Serotype 6C at Year 1:I | 0.0
  Serotype 7C at Year 1:I: number analyzed (Participants) | 135
  Serotype 7C at Year 1:I | 0.0
  Serotype 9N at Year 1:I: number analyzed (Participants) | 135
  Serotype 9N at Year 1:I | 0.0
  Serotype 10 at Year 1:I: number analyzed (Participants) | 135
  Serotype 10 at Year 1:I | 0.0
  Serotype 11 at Year 1:I: number analyzed (Participants) | 135
  Serotype 11 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 135
  Serotype 12 at Year 1:I | 0.0
  Serotype 12F at Year 1:I: number analyzed (Participants) | 135
  Serotype 12F at Year 1:I | 0.0
  Serotype 13 at Year 1:I: number analyzed (Participants) | 135
  Serotype 13 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 135
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 135
  Serotype 15B at Year 1:I | 0.0
  Serotype 15C at Year 1:I: number analyzed (Participants) | 135
  Serotype 15C at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 135
  Serotype 15F at Year 1:I | 0.0
  Serotype 16 at Year 1:I: number analyzed (Participants) | 135
  Serotype 16 at Year 1:I | 0.0
  Serotype 17 at Year 1:I: number analyzed (Participants) | 135
  Serotype 17 at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 135
  Serotype 19A at Year 1:I | 5.9
  Serotype 19F at Year 1:I: number analyzed (Participants) | 135
  Serotype 19F at Year 1:I | 0.0
  Serotype 20 at Year 1:I: number analyzed (Participants) | 135
  Serotype 20 at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 135
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 135
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 135
  Serotype 23A at Year 1:I | 0.0
  Serotype 23B at Year 1:I: number analyzed (Participants) | 135
  Serotype 23B at Year 1:I | 0.0
  Serotype 31 at Year 1:I: number analyzed (Participants) | 135
  Serotype 31 at Year 1:I | 0.0
  Serotype 33A at Year 1:I: number analyzed (Participants) | 135
  Serotype 33A at Year 1:I | 0.0
  Serotype 33F at Year 1:I: number analyzed (Participants) | 135
  Serotype 33F at Year 1:I | 0.0
  Serotype 34 at Year 1:I: number analyzed (Participants) | 135
  Serotype 34 at Year 1:I | 0.0
  Serotype 35B at Year 1:I: number analyzed (Participants) | 135
  Serotype 35B at Year 1:I | 0.0
  Serotype 35F at Year 1:I: number analyzed (Participants) | 135
  Serotype 35F at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 135
  Serotype 38 at Year 1:I | 0.0
  Serotype clumps at Year 1:I: number analyzed (Participants) | 135
  Serotype clumps at Year 1:I | 0.0
  Serotype Missing/non-viable at Year 1:I: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 111
  Serotype 3 at Year 2:I | 0.0
  Serotype 6C at Year 2:I: number analyzed (Participants) | 111
  Serotype 6C at Year 2:I | 0.0
  Serotype 7C at Year 2:I: number analyzed (Participants) | 111
  Serotype 7C at Year 2:I | 0.0
  Serotype 9N at Year 2:I: number analyzed (Participants) | 111
  Serotype 9N at Year 2:I | 0.0
  Serotype 10 at Year 2:I: number analyzed (Participants) | 111
  Serotype 10 at Year 2:I | 0.0
  Serotype 11 at Year 2:I: number analyzed (Participants) | 111
  Serotype 11 at Year 2:I | 0.0
  Serotype 12 at Year 2:I: number analyzed (Participants) | 111
  Serotype 12 at Year 2:I | 0.0
  Serotype 12F at Year 2:I: number analyzed (Participants) | 111
  Serotype 12F at Year 2:I | 0.0
  Serotype 13 at Year 2:I: number analyzed (Participants) | 111
  Serotype 13 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 111
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 111
  Serotype 15B at Year 2:I | 0.0
  Serotype 15C at Year 2:I: number analyzed (Participants) | 111
  Serotype 15C at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 111
  Serotype 15F at Year 2:I | 0.0
  Serotype 16 at Year 2:I: number analyzed (Participants) | 111
  Serotype 16 at Year 2:I | 0.0
  Serotype 17 at Year 2:I: number analyzed (Participants) | 111
  Serotype 17 at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 111
  Serotype 19A at Year 2:I | 0.0
  Serotype 19F at Year 2:I: number analyzed (Participants) | 111
  Serotype 19F at Year 2:I | 0.0
  Serotype 20 at Year 2:I: number analyzed (Participants) | 111
  Serotype 20 at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 111
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 111
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 111
  Serotype 23A at Year 2:I | 0.0
  Serotype 23B at Year 2:I: number analyzed (Participants) | 111
  Serotype 23B at Year 2:I | 0.0
  Serotype 31 at Year 2:I: number analyzed (Participants) | 111
  Serotype 31 at Year 2:I | 0.0
  Serotype 33A at Year 2:I: number analyzed (Participants) | 111
  Serotype 33A at Year 2:I | 0.0
  Serotype 33F at Year 2:I: number analyzed (Participants) | 111
  Serotype 33F at Year 2:I | 0.0
  Serotype 34 at Year 2:I: number analyzed (Participants) | 111
  Serotype 34 at Year 2:I | 0.0
  Serotype 35B at Year 2:I: number analyzed (Participants) | 111
  Serotype 35B at Year 2:I | 0.0
  Serotype 35F at Year 2:I: number analyzed (Participants) | 111
  Serotype 35F at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 111
  Serotype 38 at Year 2:I | 0.0
  Serotype clumps at Year 2:I: number analyzed (Participants) | 111
  Serotype clumps at Year 2:I | 0.0
  Serotype Missing/non-viable at Year 2:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 111
  Serotype 3 at Year 3:I | 0.0
  Serotype 6C at Year 3:I: number analyzed (Participants) | 111
  Serotype 6C at Year 3:I | 0.0
  Serotype 7C at Year 3:I: number analyzed (Participants) | 111
  Serotype 7C at Year 3:I | 0.0
  Serotype 9N at Year 3:I: number analyzed (Participants) | 111
  Serotype 9N at Year 3:I | 0.0
  Serotype 10 at Year 3:I: number analyzed (Participants) | 111
  Serotype 10 at Year 3:I | 0.0
  Serotype 11 at Year 3:I: number analyzed (Participants) | 111
  Serotype 11 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 111
  Serotype 12 at Year 3:I | 0.0
  Serotype 12F at Year 3:I: number analyzed (Participants) | 111
  Serotype 12F at Year 3:I | 0.0
  Serotype 13 at Year 3:I: number analyzed (Participants) | 111
  Serotype 13 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 111
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 111
  Serotype 15B at Year 3:I | 0.0
  Serotype 15C at Year 3:I: number analyzed (Participants) | 111
  Serotype 15C at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 111
  Serotype 15F at Year 3:I | 0.0
  Serotype 16 at Year 3:I: number analyzed (Participants) | 111
  Serotype 16 at Year 3:I | 0.0
  Serotype 17 at Year 3:I: number analyzed (Participants) | 111
  Serotype 17 at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 111
  Serotype 19A at Year 3:I | 2.7
  Serotype 19F at Year 3:I: number analyzed (Participants) | 111
  Serotype 19F at Year 3:I | 0.0
  Serotype 20 at Year 3:I: number analyzed (Participants) | 111
  Serotype 20 at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 111
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 111
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 111
  Serotype 23A at Year 3:I | 0.0
  Serotype 23B at Year 3:I: number analyzed (Participants) | 111
  Serotype 23B at Year 3:I | 0.0
  Serotype 31 at Year 3:I: number analyzed (Participants) | 111
  Serotype 31 at Year 3:I | 0.0
  Serotype 33A at Year 3:I: number analyzed (Participants) | 111
  Serotype 33A at Year 3:I | 0.0
  Serotype 33F at Year 3:I: number analyzed (Participants) | 111
  Serotype 33F at Year 3:I | 0.0
  Serotype 34 at Year 3:I: number analyzed (Participants) | 111
  Serotype 34 at Year 3:I | 0.0
  Serotype 35B at Year 3:I: number analyzed (Participants) | 111
  Serotype 35B at Year 3:I | 0.9
  Serotype 35F at Year 3:I: number analyzed (Participants) | 111
  Serotype 35F at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 111
  Serotype 38 at Year 3:I | 0.0
  Serotype clumps at Year 3:I: number analyzed (Participants) | 111
  Serotype clumps at Year 3:I | 0.0
  Serotype Missing/non-viable at Year 3:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 135
  Serotype 3 at Year 1:R | 0.0
  Serotype 6C at Year 1:R: number analyzed (Participants) | 135
  Serotype 6C at Year 1:R | 0.0
  Serotype 7C at Year 1:R: number analyzed (Participants) | 135
  Serotype 7C at Year 1:R | 0.0
  Serotype 9N at Year 1:R: number analyzed (Participants) | 135
  Serotype 9N at Year 1:R | 0.0
  Serotype 10 at Year 1:R: number analyzed (Participants) | 135
  Serotype 10 at Year 1:R | 0.0
  Serotype 11 at Year 1:R: number analyzed (Participants) | 135
  Serotype 11 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 135
  Serotype 12 at Year 1:R | 0.0
  Serotype 12F at Year 1:R: number analyzed (Participants) | 135
  Serotype 12F at Year 1:R | 0.0
  Serotype 13 at Year 1:R: number analyzed (Participants) | 135
  Serotype 13 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 135
  Serotype 15A at Year 1:R | 0.0
  Serotype 15B at Year 1:R: number analyzed (Participants) | 135
  Serotype 15B at Year 1:R | 0.0
  Serotype 15C at Year 1:R: number analyzed (Participants) | 135
  Serotype 15C at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 135
  Serotype 15F at Year 1:R | 0.0
  Serotype 16 at Year 1:R: number analyzed (Participants) | 135
  Serotype 16 at Year 1:R | 0.0
  Serotype 17 at Year 1:R: number analyzed (Participants) | 135
  Serotype 17 at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 135
  Serotype 19A at Year 1:R | 0.0
  Serotype 19F at Year 1:R: number analyzed (Participants) | 135
  Serotype 19F at Year 1:R | 0.0
  Serotype 20 at Year 1:R: number analyzed (Participants) | 135
  Serotype 20 at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 135
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 135
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 135
  Serotype 23A at Year 1:R | 0.0
  Serotype 23B at Year 1:R: number analyzed (Participants) | 135
  Serotype 23B at Year 1:R | 0.0
  Serotype 31 at Year 1:R: number analyzed (Participants) | 135
  Serotype 31 at Year 1:R | 0.0
  Serotype 33A at Year 1:R: number analyzed (Participants) | 135
  Serotype 33A at Year 1:R | 0.0
  Serotype 33F at Year 1:R: number analyzed (Participants) | 135
  Serotype 33F at Year 1:R | 0.0
  Serotype 34 at Year 1:R: number analyzed (Participants) | 135
  Serotype 34 at Year 1:R | 0.0
  Serotype 35B at Year 1:R: number analyzed (Participants) | 135
  Serotype 35B at Year 1:R | 0.0
  Serotype 35F at Year 1:R: number analyzed (Participants) | 135
  Serotype 35F at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 135
  Serotype 38 at Year 1:R | 0.0
  Serotype clumps at Year 1:R: number analyzed (Participants) | 135
  Serotype clumps at Year 1:R | 0.0
  Serotype Missing/non-viable at Year 1:R: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 111
  Serotype 3 at Year 2:R | 0.0
  Serotype 6C at Year 2:R: number analyzed (Participants) | 111
  Serotype 6C at Year 2:R | 0.0
  Serotype 7C at Year 2:R: number analyzed (Participants) | 111
  Serotype 7C at Year 2:R | 0.0
  Serotype 9N at Year 2:R: number analyzed (Participants) | 111
  Serotype 9N at Year 2:R | 0.0
  Serotype 10 at Year 2:R: number analyzed (Participants) | 111
  Serotype 10 at Year 2:R | 0.0
  Serotype 11 at Year 2:R: number analyzed (Participants) | 111
  Serotype 11 at Year 2:R | 0.0
  Serotype 12 at Year 2:R: number analyzed (Participants) | 111
  Serotype 12 at Year 2:R | 0.0
  Serotype 12F at Year 2:R: number analyzed (Participants) | 111
  Serotype 12F at Year 2:R | 0.0
  Serotype 13 at Year 2:R: number analyzed (Participants) | 111
  Serotype 13 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 111
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 111
  Serotype 15B at Year 2:R | 0.0
  Serotype 15C at Year 2:R: number analyzed (Participants) | 111
  Serotype 15C at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 111
  Serotype 15F at Year 2:R | 0.0
  Serotype 16 at Year 2:R: number analyzed (Participants) | 111
  Serotype 16 at Year 2:R | 0.0
  Serotype 17 at Year 2:R: number analyzed (Participants) | 111
  Serotype 17 at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 111
  Serotype 19A at Year 2:R | 1.8
  Serotype 19F at Year 2:R: number analyzed (Participants) | 111
  Serotype 19F at Year 2:R | 0.0
  Serotype 20 at Year 2:R: number analyzed (Participants) | 111
  Serotype 20 at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 111
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 111
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 111
  Serotype 23A at Year 2:R | 0.0
  Serotype 23B at Year 2:R: number analyzed (Participants) | 111
  Serotype 23B at Year 2:R | 0.0
  Serotype 31 at Year 2:R: number analyzed (Participants) | 111
  Serotype 31 at Year 2:R | 0.0
  Serotype 33A at Year 2:R: number analyzed (Participants) | 111
  Serotype 33A at Year 2:R | 0.0
  Serotype 33F at Year 2:R: number analyzed (Participants) | 111
  Serotype 33F at Year 2:R | 0.0
  Serotype 34 at Year 2:R: number analyzed (Participants) | 111
  Serotype 34 at Year 2:R | 0.0
  Serotype 35B at Year 2:R: number analyzed (Participants) | 111
  Serotype 35B at Year 2:R | 0.0
  Serotype 35F at Year 2:R: number analyzed (Participants) | 111
  Serotype 35F at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 111
  Serotype 38 at Year 2:R | 0.0
  Serotype clumps at Year 2:R: number analyzed (Participants) | 111
  Serotype clumps at Year 2:R | 0.0
  Serotype Missing/non-viable at Year 2:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 111
  Serotype 3 at Year 3:R | 0.0
  Serotype 6C at Year 3:R: number analyzed (Participants) | 111
  Serotype 6C at Year 3:R | 0.0
  Serotype 7C at Year 3:R: number analyzed (Participants) | 111
  Serotype 7C at Year 3:R | 0.0
  Serotype 9N at Year 3:R: number analyzed (Participants) | 111
  Serotype 9N at Year 3:R | 0.0
  Serotype 10 at Year 3:R: number analyzed (Participants) | 111
  Serotype 10 at Year 3:R | 0.0
  Serotype 11 at Year 3:R: number analyzed (Participants) | 111
  Serotype 11 at Year 3:R | 0.0
  Serotype 12 at Year 3:R: number analyzed (Participants) | 111
  Serotype 12 at Year 3:R | 0.0
  Serotype 12F at Year 3:R: number analyzed (Participants) | 111
  Serotype 12F at Year 3:R | 0.0
  Serotype 13 at Year 3:R: number analyzed (Participants) | 111
  Serotype 13 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 111
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 111
  Serotype 15B at Year 3:R | 0.0
  Serotype 15C at Year 3:R: number analyzed (Participants) | 111
  Serotype 15C at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 111
  Serotype 15F at Year 3:R | 0.0
  Serotype 16 at Year 3:R: number analyzed (Participants) | 111
  Serotype 16 at Year 3:R | 0.0
  Serotype 17 at Year 3:R: number analyzed (Participants) | 111
  Serotype 17 at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 111
  Serotype 19A at Year 3:R | 2.7
  Serotype 19F at Year 3:R: number analyzed (Participants) | 111
  Serotype 19F at Year 3:R | 0.0
  Serotype 20 at Year 3:R: number analyzed (Participants) | 111
  Serotype 20 at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 111
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 111
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 111
  Serotype 23A at Year 3:R | 0.0
  Serotype 23B at Year 3:R: number analyzed (Participants) | 111
  Serotype 23B at Year 3:R | 0.0
  Serotype 31 at Year 3:R: number analyzed (Participants) | 111
  Serotype 31 at Year 3:R | 0.0
  Serotype 33A at Year 3:R: number analyzed (Participants) | 111
  Serotype 33A at Year 3:R | 0.0
  Serotype 33F at Year 3:R: number analyzed (Participants) | 111
  Serotype 33F at Year 3:R | 0.0
  Serotype 34 at Year 3:R: number analyzed (Participants) | 111
  Serotype 34 at Year 3:R | 0.0
  Serotype 35B at Year 3:R: number analyzed (Participants) | 111
  Serotype 35B at Year 3:R | 0.0
  Serotype 35F at Year 3:R: number analyzed (Participants) | 111
  Serotype 35F at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 111
  Serotype 38 at Year 3:R | 0.0
  Serotype clumps at Year 3:R: number analyzed (Participants) | 111
  Serotype clumps at Year 3:R | 0.0
  Serotype Missing/non-viable at Year 3:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:R | 0.0

8. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Cefotaxime: Middle Ear Fluid (MEF) Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for cefotaxime from MEF samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 19 A, 19 F, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38, clumps and missing or non-viable, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: MEF population. N (number of participants analyzed) includes total number of participants in MEF population, however actual 'N' for this OM is unknown as this data were not calculated as per planned analysis and number analyzed=number of isolates for the given serotype at specified time point.
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 135
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 135
  Serotype 3 at Year 1:S | 1.5
  Serotype 6C at Year 1:S: number analyzed (Participants) | 135
  Serotype 6C at Year 1:S | 2.2
  Serotype 7C at Year 1:S: number analyzed (Participants) | 135
  Serotype 7C at Year 1:S | 0.7
  Serotype 9N at Year 1:S: number analyzed (Participants) | 135
  Serotype 9N at Year 1:S | 0.0
  Serotype 10 at Year 1:S: number analyzed (Participants) | 135
  Serotype 10 at Year 1:S | 0.7
  Serotype 11 at Year 1:S: number analyzed (Participants) | 135
  Serotype 11 at Year 1:S | 0.0
  Serotype 12 at Year 1:S: number analyzed (Participants) | 135
  Serotype 12 at Year 1:S | 0.7
  Serotype 12F at Year 1:S: number analyzed (Participants) | 135
  Serotype 12F at Year 1:S | 0.0
  Serotype 13 at Year 1:S: number analyzed (Participants) | 135
  Serotype 13 at Year 1:S | 0.0
  Serotype 15A at Year 1:S: number analyzed (Participants) | 135
  Serotype 15A at Year 1:S | 2.2
  Serotype 15B at Year 1:S: number analyzed (Participants) | 135
  Serotype 15B at Year 1:S | 2.2
  Serotype 15C at Year 1:S: number analyzed (Participants) | 135
  Serotype 15C at Year 1:S | 0.7
  Serotype 15F at Year 1:S: number analyzed (Participants) | 135
  Serotype 15F at Year 1:S | 0.0
  Serotype 16 at Year 1:S: number analyzed (Participants) | 135
  Serotype 16 at Year 1:S | 0.7
  Serotype 17 at Year 1:S: number analyzed (Participants) | 135
  Serotype 17 at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 135
  Serotype 19A at Year 1:S | 5.9
  Serotype 19F at Year 1:S: number analyzed (Participants) | 135
  Serotype 19F at Year 1:S | 0.0
  Serotype 20 at Year 1:S: number analyzed (Participants) | 135
  Serotype 20 at Year 1:S | 0.0
  Serotype 21 at Year 1:S: number analyzed (Participants) | 135
  Serotype 21 at Year 1:S | 0.7
  Serotype 22F at Year 1:S: number analyzed (Participants) | 135
  Serotype 22F at Year 1:S | 0.7
  Serotype 23A at Year 1:S: number analyzed (Participants) | 135
  Serotype 23A at Year 1:S | 0.7
  Serotype 23B at Year 1:S: number analyzed (Participants) | 135
  Serotype 23B at Year 1:S | 0.7
  Serotype 31 at Year 1:S: number analyzed (Participants) | 135
  Serotype 31 at Year 1:S | 2.2
  Serotype 33A at Year 1:S: number analyzed (Participants) | 135
  Serotype 33A at Year 1:S | 0.0
  Serotype 33F at Year 1:S: number analyzed (Participants) | 135
  Serotype 33F at Year 1:S | 2.2
  Serotype 34 at Year 1:S: number analyzed (Participants) | 135
  Serotype 34 at Year 1:S | 0.0
  Serotype 35B at Year 1:S: number analyzed (Participants) | 135
  Serotype 35B at Year 1:S | 3.0
  Serotype 35F at Year 1:S: number analyzed (Participants) | 135
  Serotype 35F at Year 1:S | 0.0
  Serotype 38 at Year 1:S: number analyzed (Participants) | 135
  Serotype 38 at Year 1:S | 0.0
  Serotype clumps at Year 1:S: number analyzed (Participants) | 135
  Serotype clumps at Year 1:S | 1.5
  Serotype Missing/non-viable at Year 1:S: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:S | 0.7
  Serotype 3 at Year 2:S: number analyzed (Participants) | 111
  Serotype 3 at Year 2:S | 2.7
  Serotype 6C at Year 2:S: number analyzed (Participants) | 111
  Serotype 6C at Year 2:S | 1.8
  Serotype 7C at Year 2:S: number analyzed (Participants) | 111
  Serotype 7C at Year 2:S | 0.0
  Serotype 9N at Year 2:S: number analyzed (Participants) | 111
  Serotype 9N at Year 2:S | 0.0
  Serotype 10 at Year 2:S: number analyzed (Participants) | 111
  Serotype 10 at Year 2:S | 0.0
  Serotype 11 at Year 2:S: number analyzed (Participants) | 111
  Serotype 11 at Year 2:S | 2.7
  Serotype 12 at Year 2:S: number analyzed (Participants) | 111
  Serotype 12 at Year 2:S | 0.0
  Serotype 12F at Year 2:S: number analyzed (Participants) | 111
  Serotype 12F at Year 2:S | 0.0
  Serotype 13 at Year 2:S: number analyzed (Participants) | 111
  Serotype 13 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 111
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 111
  Serotype 15B at Year 2:S | 2.7
  Serotype 15C at Year 2:S: number analyzed (Participants) | 111
  Serotype 15C at Year 2:S | 0.0
  Serotype 15F at Year 2:S: number analyzed (Participants) | 111
  Serotype 15F at Year 2:S | 0.0
  Serotype 16 at Year 2:S: number analyzed (Participants) | 111
  Serotype 16 at Year 2:S | 0.9
  Serotype 17 at Year 2:S: number analyzed (Participants) | 111
  Serotype 17 at Year 2:S | 0.0
  Serotype 19A at Year 2:S: number analyzed (Participants) | 111
  Serotype 19A at Year 2:S | 2.7
  Serotype 19F at Year 2:S: number analyzed (Participants) | 111
  Serotype 19F at Year 2:S | 0.0
  Serotype 20 at Year 2:S: number analyzed (Participants) | 111
  Serotype 20 at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 111
  Serotype 21 at Year 2:S | 4.5
  Serotype 22F at Year 2:S: number analyzed (Participants) | 111
  Serotype 22F at Year 2:S | 0.9
  Serotype 23A at Year 2:S: number analyzed (Participants) | 111
  Serotype 23A at Year 2:S | 1.8
  Serotype 23B at Year 2:S: number analyzed (Participants) | 111
  Serotype 23B at Year 2:S | 2.7
  Serotype 31 at Year 2:S: number analyzed (Participants) | 111
  Serotype 31 at Year 2:S | 0.0
  Serotype 33A at Year 2:S: number analyzed (Participants) | 111
  Serotype 33A at Year 2:S | 0.0
  Serotype 33F at Year 2:S: number analyzed (Participants) | 111
  Serotype 33F at Year 2:S | 0.0
  Serotype 34 at Year 2:S: number analyzed (Participants) | 111
  Serotype 34 at Year 2:S | 0.0
  Serotype 35B at Year 2:S: number analyzed (Participants) | 111
  Serotype 35B at Year 2:S | 4.5
  Serotype 35F at Year 2:S: number analyzed (Participants) | 111
  Serotype 35F at Year 2:S | 0.0
  Serotype 38 at Year 2:S: number analyzed (Participants) | 111
  Serotype 38 at Year 2:S | 0.0
  Serotype clumps at Year 2:S: number analyzed (Participants) | 111
  Serotype clumps at Year 2:S | 0.9
  Serotype Missing/non-viable at Year 2:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:S | 0.0
  Serotype 3 at Year 3:S: number analyzed (Participants) | 111
  Serotype 3 at Year 3:S | 0.9
  Serotype 6C at Year 3:S: number analyzed (Participants) | 111
  Serotype 6C at Year 3:S | 0.9
  Serotype 7C at Year 3:S: number analyzed (Participants) | 111
  Serotype 7C at Year 3:S | 0.0
  Serotype 9N at Year 3:S: number analyzed (Participants) | 111
  Serotype 9N at Year 3:S | 0.0
  Serotype 10 at Year 3:S: number analyzed (Participants) | 111
  Serotype 10 at Year 3:S | 0.0
  Serotype 11 at Year 3:S: number analyzed (Participants) | 111
  Serotype 11 at Year 3:S | 0.9
  Serotype 12 at Year 3:S: number analyzed (Participants) | 111
  Serotype 12 at Year 3:S | 0.0
  Serotype 12F at Year 3:S: number analyzed (Participants) | 111
  Serotype 12F at Year 3:S | 0.0
  Serotype 13 at Year 3:S: number analyzed (Participants) | 111
  Serotype 13 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 111
  Serotype 15A at Year 3:S | 1.8
  Serotype 15B at Year 3:S: number analyzed (Participants) | 111
  Serotype 15B at Year 3:S | 0.0
  Serotype 15C at Year 3:S: number analyzed (Participants) | 111
  Serotype 15C at Year 3:S | 2.7
  Serotype 15F at Year 3:S: number analyzed (Participants) | 111
  Serotype 15F at Year 3:S | 0.0
  Serotype 16 at Year 3:S: number analyzed (Participants) | 111
  Serotype 16 at Year 3:S | 0.0
  Serotype 17 at Year 3:S: number analyzed (Participants) | 111
  Serotype 17 at Year 3:S | 0.0
  Serotype 19A at Year 3:S: number analyzed (Participants) | 111
  Serotype 19A at Year 3:S | 1.8
  Serotype 19F at Year 3:S: number analyzed (Participants) | 111
  Serotype 19F at Year 3:S | 2.7
  Serotype 20 at Year 3:S: number analyzed (Participants) | 111
  Serotype 20 at Year 3:S | 0.0
  Serotype 21 at Year 3:S: number analyzed (Participants) | 111
  Serotype 21 at Year 3:S | 0.9
  Serotype 22F at Year 3:S: number analyzed (Participants) | 111
  Serotype 22F at Year 3:S | 0.0
  Serotype 23A at Year 3:S: number analyzed (Participants) | 111
  Serotype 23A at Year 3:S | 0.0
  Serotype 23B at Year 3:S: number analyzed (Participants) | 111
  Serotype 23B at Year 3:S | 0.9
  Serotype 31 at Year 3:S: number analyzed (Participants) | 111
  Serotype 31 at Year 3:S | 0.9
  Serotype 33A at Year 3:S: number analyzed (Participants) | 111
  Serotype 33A at Year 3:S | 0.0
  Serotype 33F at Year 3:S: number analyzed (Participants) | 111
  Serotype 33F at Year 3:S | 1.8
  Serotype 34 at Year 3:S: number analyzed (Participants) | 111
  Serotype 34 at Year 3:S | 0.0
  Serotype 35B at Year 3:S: number analyzed (Participants) | 111
  Serotype 35B at Year 3:S | 2.7
  Serotype 35F at Year 3:S: number analyzed (Participants) | 111
  Serotype 35F at Year 3:S | 0.9
  Serotype 38 at Year 3:S: number analyzed (Participants) | 111
  Serotype 38 at Year 3:S | 0.0
  Serotype clumps at Year 3:S: number analyzed (Participants) | 111
  Serotype clumps at Year 3:S | 0.0
  Serotype Missing/non-viable at Year 3:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:S | 0.9
  Serotype 3 at Year 1:I: number analyzed (Participants) | 135
  Serotype 3 at Year 1:I | 0.0
  Serotype 6C at Year 1:I: number analyzed (Participants) | 135
  Serotype 6C at Year 1:I | 0.0
  Serotype 7C at Year 1:I: number analyzed (Participants) | 135
  Serotype 7C at Year 1:I | 0.0
  Serotype 9N at Year 1:I: number analyzed (Participants) | 135
  Serotype 9N at Year 1:I | 0.0
  Serotype 10 at Year 1:I: number analyzed (Participants) | 135
  Serotype 10 at Year 1:I | 0.0
  Serotype 11 at Year 1:I: number analyzed (Participants) | 135
  Serotype 11 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 135
  Serotype 12 at Year 1:I | 0.0
  Serotype 12F at Year 1:I: number analyzed (Participants) | 135
  Serotype 12F at Year 1:I | 0.0
  Serotype 13 at Year 1:I: number analyzed (Participants) | 135
  Serotype 13 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 135
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 135
  Serotype 15B at Year 1:I | 0.0
  Serotype 15C at Year 1:I: number analyzed (Participants) | 135
  Serotype 15C at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 135
  Serotype 15F at Year 1:I | 0.0
  Serotype 16 at Year 1:I: number analyzed (Participants) | 135
  Serotype 16 at Year 1:I | 0.0
  Serotype 17 at Year 1:I: number analyzed (Participants) | 135
  Serotype 17 at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 135
  Serotype 19A at Year 1:I | 7.4
  Serotype 19F at Year 1:I: number analyzed (Participants) | 135
  Serotype 19F at Year 1:I | 0.7
  Serotype 20 at Year 1:I: number analyzed (Participants) | 135
  Serotype 20 at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 135
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 135
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 135
  Serotype 23A at Year 1:I | 0.0
  Serotype 23B at Year 1:I: number analyzed (Participants) | 135
  Serotype 23B at Year 1:I | 0.0
  Serotype 31 at Year 1:I: number analyzed (Participants) | 135
  Serotype 31 at Year 1:I | 0.0
  Serotype 33A at Year 1:I: number analyzed (Participants) | 135
  Serotype 33A at Year 1:I | 0.0
  Serotype 33F at Year 1:I: number analyzed (Participants) | 135
  Serotype 33F at Year 1:I | 0.0
  Serotype 34 at Year 1:I: number analyzed (Participants) | 135
  Serotype 34 at Year 1:I | 0.0
  Serotype 35B at Year 1:I: number analyzed (Participants) | 135
  Serotype 35B at Year 1:I | 0.7
  Serotype 35F at Year 1:I: number analyzed (Participants) | 135
  Serotype 35F at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 135
  Serotype 38 at Year 1:I | 0.0
  Serotype clumps at Year 1:I: number analyzed (Participants) | 135
  Serotype clumps at Year 1:I | 0.0
  Serotype Missing/non-viable at Year 1:I: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 111
  Serotype 3 at Year 2:I | 0.0
  Serotype 6C at Year 2:I: number analyzed (Participants) | 111
  Serotype 6C at Year 2:I | 0.0
  Serotype 7C at Year 2:I: number analyzed (Participants) | 111
  Serotype 7C at Year 2:I | 0.0
  Serotype 9N at Year 2:I: number analyzed (Participants) | 111
  Serotype 9N at Year 2:I | 0.0
  Serotype 10 at Year 2:I: number analyzed (Participants) | 111
  Serotype 10 at Year 2:I | 0.0
  Serotype 11 at Year 2:I: number analyzed (Participants) | 111
  Serotype 11 at Year 2:I | 0.9
  Serotype 12 at Year 2:I: number analyzed (Participants) | 111
  Serotype 12 at Year 2:I | 0.0
  Serotype 12F at Year 2:I: number analyzed (Participants) | 111
  Serotype 12F at Year 2:I | 0.0
  Serotype 13 at Year 2:I: number analyzed (Participants) | 111
  Serotype 13 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 111
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 111
  Serotype 15B at Year 2:I | 0.0
  Serotype 15C at Year 2:I: number analyzed (Participants) | 111
  Serotype 15C at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 111
  Serotype 15F at Year 2:I | 0.0
  Serotype 16 at Year 2:I: number analyzed (Participants) | 111
  Serotype 16 at Year 2:I | 0.0
  Serotype 17 at Year 2:I: number analyzed (Participants) | 111
  Serotype 17 at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 111
  Serotype 19A at Year 2:I | 4.5
  Serotype 19F at Year 2:I: number analyzed (Participants) | 111
  Serotype 19F at Year 2:I | 0.0
  Serotype 20 at Year 2:I: number analyzed (Participants) | 111
  Serotype 20 at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 111
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 111
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 111
  Serotype 23A at Year 2:I | 0.0
  Serotype 23B at Year 2:I: number analyzed (Participants) | 111
  Serotype 23B at Year 2:I | 0.9
  Serotype 31 at Year 2:I: number analyzed (Participants) | 111
  Serotype 31 at Year 2:I | 0.0
  Serotype 33A at Year 2:I: number analyzed (Participants) | 111
  Serotype 33A at Year 2:I | 0.0
  Serotype 33F at Year 2:I: number analyzed (Participants) | 111
  Serotype 33F at Year 2:I | 0.0
  Serotype 34 at Year 2:I: number analyzed (Participants) | 111
  Serotype 34 at Year 2:I | 0.0
  Serotype 35B at Year 2:I: number analyzed (Participants) | 111
  Serotype 35B at Year 2:I | 0.9
  Serotype 35F at Year 2:I: number analyzed (Participants) | 111
  Serotype 35F at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 111
  Serotype 38 at Year 2:I | 0.0
  Serotype clumps at Year 2:I: number analyzed (Participants) | 111
  Serotype clumps at Year 2:I | 0.0
  Serotype Missing/non-viable at Year 2:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 111
  Serotype 3 at Year 3:I | 0.0
  Serotype 6C at Year 3:I: number analyzed (Participants) | 111
  Serotype 6C at Year 3:I | 0.0
  Serotype 7C at Year 3:I: number analyzed (Participants) | 111
  Serotype 7C at Year 3:I | 0.0
  Serotype 9N at Year 3:I: number analyzed (Participants) | 111
  Serotype 9N at Year 3:I | 0.0
  Serotype 10 at Year 3:I: number analyzed (Participants) | 111
  Serotype 10 at Year 3:I | 0.0
  Serotype 11 at Year 3:I: number analyzed (Participants) | 111
  Serotype 11 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 111
  Serotype 12 at Year 3:I | 0.0
  Serotype 12F at Year 3:I: number analyzed (Participants) | 111
  Serotype 12F at Year 3:I | 0.0
  Serotype 13 at Year 3:I: number analyzed (Participants) | 111
  Serotype 13 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 111
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 111
  Serotype 15B at Year 3:I | 0.0
  Serotype 15C at Year 3:I: number analyzed (Participants) | 111
  Serotype 15C at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 111
  Serotype 15F at Year 3:I | 0.0
  Serotype 16 at Year 3:I: number analyzed (Participants) | 111
  Serotype 16 at Year 3:I | 0.0
  Serotype 17 at Year 3:I: number analyzed (Participants) | 111
  Serotype 17 at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 111
  Serotype 19A at Year 3:I | 0.0
  Serotype 19F at Year 3:I: number analyzed (Participants) | 111
  Serotype 19F at Year 3:I | 0.9
  Serotype 20 at Year 3:I: number analyzed (Participants) | 111
  Serotype 20 at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 111
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 111
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 111
  Serotype 23A at Year 3:I | 0.0
  Serotype 23B at Year 3:I: number analyzed (Participants) | 111
  Serotype 23B at Year 3:I | 0.0
  Serotype 31 at Year 3:I: number analyzed (Participants) | 111
  Serotype 31 at Year 3:I | 0.0
  Serotype 33A at Year 3:I: number analyzed (Participants) | 111
  Serotype 33A at Year 3:I | 0.0
  Serotype 33F at Year 3:I: number analyzed (Participants) | 111
  Serotype 33F at Year 3:I | 0.0
  Serotype 34 at Year 3:I: number analyzed (Participants) | 111
  Serotype 34 at Year 3:I | 0.0
  Serotype 35B at Year 3:I: number analyzed (Participants) | 111
  Serotype 35B at Year 3:I | 0.0
  Serotype 35F at Year 3:I: number analyzed (Participants) | 111
  Serotype 35F at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 111
  Serotype 38 at Year 3:I | 0.0
  Serotype clumps at Year 3:I: number analyzed (Participants) | 111
  Serotype clumps at Year 3:I | 0.0
  Serotype Missing/non-viable at Year 3:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 135
  Serotype 3 at Year 1:R | 0.0
  Serotype 6C at Year 1:R: number analyzed (Participants) | 135
  Serotype 6C at Year 1:R | 0.0
  Serotype 7C at Year 1:R: number analyzed (Participants) | 135
  Serotype 7C at Year 1:R | 0.0
  Serotype 9N at Year 1:R: number analyzed (Participants) | 135
  Serotype 9N at Year 1:R | 0.0
  Serotype 10 at Year 1:R: number analyzed (Participants) | 135
  Serotype 10 at Year 1:R | 0.0
  Serotype 11 at Year 1:R: number analyzed (Participants) | 135
  Serotype 11 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 135
  Serotype 12 at Year 1:R | 0.0
  Serotype 12F at Year 1:R: number analyzed (Participants) | 135
  Serotype 12F at Year 1:R | 0.0
  Serotype 13 at Year 1:R: number analyzed (Participants) | 135
  Serotype 13 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 135
  Serotype 15A at Year 1:R | 0.0
  Serotype 15B at Year 1:R: number analyzed (Participants) | 135
  Serotype 15B at Year 1:R | 0.0
  Serotype 15C at Year 1:R: number analyzed (Participants) | 135
  Serotype 15C at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 135
  Serotype 15F at Year 1:R | 0.0
  Serotype 16 at Year 1:R: number analyzed (Participants) | 135
  Serotype 16 at Year 1:R | 0.0
  Serotype 17 at Year 1:R: number analyzed (Participants) | 135
  Serotype 17 at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 135
  Serotype 19A at Year 1:R | 1.5
  Serotype 19F at Year 1:R: number analyzed (Participants) | 135
  Serotype 19F at Year 1:R | 0.0
  Serotype 20 at Year 1:R: number analyzed (Participants) | 135
  Serotype 20 at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 135
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 135
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 135
  Serotype 23A at Year 1:R | 0.0
  Serotype 23B at Year 1:R: number analyzed (Participants) | 135
  Serotype 23B at Year 1:R | 0.0
  Serotype 31 at Year 1:R: number analyzed (Participants) | 135
  Serotype 31 at Year 1:R | 0.0
  Serotype 33A at Year 1:R: number analyzed (Participants) | 135
  Serotype 33A at Year 1:R | 0.0
  Serotype 33F at Year 1:R: number analyzed (Participants) | 135
  Serotype 33F at Year 1:R | 0.0
  Serotype 34 at Year 1:R: number analyzed (Participants) | 135
  Serotype 34 at Year 1:R | 0.0
  Serotype 35B at Year 1:R: number analyzed (Participants) | 135
  Serotype 35B at Year 1:R | 0.0
  Serotype 35F at Year 1:R: number analyzed (Participants) | 135
  Serotype 35F at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 135
  Serotype 38 at Year 1:R | 0.0
  Serotype clumps at Year 1:R: number analyzed (Participants) | 135
  Serotype clumps at Year 1:R | 0.0
  Serotype Missing/non-viable at Year 1:R: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 111
  Serotype 3 at Year 2:R | 0.0
  Serotype 6C at Year 2:R: number analyzed (Participants) | 111
  Serotype 6C at Year 2:R | 0.0
  Serotype 7C at Year 2:R: number analyzed (Participants) | 111
  Serotype 7C at Year 2:R | 0.0
  Serotype 9N at Year 2:R: number analyzed (Participants) | 111
  Serotype 9N at Year 2:R | 0.0
  Serotype 10 at Year 2:R: number analyzed (Participants) | 111
  Serotype 10 at Year 2:R | 0.0
  Serotype 11 at Year 2:R: number analyzed (Participants) | 111
  Serotype 11 at Year 2:R | 0.0
  Serotype 12 at Year 2:R: number analyzed (Participants) | 111
  Serotype 12 at Year 2:R | 0.0
  Serotype 12F at Year 2:R: number analyzed (Participants) | 111
  Serotype 12F at Year 2:R | 0.0
  Serotype 13 at Year 2:R: number analyzed (Participants) | 111
  Serotype 13 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 111
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 111
  Serotype 15B at Year 2:R | 0.0
  Serotype 15C at Year 2:R: number analyzed (Participants) | 111
  Serotype 15C at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 111
  Serotype 15F at Year 2:R | 0.0
  Serotype 16 at Year 2:R: number analyzed (Participants) | 111
  Serotype 16 at Year 2:R | 0.0
  Serotype 17 at Year 2:R: number analyzed (Participants) | 111
  Serotype 17 at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 111
  Serotype 19A at Year 2:R | 0.0
  Serotype 19F at Year 2:R: number analyzed (Participants) | 111
  Serotype 19F at Year 2:R | 0.0
  Serotype 20 at Year 2:R: number analyzed (Participants) | 111
  Serotype 20 at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 111
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 111
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 111
  Serotype 23A at Year 2:R | 0.0
  Serotype 23B at Year 2:R: number analyzed (Participants) | 111
  Serotype 23B at Year 2:R | 0.0
  Serotype 31 at Year 2:R: number analyzed (Participants) | 111
  Serotype 31 at Year 2:R | 0.0
  Serotype 33A at Year 2:R: number analyzed (Participants) | 111
  Serotype 33A at Year 2:R | 0.0
  Serotype 33F at Year 2:R: number analyzed (Participants) | 111
  Serotype 33F at Year 2:R | 0.0
  Serotype 34 at Year 2:R: number analyzed (Participants) | 111
  Serotype 34 at Year 2:R | 0.0
  Serotype 35B at Year 2:R: number analyzed (Participants) | 111
  Serotype 35B at Year 2:R | 0.0
  Serotype 35F at Year 2:R: number analyzed (Participants) | 111
  Serotype 35F at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 111
  Serotype 38 at Year 2:R | 0.0
  Serotype clumps at Year 2:R: number analyzed (Participants) | 111
  Serotype clumps at Year 2:R | 0.0
  Serotype Missing/non-viable at Year 2:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 111
  Serotype 3 at Year 3:R | 0.0
  Serotype 6C at Year 3:R: number analyzed (Participants) | 111
  Serotype 6C at Year 3:R | 0.0
  Serotype 7C at Year 3:R: number analyzed (Participants) | 111
  Serotype 7C at Year 3:R | 0.0
  Serotype 9N at Year 3:R: number analyzed (Participants) | 111
  Serotype 9N at Year 3:R | 0.0
  Serotype 10 at Year 3:R: number analyzed (Participants) | 111
  Serotype 10 at Year 3:R | 0.0
  Serotype 11 at Year 3:R: number analyzed (Participants) | 111
  Serotype 11 at Year 3:R | 0.0
  Serotype 12 at Year 3:R: number analyzed (Participants) | 111
  Serotype 12 at Year 3:R | 0.0
  Serotype 12F at Year 3:R: number analyzed (Participants) | 111
  Serotype 12F at Year 3:R | 0.0
  Serotype 13 at Year 3:R: number analyzed (Participants) | 111
  Serotype 13 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 111
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 111
  Serotype 15B at Year 3:R | 0.0
  Serotype 15C at Year 3:R: number analyzed (Participants) | 111
  Serotype 15C at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 111
  Serotype 15F at Year 3:R | 0.0
  Serotype 16 at Year 3:R: number analyzed (Participants) | 111
  Serotype 16 at Year 3:R | 0.0
  Serotype 17 at Year 3:R: number analyzed (Participants) | 111
  Serotype 17 at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 111
  Serotype 19A at Year 3:R | 0.0
  Serotype 19F at Year 3:R: number analyzed (Participants) | 111
  Serotype 19F at Year 3:R | 0.0
  Serotype 20 at Year 3:R: number analyzed (Participants) | 111
  Serotype 20 at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 111
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 111
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 111
  Serotype 23A at Year 3:R | 0.0
  Serotype 23B at Year 3:R: number analyzed (Participants) | 111
  Serotype 23B at Year 3:R | 0.0
  Serotype 31 at Year 3:R: number analyzed (Participants) | 111
  Serotype 31 at Year 3:R | 0.0
  Serotype 33A at Year 3:R: number analyzed (Participants) | 111
  Serotype 33A at Year 3:R | 0.0
  Serotype 33F at Year 3:R: number analyzed (Participants) | 111
  Serotype 33F at Year 3:R | 0.0
  Serotype 34 at Year 3:R: number analyzed (Participants) | 111
  Serotype 34 at Year 3:R | 0.0
  Serotype 35B at Year 3:R: number analyzed (Participants) | 111
  Serotype 35B at Year 3:R | 0.0
  Serotype 35F at Year 3:R: number analyzed (Participants) | 111
  Serotype 35F at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 111
  Serotype 38 at Year 3:R | 0.0
  Serotype clumps at Year 3:R: number analyzed (Participants) | 111
  Serotype clumps at Year 3:R | 0.0
  Serotype Missing/non-viable at Year 3:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:R | 0.0

9. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Ceftriaxone: Middle Ear Fluid (MEF) Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for ceftriaxone from MEF samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 19 A, 19 F, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38, clumps and missing or non-viable, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: MEF population. N (number of participants analyzed) includes total number of participants in MEF population, however actual 'N' for this OM is unknown as this data were not calculated as per planned analysis and n=number of isolates for the given serotype at specified time point.
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 135
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 135
  Serotype 3 at Year 1:S | 5.9
  Serotype 6C at Year 1:S: number analyzed (Participants) | 135
  Serotype 6C at Year 1:S | 6.7
  Serotype 7C at Year 1:S: number analyzed (Participants) | 135
  Serotype 7C at Year 1:S | 1.5
  Serotype 9N at Year 1:S: number analyzed (Participants) | 135
  Serotype 9N at Year 1:S | 2.2
  Serotype 10 at Year 1:S: number analyzed (Participants) | 135
  Serotype 10 at Year 1:S | 3.0
  Serotype 11 at Year 1:S: number analyzed (Participants) | 135
  Serotype 11 at Year 1:S | 3.7
  Serotype 12 at Year 1:S: number analyzed (Participants) | 135
  Serotype 12 at Year 1:S | 0.7
  Serotype 12F at Year 1:S: number analyzed (Participants) | 135
  Serotype 12F at Year 1:S | 0.0
  Serotype 13 at Year 1:S: number analyzed (Participants) | 135
  Serotype 13 at Year 1:S | 0.7
  Serotype 15A at Year 1:S: number analyzed (Participants) | 135
  Serotype 15A at Year 1:S | 3.7
  Serotype 15B at Year 1:S: number analyzed (Participants) | 135
  Serotype 15B at Year 1:S | 4.4
  Serotype 15C at Year 1:S: number analyzed (Participants) | 135
  Serotype 15C at Year 1:S | 3.7
  Serotype 15F at Year 1:S: number analyzed (Participants) | 135
  Serotype 15F at Year 1:S | 0.0
  Serotype 16 at Year 1:S: number analyzed (Participants) | 135
  Serotype 16 at Year 1:S | 1.5
  Serotype 17 at Year 1:S: number analyzed (Participants) | 135
  Serotype 17 at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 135
  Serotype 19A at Year 1:S | 20.7
  Serotype 19F at Year 1:S: number analyzed (Participants) | 135
  Serotype 19F at Year 1:S | 1.5
  Serotype 20 at Year 1:S: number analyzed (Participants) | 135
  Serotype 20 at Year 1:S | 0.0
  Serotype 21 at Year 1:S: number analyzed (Participants) | 135
  Serotype 21 at Year 1:S | 3.0
  Serotype 22F at Year 1:S: number analyzed (Participants) | 135
  Serotype 22F at Year 1:S | 1.5
  Serotype 23A at Year 1:S: number analyzed (Participants) | 135
  Serotype 23A at Year 1:S | 3.0
  Serotype 23B at Year 1:S: number analyzed (Participants) | 135
  Serotype 23B at Year 1:S | 0.7
  Serotype 31 at Year 1:S: number analyzed (Participants) | 135
  Serotype 31 at Year 1:S | 2.2
  Serotype 33A at Year 1:S: number analyzed (Participants) | 135
  Serotype 33A at Year 1:S | 0.7
  Serotype 33F at Year 1:S: number analyzed (Participants) | 135
  Serotype 33F at Year 1:S | 3.0
  Serotype 34 at Year 1:S: number analyzed (Participants) | 135
  Serotype 34 at Year 1:S | 0.0
  Serotype 35B at Year 1:S: number analyzed (Participants) | 135
  Serotype 35B at Year 1:S | 6.7
  Serotype 35F at Year 1:S: number analyzed (Participants) | 135
  Serotype 35F at Year 1:S | 0.0
  Serotype 38 at Year 1:S: number analyzed (Participants) | 135
  Serotype 38 at Year 1:S | 0.7
  Serotype clumps at Year 1:S: number analyzed (Participants) | 135
  Serotype clumps at Year 1:S | 0.7
  Serotype Missing/non-viable at Year 1:S: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:S | 0.7
  Serotype 3 at Year 2:S: number analyzed (Participants) | 111
  Serotype 3 at Year 2:S | 6.3
  Serotype 6C at Year 2:S: number analyzed (Participants) | 111
  Serotype 6C at Year 2:S | 3.6
  Serotype 7C at Year 2:S: number analyzed (Participants) | 111
  Serotype 7C at Year 2:S | 0.0
  Serotype 9N at Year 2:S: number analyzed (Participants) | 111
  Serotype 9N at Year 2:S | 0.0
  Serotype 10 at Year 2:S: number analyzed (Participants) | 111
  Serotype 10 at Year 2:S | 0.9
  Serotype 11 at Year 2:S: number analyzed (Participants) | 111
  Serotype 11 at Year 2:S | 6.3
  Serotype 12 at Year 2:S: number analyzed (Participants) | 111
  Serotype 12 at Year 2:S | 0.0
  Serotype 12F at Year 2:S: number analyzed (Participants) | 111
  Serotype 12F at Year 2:S | 0.9
  Serotype 13 at Year 2:S: number analyzed (Participants) | 111
  Serotype 13 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 111
  Serotype 15A at Year 2:S | 0.9
  Serotype 15B at Year 2:S: number analyzed (Participants) | 111
  Serotype 15B at Year 2:S | 3.6
  Serotype 15C at Year 2:S: number analyzed (Participants) | 111
  Serotype 15C at Year 2:S | 2.7
  Serotype 15F at Year 2:S: number analyzed (Participants) | 111
  Serotype 15F at Year 2:S | 0.0
  Serotype 16 at Year 2:S: number analyzed (Participants) | 111
  Serotype 16 at Year 2:S | 2.7
  Serotype 17 at Year 2:S: number analyzed (Participants) | 111
  Serotype 17 at Year 2:S | 1.8
  Serotype 19A at Year 2:S: number analyzed (Participants) | 111
  Serotype 19A at Year 2:S | 13.5
  Serotype 19F at Year 2:S: number analyzed (Participants) | 111
  Serotype 19F at Year 2:S | 0.9
  Serotype 20 at Year 2:S: number analyzed (Participants) | 111
  Serotype 20 at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 111
  Serotype 21 at Year 2:S | 9.0
  Serotype 22F at Year 2:S: number analyzed (Participants) | 111
  Serotype 22F at Year 2:S | 0.9
  Serotype 23A at Year 2:S: number analyzed (Participants) | 111
  Serotype 23A at Year 2:S | 4.5
  Serotype 23B at Year 2:S: number analyzed (Participants) | 111
  Serotype 23B at Year 2:S | 6.3
  Serotype 31 at Year 2:S: number analyzed (Participants) | 111
  Serotype 31 at Year 2:S | 1.8
  Serotype 33A at Year 2:S: number analyzed (Participants) | 111
  Serotype 33A at Year 2:S | 0.0
  Serotype 33F at Year 2:S: number analyzed (Participants) | 111
  Serotype 33F at Year 2:S | 0.0
  Serotype 34 at Year 2:S: number analyzed (Participants) | 111
  Serotype 34 at Year 2:S | 0.9
  Serotype 35B at Year 2:S: number analyzed (Participants) | 111
  Serotype 35B at Year 2:S | 11.7
  Serotype 35F at Year 2:S: number analyzed (Participants) | 111
  Serotype 35F at Year 2:S | 0.9
  Serotype 38 at Year 2:S: number analyzed (Participants) | 111
  Serotype 38 at Year 2:S | 0.9
  Serotype clumps at Year 2:S: number analyzed (Participants) | 111
  Serotype clumps at Year 2:S | 0.9
  Serotype Missing/non-viable at Year 2:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:S | 0.9
  Serotype 3 at Year 3:S: number analyzed (Participants) | 111
  Serotype 3 at Year 3:S | 6.3
  Serotype 6C at Year 3:S: number analyzed (Participants) | 111
  Serotype 6C at Year 3:S | 1.8
  Serotype 7C at Year 3:S: number analyzed (Participants) | 111
  Serotype 7C at Year 3:S | 0.0
  Serotype 9N at Year 3:S: number analyzed (Participants) | 111
  Serotype 9N at Year 3:S | 0.9
  Serotype 10 at Year 3:S: number analyzed (Participants) | 111
  Serotype 10 at Year 3:S | 2.7
  Serotype 11 at Year 3:S: number analyzed (Participants) | 111
  Serotype 11 at Year 3:S | 3.6
  Serotype 12 at Year 3:S: number analyzed (Participants) | 111
  Serotype 12 at Year 3:S | 0.0
  Serotype 12F at Year 3:S: number analyzed (Participants) | 111
  Serotype 12F at Year 3:S | 0.0
  Serotype 13 at Year 3:S: number analyzed (Participants) | 111
  Serotype 13 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 111
  Serotype 15A at Year 3:S | 6.3
  Serotype 15B at Year 3:S: number analyzed (Participants) | 111
  Serotype 15B at Year 3:S | 4.5
  Serotype 15C at Year 3:S: number analyzed (Participants) | 111
  Serotype 15C at Year 3:S | 5.4
  Serotype 15F at Year 3:S: number analyzed (Participants) | 111
  Serotype 15F at Year 3:S | 0.9
  Serotype 16 at Year 3:S: number analyzed (Participants) | 111
  Serotype 16 at Year 3:S | 4.5
  Serotype 17 at Year 3:S: number analyzed (Participants) | 111
  Serotype 17 at Year 3:S | 0.9
  Serotype 19A at Year 3:S: number analyzed (Participants) | 111
  Serotype 19A at Year 3:S | 5.4
  Serotype 19F at Year 3:S: number analyzed (Participants) | 111
  Serotype 19F at Year 3:S | 4.5
  Serotype 20 at Year 3:S: number analyzed (Participants) | 111
  Serotype 20 at Year 3:S | 0.9
  Serotype 21 at Year 3:S: number analyzed (Participants) | 111
  Serotype 21 at Year 3:S | 5.4
  Serotype 22F at Year 3:S: number analyzed (Participants) | 111
  Serotype 22F at Year 3:S | 1.8
  Serotype 23A at Year 3:S: number analyzed (Participants) | 111
  Serotype 23A at Year 3:S | 2.7
  Serotype 23B at Year 3:S: number analyzed (Participants) | 111
  Serotype 23B at Year 3:S | 8.1
  Serotype 31 at Year 3:S: number analyzed (Participants) | 111
  Serotype 31 at Year 3:S | 4.5
  Serotype 33A at Year 3:S: number analyzed (Participants) | 111
  Serotype 33A at Year 3:S | 0.0
  Serotype 33F at Year 3:S: number analyzed (Participants) | 111
  Serotype 33F at Year 3:S | 1.8
  Serotype 34 at Year 3:S: number analyzed (Participants) | 111
  Serotype 34 at Year 3:S | 0.9
  Serotype 35B at Year 3:S: number analyzed (Participants) | 111
  Serotype 35B at Year 3:S | 9.9
  Serotype 35F at Year 3:S: number analyzed (Participants) | 111
  Serotype 35F at Year 3:S | 1.8
  Serotype 38 at Year 3:S: number analyzed (Participants) | 111
  Serotype 38 at Year 3:S | 0.9
  Serotype clumps at Year 3:S: number analyzed (Participants) | 111
  Serotype clumps at Year 3:S | 0.0
  Serotype Missing/non-viable at Year 3:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:S | 0.9
  Serotype 3 at Year 1:I: number analyzed (Participants) | 135
  Serotype 3 at Year 1:I | 0.0
  Serotype 6C at Year 1:I: number analyzed (Participants) | 135
  Serotype 6C at Year 1:I | 0.0
  Serotype 7C at Year 1:I: number analyzed (Participants) | 135
  Serotype 7C at Year 1:I | 0.0
  Serotype 9N at Year 1:I: number analyzed (Participants) | 135
  Serotype 9N at Year 1:I | 0.0
  Serotype 10 at Year 1:I: number analyzed (Participants) | 135
  Serotype 10 at Year 1:I | 0.0
  Serotype 11 at Year 1:I: number analyzed (Participants) | 135
  Serotype 11 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 135
  Serotype 12 at Year 1:I | 0.0
  Serotype 12F at Year 1:I: number analyzed (Participants) | 135
  Serotype 12F at Year 1:I | 0.0
  Serotype 13 at Year 1:I: number analyzed (Participants) | 135
  Serotype 13 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 135
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 135
  Serotype 15B at Year 1:I | 0.0
  Serotype 15C at Year 1:I: number analyzed (Participants) | 135
  Serotype 15C at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 135
  Serotype 15F at Year 1:I | 0.0
  Serotype 16 at Year 1:I: number analyzed (Participants) | 135
  Serotype 16 at Year 1:I | 0.0
  Serotype 17 at Year 1:I: number analyzed (Participants) | 135
  Serotype 17 at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 135
  Serotype 19A at Year 1:I | 8.1
  Serotype 19F at Year 1:I: number analyzed (Participants) | 135
  Serotype 19F at Year 1:I | 0.7
  Serotype 20 at Year 1:I: number analyzed (Participants) | 135
  Serotype 20 at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 135
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 135
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 135
  Serotype 23A at Year 1:I | 0.0
  Serotype 23B at Year 1:I: number analyzed (Participants) | 135
  Serotype 23B at Year 1:I | 0.0
  Serotype 31 at Year 1:I: number analyzed (Participants) | 135
  Serotype 31 at Year 1:I | 0.0
  Serotype 33A at Year 1:I: number analyzed (Participants) | 135
  Serotype 33A at Year 1:I | 0.0
  Serotype 33F at Year 1:I: number analyzed (Participants) | 135
  Serotype 33F at Year 1:I | 0.0
  Serotype 34 at Year 1:I: number analyzed (Participants) | 135
  Serotype 34 at Year 1:I | 0.0
  Serotype 35B at Year 1:I: number analyzed (Participants) | 135
  Serotype 35B at Year 1:I | 0.0
  Serotype 35F at Year 1:I: number analyzed (Participants) | 135
  Serotype 35F at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 135
  Serotype 38 at Year 1:I | 0.0
  Serotype clumps at Year 1:I: number analyzed (Participants) | 135
  Serotype clumps at Year 1:I | 0.0
  Serotype Missing/non-viable at Year 1:I: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 111
  Serotype 3 at Year 2:I | 0.0
  Serotype 6C at Year 2:I: number analyzed (Participants) | 111
  Serotype 6C at Year 2:I | 0.0
  Serotype 7C at Year 2:I: number analyzed (Participants) | 111
  Serotype 7C at Year 2:I | 0.0
  Serotype 9N at Year 2:I: number analyzed (Participants) | 111
  Serotype 9N at Year 2:I | 0.0
  Serotype 10 at Year 2:I: number analyzed (Participants) | 111
  Serotype 10 at Year 2:I | 0.0
  Serotype 11 at Year 2:I: number analyzed (Participants) | 111
  Serotype 11 at Year 2:I | 0.9
  Serotype 12 at Year 2:I: number analyzed (Participants) | 111
  Serotype 12 at Year 2:I | 0.0
  Serotype 12F at Year 2:I: number analyzed (Participants) | 111
  Serotype 12F at Year 2:I | 0.0
  Serotype 13 at Year 2:I: number analyzed (Participants) | 111
  Serotype 13 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 111
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 111
  Serotype 15B at Year 2:I | 0.0
  Serotype 15C at Year 2:I: number analyzed (Participants) | 111
  Serotype 15C at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 111
  Serotype 15F at Year 2:I | 0.0
  Serotype 16 at Year 2:I: number analyzed (Participants) | 111
  Serotype 16 at Year 2:I | 0.0
  Serotype 17 at Year 2:I: number analyzed (Participants) | 111
  Serotype 17 at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 111
  Serotype 19A at Year 2:I | 7.2
  Serotype 19F at Year 2:I: number analyzed (Participants) | 111
  Serotype 19F at Year 2:I | 0.0
  Serotype 20 at Year 2:I: number analyzed (Participants) | 111
  Serotype 20 at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 111
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 111
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 111
  Serotype 23A at Year 2:I | 0.0
  Serotype 23B at Year 2:I: number analyzed (Participants) | 111
  Serotype 23B at Year 2:I | 0.9
  Serotype 31 at Year 2:I: number analyzed (Participants) | 111
  Serotype 31 at Year 2:I | 0.0
  Serotype 33A at Year 2:I: number analyzed (Participants) | 111
  Serotype 33A at Year 2:I | 0.0
  Serotype 33F at Year 2:I: number analyzed (Participants) | 111
  Serotype 33F at Year 2:I | 0.0
  Serotype 34 at Year 2:I: number analyzed (Participants) | 111
  Serotype 34 at Year 2:I | 0.0
  Serotype 35B at Year 2:I: number analyzed (Participants) | 111
  Serotype 35B at Year 2:I | 0.0
  Serotype 35F at Year 2:I: number analyzed (Participants) | 111
  Serotype 35F at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 111
  Serotype 38 at Year 2:I | 0.0
  Serotype clumps at Year 2:I: number analyzed (Participants) | 111
  Serotype clumps at Year 2:I | 0.0
  Serotype Missing/non-viable at Year 2:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 111
  Serotype 3 at Year 3:I | 0.9
  Serotype 6C at Year 3:I: number analyzed (Participants) | 111
  Serotype 6C at Year 3:I | 0.0
  Serotype 7C at Year 3:I: number analyzed (Participants) | 111
  Serotype 7C at Year 3:I | 0.0
  Serotype 9N at Year 3:I: number analyzed (Participants) | 111
  Serotype 9N at Year 3:I | 0.0
  Serotype 10 at Year 3:I: number analyzed (Participants) | 111
  Serotype 10 at Year 3:I | 0.0
  Serotype 11 at Year 3:I: number analyzed (Participants) | 111
  Serotype 11 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 111
  Serotype 12 at Year 3:I | 0.0
  Serotype 12F at Year 3:I: number analyzed (Participants) | 111
  Serotype 12F at Year 3:I | 0.0
  Serotype 13 at Year 3:I: number analyzed (Participants) | 111
  Serotype 13 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 111
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 111
  Serotype 15B at Year 3:I | 0.0
  Serotype 15C at Year 3:I: number analyzed (Participants) | 111
  Serotype 15C at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 111
  Serotype 15F at Year 3:I | 0.0
  Serotype 16 at Year 3:I: number analyzed (Participants) | 111
  Serotype 16 at Year 3:I | 0.0
  Serotype 17 at Year 3:I: number analyzed (Participants) | 111
  Serotype 17 at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 111
  Serotype 19A at Year 3:I | 2.7
  Serotype 19F at Year 3:I: number analyzed (Participants) | 111
  Serotype 19F at Year 3:I | 0.9
  Serotype 20 at Year 3:I: number analyzed (Participants) | 111
  Serotype 20 at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 111
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 111
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 111
  Serotype 23A at Year 3:I | 0.0
  Serotype 23B at Year 3:I: number analyzed (Participants) | 111
  Serotype 23B at Year 3:I | 0.0
  Serotype 31 at Year 3:I: number analyzed (Participants) | 111
  Serotype 31 at Year 3:I | 0.0
  Serotype 33A at Year 3:I: number analyzed (Participants) | 111
  Serotype 33A at Year 3:I | 0.0
  Serotype 33F at Year 3:I: number analyzed (Participants) | 111
  Serotype 33F at Year 3:I | 0.0
  Serotype 34 at Year 3:I: number analyzed (Participants) | 111
  Serotype 34 at Year 3:I | 0.0
  Serotype 35B at Year 3:I: number analyzed (Participants) | 111
  Serotype 35B at Year 3:I | 0.0
  Serotype 35F at Year 3:I: number analyzed (Participants) | 111
  Serotype 35F at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 111
  Serotype 38 at Year 3:I | 0.0
  Serotype clumps at Year 3:I: number analyzed (Participants) | 111
  Serotype clumps at Year 3:I | 0.0
  Serotype Missing/non-viable at Year 3:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 135
  Serotype 3 at Year 1:R | 0.0
  Serotype 6C at Year 1:R: number analyzed (Participants) | 135
  Serotype 6C at Year 1:R | 0.0
  Serotype 7C at Year 1:R: number analyzed (Participants) | 135
  Serotype 7C at Year 1:R | 0.0
  Serotype 9N at Year 1:R: number analyzed (Participants) | 135
  Serotype 9N at Year 1:R | 0.0
  Serotype 10 at Year 1:R: number analyzed (Participants) | 135
  Serotype 10 at Year 1:R | 0.0
  Serotype 11 at Year 1:R: number analyzed (Participants) | 135
  Serotype 11 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 135
  Serotype 12 at Year 1:R | 0.0
  Serotype 12F at Year 1:R: number analyzed (Participants) | 135
  Serotype 12F at Year 1:R | 0.0
  Serotype 13 at Year 1:R: number analyzed (Participants) | 135
  Serotype 13 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 135
  Serotype 15A at Year 1:R | 0.0
  Serotype 15B at Year 1:R: number analyzed (Participants) | 135
  Serotype 15B at Year 1:R | 0.0
  Serotype 15C at Year 1:R: number analyzed (Participants) | 135
  Serotype 15C at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 135
  Serotype 15F at Year 1:R | 0.0
  Serotype 16 at Year 1:R: number analyzed (Participants) | 135
  Serotype 16 at Year 1:R | 0.0
  Serotype 17 at Year 1:R: number analyzed (Participants) | 135
  Serotype 17 at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 135
  Serotype 19A at Year 1:R | 1.5
  Serotype 19F at Year 1:R: number analyzed (Participants) | 135
  Serotype 19F at Year 1:R | 0.0
  Serotype 20 at Year 1:R: number analyzed (Participants) | 135
  Serotype 20 at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 135
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 135
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 135
  Serotype 23A at Year 1:R | 0.0
  Serotype 23B at Year 1:R: number analyzed (Participants) | 135
  Serotype 23B at Year 1:R | 0.0
  Serotype 31 at Year 1:R: number analyzed (Participants) | 135
  Serotype 31 at Year 1:R | 0.0
  Serotype 33A at Year 1:R: number analyzed (Participants) | 135
  Serotype 33A at Year 1:R | 0.0
  Serotype 33F at Year 1:R: number analyzed (Participants) | 135
  Serotype 33F at Year 1:R | 0.0
  Serotype 34 at Year 1:R: number analyzed (Participants) | 135
  Serotype 34 at Year 1:R | 0.0
  Serotype 35B at Year 1:R: number analyzed (Participants) | 135
  Serotype 35B at Year 1:R | 0.0
  Serotype 35F at Year 1:R: number analyzed (Participants) | 135
  Serotype 35F at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 135
  Serotype 38 at Year 1:R | 0.0
  Serotype clumps at Year 1:R: number analyzed (Participants) | 135
  Serotype clumps at Year 1:R | 0.0
  Serotype Missing/non-viable at Year 1:R: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 111
  Serotype 3 at Year 2:R | 0.0
  Serotype 6C at Year 2:R: number analyzed (Participants) | 111
  Serotype 6C at Year 2:R | 0.0
  Serotype 7C at Year 2:R: number analyzed (Participants) | 111
  Serotype 7C at Year 2:R | 0.0
  Serotype 9N at Year 2:R: number analyzed (Participants) | 111
  Serotype 9N at Year 2:R | 0.0
  Serotype 10 at Year 2:R: number analyzed (Participants) | 111
  Serotype 10 at Year 2:R | 0.0
  Serotype 11 at Year 2:R: number analyzed (Participants) | 111
  Serotype 11 at Year 2:R | 0.0
  Serotype 12 at Year 2:R: number analyzed (Participants) | 111
  Serotype 12 at Year 2:R | 0.0
  Serotype 12F at Year 2:R: number analyzed (Participants) | 111
  Serotype 12F at Year 2:R | 0.0
  Serotype 13 at Year 2:R: number analyzed (Participants) | 111
  Serotype 13 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 111
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 111
  Serotype 15B at Year 2:R | 0.0
  Serotype 15C at Year 2:R: number analyzed (Participants) | 111
  Serotype 15C at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 111
  Serotype 15F at Year 2:R | 0.0
  Serotype 16 at Year 2:R: number analyzed (Participants) | 111
  Serotype 16 at Year 2:R | 0.0
  Serotype 17 at Year 2:R: number analyzed (Participants) | 111
  Serotype 17 at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 111
  Serotype 19A at Year 2:R | 0.0
  Serotype 19F at Year 2:R: number analyzed (Participants) | 111
  Serotype 19F at Year 2:R | 0.0
  Serotype 20 at Year 2:R: number analyzed (Participants) | 111
  Serotype 20 at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 111
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 111
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 111
  Serotype 23A at Year 2:R | 0.0
  Serotype 23B at Year 2:R: number analyzed (Participants) | 111
  Serotype 23B at Year 2:R | 0.0
  Serotype 31 at Year 2:R: number analyzed (Participants) | 111
  Serotype 31 at Year 2:R | 0.0
  Serotype 33A at Year 2:R: number analyzed (Participants) | 111
  Serotype 33A at Year 2:R | 0.0
  Serotype 33F at Year 2:R: number analyzed (Participants) | 111
  Serotype 33F at Year 2:R | 0.0
  Serotype 34 at Year 2:R: number analyzed (Participants) | 111
  Serotype 34 at Year 2:R | 0.0
  Serotype 35B at Year 2:R: number analyzed (Participants) | 111
  Serotype 35B at Year 2:R | 0.0
  Serotype 35F at Year 2:R: number analyzed (Participants) | 111
  Serotype 35F at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 111
  Serotype 38 at Year 2:R | 0.0
  Serotype clumps at Year 2:R: number analyzed (Participants) | 111
  Serotype clumps at Year 2:R | 0.0
  Serotype Missing/non-viable at Year 2:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 111
  Serotype 3 at Year 3:R | 0.0
  Serotype 6C at Year 3:R: number analyzed (Participants) | 111
  Serotype 6C at Year 3:R | 0.0
  Serotype 7C at Year 3:R: number analyzed (Participants) | 111
  Serotype 7C at Year 3:R | 0.0
  Serotype 9N at Year 3:R: number analyzed (Participants) | 111
  Serotype 9N at Year 3:R | 0.0
  Serotype 10 at Year 3:R: number analyzed (Participants) | 111
  Serotype 10 at Year 3:R | 0.0
  Serotype 11 at Year 3:R: number analyzed (Participants) | 111
  Serotype 11 at Year 3:R | 0.0
  Serotype 12 at Year 3:R: number analyzed (Participants) | 111
  Serotype 12 at Year 3:R | 0.0
  Serotype 12F at Year 3:R: number analyzed (Participants) | 111
  Serotype 12F at Year 3:R | 0.0
  Serotype 13 at Year 3:R: number analyzed (Participants) | 111
  Serotype 13 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 111
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 111
  Serotype 15B at Year 3:R | 0.0
  Serotype 15C at Year 3:R: number analyzed (Participants) | 111
  Serotype 15C at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 111
  Serotype 15F at Year 3:R | 0.0
  Serotype 16 at Year 3:R: number analyzed (Participants) | 111
  Serotype 16 at Year 3:R | 0.0
  Serotype 17 at Year 3:R: number analyzed (Participants) | 111
  Serotype 17 at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 111
  Serotype 19A at Year 3:R | 0.9
  Serotype 19F at Year 3:R: number analyzed (Participants) | 111
  Serotype 19F at Year 3:R | 0.0
  Serotype 20 at Year 3:R: number analyzed (Participants) | 111
  Serotype 20 at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 111
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 111
  Serotype 22F at Year 3:R | 0.9
  Serotype 23A at Year 3:R: number analyzed (Participants) | 111
  Serotype 23A at Year 3:R | 0.0
  Serotype 23B at Year 3:R: number analyzed (Participants) | 111
  Serotype 23B at Year 3:R | 0.0
  Serotype 31 at Year 3:R: number analyzed (Participants) | 111
  Serotype 31 at Year 3:R | 0.0
  Serotype 33A at Year 3:R: number analyzed (Participants) | 111
  Serotype 33A at Year 3:R | 0.0
  Serotype 33F at Year 3:R: number analyzed (Participants) | 111
  Serotype 33F at Year 3:R | 0.0
  Serotype 34 at Year 3:R: number analyzed (Participants) | 111
  Serotype 34 at Year 3:R | 0.0
  Serotype 35B at Year 3:R: number analyzed (Participants) | 111
  Serotype 35B at Year 3:R | 0.0
  Serotype 35F at Year 3:R: number analyzed (Participants) | 111
  Serotype 35F at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 111
  Serotype 38 at Year 3:R | 0.0
  Serotype clumps at Year 3:R: number analyzed (Participants) | 111
  Serotype clumps at Year 3:R | 0.0
  Serotype Missing/non-viable at Year 3:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:R | 0.0

10. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Clindamycin: Middle Ear Fluid (MEF) Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for clindamycin from MEF samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 19 A, 19 F, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38, clumps and missing or non-viable, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: as for outcome 8
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 135
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 135
  Serotype 3 at Year 1:S | 4.4
  Serotype 9N at Year 1:S: number analyzed (Participants) | 135
  Serotype 9N at Year 1:S | 0.0
  Serotype 10 at Year 1:S: number analyzed (Participants) | 135
  Serotype 10 at Year 1:S | 1.5
  Serotype 11 at Year 1:S: number analyzed (Participants) | 135
  Serotype 11 at Year 1:S | 1.5
  Serotype 12 at Year 1:S: number analyzed (Participants) | 135
  Serotype 12 at Year 1:S | 0.7
  Serotype 12F at Year 1:S: number analyzed (Participants) | 135
  Serotype 12F at Year 1:S | 0.0
  Serotype 13 at Year 1:S: number analyzed (Participants) | 135
  Serotype 13 at Year 1:S | 0.0
  Serotype 15A at Year 1:S: number analyzed (Participants) | 135
  Serotype 15A at Year 1:S | 0.7
  Serotype 15B at Year 1:S: number analyzed (Participants) | 135
  Serotype 15B at Year 1:S | 2.2
  Serotype 15C at Year 1:S: number analyzed (Participants) | 135
  Serotype 15C at Year 1:S | 3.0
  Serotype 15F at Year 1:S: number analyzed (Participants) | 135
  Serotype 15F at Year 1:S | 0.0
  Serotype 16 at Year 1:S: number analyzed (Participants) | 135
  Serotype 16 at Year 1:S | 0.0
  Serotype 17 at Year 1:S: number analyzed (Participants) | 135
  Serotype 17 at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 135
  Serotype 19A at Year 1:S | 3.0
  Serotype 19F at Year 1:S: number analyzed (Participants) | 135
  Serotype 19F at Year 1:S | 0.7
  Serotype 20 at Year 1:S: number analyzed (Participants) | 135
  Serotype 20 at Year 1:S | 0.0
  Serotype 21 at Year 1:S: number analyzed (Participants) | 135
  Serotype 21 at Year 1:S | 1.5
  Serotype 22F at Year 1:S: number analyzed (Participants) | 135
  Serotype 22F at Year 1:S | 0.0
  Serotype 23A at Year 1:S: number analyzed (Participants) | 135
  Serotype 23A at Year 1:S | 2.2
  Serotype 23B at Year 1:S: number analyzed (Participants) | 135
  Serotype 23B at Year 1:S | 0.7
  Serotype 31 at Year 1:S: number analyzed (Participants) | 135
  Serotype 31 at Year 1:S | 1.5
  Serotype 33A at Year 1:S: number analyzed (Participants) | 135
  Serotype 33A at Year 1:S | 0.7
  Serotype 33F at Year 1:S: number analyzed (Participants) | 135
  Serotype 33F at Year 1:S | 0.7
  Serotype 34 at Year 1:S: number analyzed (Participants) | 135
  Serotype 34 at Year 1:S | 0.0
  Serotype 35B at Year 1:S: number analyzed (Participants) | 135
  Serotype 35B at Year 1:S | 5.9
  Serotype 35F at Year 1:S: number analyzed (Participants) | 135
  Serotype 35F at Year 1:S | 0.0
  Serotype 38 at Year 1:S: number analyzed (Participants) | 135
  Serotype 38 at Year 1:S | 0.0
  Serotype clumps at Year 1:S: number analyzed (Participants) | 135
  Serotype clumps at Year 1:S | 0.0
  Serotype Missing/non-viable at Year 1:S: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:S | 0.0
  Serotype 3 at Year 2:S: number analyzed (Participants) | 111
  Serotype 3 at Year 2:S | 4.5
  Serotype 6C at Year 2:S: number analyzed (Participants) | 111
  Serotype 6C at Year 2:S | 2.7
  Serotype 7C at Year 2:S: number analyzed (Participants) | 111
  Serotype 7C at Year 2:S | 0.0
  Serotype 9N at Year 2:S: number analyzed (Participants) | 111
  Serotype 9N at Year 2:S | 0.0
  Serotype 10 at Year 2:S: number analyzed (Participants) | 111
  Serotype 10 at Year 2:S | 0.9
  Serotype 11 at Year 2:S: number analyzed (Participants) | 111
  Serotype 11 at Year 2:S | 3.6
  Serotype 12 at Year 2:S: number analyzed (Participants) | 111
  Serotype 12 at Year 2:S | 0.0
  Serotype 12F at Year 2:S: number analyzed (Participants) | 111
  Serotype 12F at Year 2:S | 0.9
  Serotype 13 at Year 2:S: number analyzed (Participants) | 111
  Serotype 13 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 111
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 111
  Serotype 15B at Year 2:S | 1.8
  Serotype 15C at Year 2:S: number analyzed (Participants) | 111
  Serotype 15C at Year 2:S | 2.7
  Serotype 15F at Year 2:S: number analyzed (Participants) | 111
  Serotype 15F at Year 2:S | 0.0
  Serotype 16 at Year 2:S: number analyzed (Participants) | 111
  Serotype 16 at Year 2:S | 1.8
  Serotype 17 at Year 2:S: number analyzed (Participants) | 111
  Serotype 17 at Year 2:S | 1.8
  Serotype 19A at Year 2:S: number analyzed (Participants) | 111
  Serotype 19A at Year 2:S | 2.7
  Serotype 19F at Year 2:S: number analyzed (Participants) | 111
  Serotype 19F at Year 2:S | 0.9
  Serotype 20 at Year 2:S: number analyzed (Participants) | 111
  Serotype 20 at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 111
  Serotype 21 at Year 2:S | 5.4
  Serotype 22F at Year 2:S: number analyzed (Participants) | 111
  Serotype 22F at Year 2:S | 0.0
  Serotype 23A at Year 2:S: number analyzed (Participants) | 111
  Serotype 23A at Year 2:S | 1.8
  Serotype 23B at Year 2:S: number analyzed (Participants) | 111
  Serotype 23B at Year 2:S | 6.3
  Serotype 31 at Year 2:S: number analyzed (Participants) | 111
  Serotype 31 at Year 2:S | 1.8
  Serotype 33A at Year 2:S: number analyzed (Participants) | 111
  Serotype 33A at Year 2:S | 0.0
  Serotype 33F at Year 2:S: number analyzed (Participants) | 111
  Serotype 33F at Year 2:S | 0.0
  Serotype 34 at Year 2:S: number analyzed (Participants) | 111
  Serotype 34 at Year 2:S | 0.9
  Serotype 35B at Year 2:S: number analyzed (Participants) | 111
  Serotype 35B at Year 2:S | 9.0
  Serotype 35F at Year 2:S: number analyzed (Participants) | 111
  Serotype 35F at Year 2:S | 0.9
  Serotype 38 at Year 2:S: number analyzed (Participants) | 111
  Serotype 38 at Year 2:S | 0.9
  Serotype clumps at Year 2:S: number analyzed (Participants) | 111
  Serotype clumps at Year 2:S | 0.0
  Serotype Missing/non-viable at Year 2:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:S | 0.9
  Serotype 3 at Year 3:S: number analyzed (Participants) | 111
  Serotype 3 at Year 3:S | 3.6
  Serotype 6C at Year 3:S: number analyzed (Participants) | 111
  Serotype 6C at Year 3:S | 0.0
  Serotype 7C at Year 3:S: number analyzed (Participants) | 111
  Serotype 7C at Year 3:S | 0.0
  Serotype 9N at Year 3:S: number analyzed (Participants) | 111
  Serotype 9N at Year 3:S | 0.9
  Serotype 10 at Year 3:S: number analyzed (Participants) | 111
  Serotype 10 at Year 3:S | 1.8
  Serotype 11 at Year 3:S: number analyzed (Participants) | 111
  Serotype 11 at Year 3:S | 1.8
  Serotype 12 at Year 3:S: number analyzed (Participants) | 111
  Serotype 12 at Year 3:S | 0.0
  Serotype 12F at Year 3:S: number analyzed (Participants) | 111
  Serotype 12F at Year 3:S | 0.0
  Serotype 13 at Year 3:S: number analyzed (Participants) | 111
  Serotype 13 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 111
  Serotype 15A at Year 3:S | 2.7
  Serotype 15B at Year 3:S: number analyzed (Participants) | 111
  Serotype 15B at Year 3:S | 2.7
  Serotype 15C at Year 3:S: number analyzed (Participants) | 111
  Serotype 15C at Year 3:S | 2.7
  Serotype 15F at Year 3:S: number analyzed (Participants) | 111
  Serotype 15F at Year 3:S | 0.0
  Serotype 16 at Year 3:S: number analyzed (Participants) | 111
  Serotype 16 at Year 3:S | 3.6
  Serotype 17 at Year 3:S: number analyzed (Participants) | 111
  Serotype 17 at Year 3:S | 0.9
  Serotype 19A at Year 3:S: number analyzed (Participants) | 111
  Serotype 19A at Year 3:S | 1.8
  Serotype 19F at Year 3:S: number analyzed (Participants) | 111
  Serotype 19F at Year 3:S | 2.7
  Serotype 20 at Year 3:S: number analyzed (Participants) | 111
  Serotype 20 at Year 3:S | 0.9
  Serotype 21 at Year 3:S: number analyzed (Participants) | 111
  Serotype 21 at Year 3:S | 1.8
  Serotype 22F at Year 3:S: number analyzed (Participants) | 111
  Serotype 22F at Year 3:S | 0.0
  Serotype 23A at Year 3:S: number analyzed (Participants) | 111
  Serotype 23A at Year 3:S | 2.7
  Serotype 23B at Year 3:S: number analyzed (Participants) | 111
  Serotype 23B at Year 3:S | 7.2
  Serotype 31 at Year 3:S: number analyzed (Participants) | 111
  Serotype 31 at Year 3:S | 2.7
  Serotype 33A at Year 3:S: number analyzed (Participants) | 111
  Serotype 33A at Year 3:S | 0.0
  Serotype 33F at Year 3:S: number analyzed (Participants) | 111
  Serotype 33F at Year 3:S | 1.8
  Serotype 34 at Year 3:S: number analyzed (Participants) | 111
  Serotype 34 at Year 3:S | 0.0
  Serotype 35B at Year 3:S: number analyzed (Participants) | 111
  Serotype 35B at Year 3:S | 6.3
  Serotype 35F at Year 3:S: number analyzed (Participants) | 111
  Serotype 35F at Year 3:S | 0.9
  Serotype 38 at Year 3:S: number analyzed (Participants) | 111
  Serotype 38 at Year 3:S | 0.9
  Serotype clumps at Year 3:S: number analyzed (Participants) | 111
  Serotype clumps at Year 3:S | 0.0
  Serotype Missing/non-viable at Year 3:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:S | 1.8
  Serotype 6C at Year 1:S: number analyzed (Participants) | 135
  Serotype 6C at Year 1:S | 4.4
  Serotype 7C at Year 1:S: number analyzed (Participants) | 135
  Serotype 7C at Year 1:S | 0.0
  Serotype 3 at Year 1:I: number analyzed (Participants) | 135
  Serotype 3 at Year 1:I | 0.0
  Serotype 6C at Year 1:I: number analyzed (Participants) | 135
  Serotype 6C at Year 1:I | 0.0
  Serotype 7C at Year 1:I: number analyzed (Participants) | 135
  Serotype 7C at Year 1:I | 0.0
  Serotype 9N at Year 1:I: number analyzed (Participants) | 135
  Serotype 9N at Year 1:I | 0.7
  Serotype 10 at Year 1:I: number analyzed (Participants) | 135
  Serotype 10 at Year 1:I | 0.0
  Serotype 11 at Year 1:I: number analyzed (Participants) | 135
  Serotype 11 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 135
  Serotype 12 at Year 1:I | 0.0
  Serotype 12F at Year 1:I: number analyzed (Participants) | 135
  Serotype 12F at Year 1:I | 0.0
  Serotype 13 at Year 1:I: number analyzed (Participants) | 135
  Serotype 13 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 135
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 135
  Serotype 15B at Year 1:I | 0.0
  Serotype 15C at Year 1:I: number analyzed (Participants) | 135
  Serotype 15C at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 135
  Serotype 15F at Year 1:I | 0.0
  Serotype 16 at Year 1:I: number analyzed (Participants) | 135
  Serotype 16 at Year 1:I | 0.0
  Serotype 17 at Year 1:I: number analyzed (Participants) | 135
  Serotype 17 at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 135
  Serotype 19A at Year 1:I | 5.2
  Serotype 19F at Year 1:I: number analyzed (Participants) | 135
  Serotype 19F at Year 1:I | 0.0
  Serotype 20 at Year 1:I: number analyzed (Participants) | 135
  Serotype 20 at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 135
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 135
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 135
  Serotype 23A at Year 1:I | 0.0
  Serotype 23B at Year 1:I: number analyzed (Participants) | 135
  Serotype 23B at Year 1:I | 0.0
  Serotype 31 at Year 1:I: number analyzed (Participants) | 135
  Serotype 31 at Year 1:I | 0.0
  Serotype 33A at Year 1:I: number analyzed (Participants) | 135
  Serotype 33A at Year 1:I | 0.0
  Serotype 33F at Year 1:I: number analyzed (Participants) | 135
  Serotype 33F at Year 1:I | 0.7
  Serotype 34 at Year 1:I: number analyzed (Participants) | 135
  Serotype 34 at Year 1:I | 0.0
  Serotype 35B at Year 1:I: number analyzed (Participants) | 135
  Serotype 35B at Year 1:I | 0.0
  Serotype 35F at Year 1:I: number analyzed (Participants) | 135
  Serotype 35F at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 135
  Serotype 38 at Year 1:I | 0.0
  Serotype clumps at Year 1:I: number analyzed (Participants) | 135
  Serotype clumps at Year 1:I | 0.0
  Serotype Missing/non-viable at Year 1:I: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 111
  Serotype 3 at Year 2:I | 0.0
  Serotype 6C at Year 2:I: number analyzed (Participants) | 111
  Serotype 6C at Year 2:I | 0.0
  Serotype 7C at Year 2:I: number analyzed (Participants) | 111
  Serotype 7C at Year 2:I | 0.0
  Serotype 9N at Year 2:I: number analyzed (Participants) | 111
  Serotype 9N at Year 2:I | 0.0
  Serotype 10 at Year 2:I: number analyzed (Participants) | 111
  Serotype 10 at Year 2:I | 0.0
  Serotype 11 at Year 2:I: number analyzed (Participants) | 111
  Serotype 11 at Year 2:I | 0.0
  Serotype 12 at Year 2:I: number analyzed (Participants) | 111
  Serotype 12 at Year 2:I | 0.0
  Serotype 12F at Year 2:I: number analyzed (Participants) | 111
  Serotype 12F at Year 2:I | 0.0
  Serotype 13 at Year 2:I: number analyzed (Participants) | 111
  Serotype 13 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 111
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 111
  Serotype 15B at Year 2:I | 0.0
  Serotype 15C at Year 2:I: number analyzed (Participants) | 111
  Serotype 15C at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 111
  Serotype 15F at Year 2:I | 0.0
  Serotype 16 at Year 2:I: number analyzed (Participants) | 111
  Serotype 16 at Year 2:I | 0.0
  Serotype 17 at Year 2:I: number analyzed (Participants) | 111
  Serotype 17 at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 111
  Serotype 19A at Year 2:I | 0.9
  Serotype 19F at Year 2:I: number analyzed (Participants) | 111
  Serotype 19F at Year 2:I | 0.0
  Serotype 20 at Year 2:I: number analyzed (Participants) | 111
  Serotype 20 at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 111
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 111
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 111
  Serotype 23A at Year 2:I | 0.9
  Serotype 23B at Year 2:I: number analyzed (Participants) | 111
  Serotype 23B at Year 2:I | 0.0
  Serotype 31 at Year 2:I: number analyzed (Participants) | 111
  Serotype 31 at Year 2:I | 0.0
  Serotype 33A at Year 2:I: number analyzed (Participants) | 111
  Serotype 33A at Year 2:I | 0.0
  Serotype 33F at Year 2:I: number analyzed (Participants) | 111
  Serotype 33F at Year 2:I | 0.0
  Serotype 34 at Year 2:I: number analyzed (Participants) | 111
  Serotype 34 at Year 2:I | 0.0
  Serotype 35B at Year 2:I1: number analyzed (Participants) | 111
  Serotype 35B at Year 2:I1 | 0.9
  Serotype 35F at Year 2:I: number analyzed (Participants) | 111
  Serotype 35F at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 111
  Serotype 38 at Year 2:I | 0.0
  Serotype clumps at Year 2:I: number analyzed (Participants) | 111
  Serotype clumps at Year 2:I | 0.0
  Serotype Missing/non-viable at Year 2:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 111
  Serotype 3 at Year 3:I | 0.0
  Serotype 6C at Year 3:I: number analyzed (Participants) | 111
  Serotype 6C at Year 3:I | 0.0
  Serotype 7C at Year 3:I: number analyzed (Participants) | 111
  Serotype 7C at Year 3:I | 0.0
  Serotype 9N at Year 3:I: number analyzed (Participants) | 111
  Serotype 9N at Year 3:I | 0.0
  Serotype 10 at Year 3:I: number analyzed (Participants) | 111
  Serotype 10 at Year 3:I | 0.0
  Serotype 11 at Year 3:I: number analyzed (Participants) | 111
  Serotype 11 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 111
  Serotype 12 at Year 3:I | 0.0
  Serotype 12F at Year 3:I: number analyzed (Participants) | 111
  Serotype 12F at Year 3:I | 0.0
  Serotype 13 at Year 3:I: number analyzed (Participants) | 111
  Serotype 13 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 111
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 111
  Serotype 15B at Year 3:I | 0.9
  Serotype 15C at Year 3:I: number analyzed (Participants) | 111
  Serotype 15C at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 111
  Serotype 15F at Year 3:I | 0.0
  Serotype 16 at Year 3:I: number analyzed (Participants) | 111
  Serotype 16 at Year 3:I | 0.0
  Serotype 17 at Year 3:I: number analyzed (Participants) | 111
  Serotype 17 at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 111
  Serotype 19A at Year 3:I | 0.0
  Serotype 19F at Year 3:I: number analyzed (Participants) | 111
  Serotype 19F at Year 3:I | 0.9
  Serotype 20 at Year 3:I: number analyzed (Participants) | 111
  Serotype 20 at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 111
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 111
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 111
  Serotype 23A at Year 3:I | 0.0
  Serotype 23B at Year 3:I: number analyzed (Participants) | 111
  Serotype 23B at Year 3:I | 0.0
  Serotype 31 at Year 3:I: number analyzed (Participants) | 111
  Serotype 31 at Year 3:I | 0.0
  Serotype 33A at Year 3:I: number analyzed (Participants) | 111
  Serotype 33A at Year 3:I | 0.0
  Serotype 33F at Year 3:I: number analyzed (Participants) | 111
  Serotype 33F at Year 3:I | 0.0
  Serotype 34 at Year 3:I: number analyzed (Participants) | 111
  Serotype 34 at Year 3:I | 0.0
  Serotype 35B at Year 3:I: number analyzed (Participants) | 111
  Serotype 35B at Year 3:I | 2.7
  Serotype 35F at Year 3:I: number analyzed (Participants) | 111
  Serotype 35F at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 111
  Serotype 38 at Year 3:I | 0.0
  Serotype clumps at Year 3:I: number analyzed (Participants) | 111
  Serotype clumps at Year 3:I | 0.0
  Serotype Missing/non-viable at Year 3:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 135
  Serotype 3 at Year 1:R | 0.0
  Serotype 6C at Year 1:R: number analyzed (Participants) | 135
  Serotype 6C at Year 1:R | 0.0
  Serotype 7C at Year 1:R: number analyzed (Participants) | 135
  Serotype 7C at Year 1:R | 0.0
  Serotype 9N at Year 1:R: number analyzed (Participants) | 135
  Serotype 9N at Year 1:R | 0.0
  Serotype 10 at Year 1:R: number analyzed (Participants) | 135
  Serotype 10 at Year 1:R | 0.0
  Serotype 11 at Year 1:R: number analyzed (Participants) | 135
  Serotype 11 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 135
  Serotype 12 at Year 1:R | 0.0
  Serotype 12F at Year 1:R: number analyzed (Participants) | 135
  Serotype 12F at Year 1:R | 0.0
  Serotype 13 at Year 1:R: number analyzed (Participants) | 135
  Serotype 13 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 135
  Serotype 15A at Year 1:R | 2.2
  Serotype 15B at Year 1:R: number analyzed (Participants) | 135
  Serotype 15B at Year 1:R | 0.0
  Serotype 15C at Year 1:R: number analyzed (Participants) | 135
  Serotype 15C at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 135
  Serotype 15F at Year 1:R | 0.0
  Serotype 16 at Year 1:R: number analyzed (Participants) | 135
  Serotype 16 at Year 1:R | 0.0
  Serotype 17 at Year 1:R: number analyzed (Participants) | 135
  Serotype 17 at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 135
  Serotype 19A at Year 1:R | 12.6
  Serotype 19F at Year 1:R: number analyzed (Participants) | 135
  Serotype 19F at Year 1:R | 0.0
  Serotype 20 at Year 1:R: number analyzed (Participants) | 135
  Serotype 20 at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 135
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 135
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 135
  Serotype 23A at Year 1:R | 0.0
  Serotype 23B at Year 1:R: number analyzed (Participants) | 135
  Serotype 23B at Year 1:R | 0.0
  Serotype 31 at Year 1:R: number analyzed (Participants) | 135
  Serotype 31 at Year 1:R | 0.0
  Serotype 33A at Year 1:R: number analyzed (Participants) | 135
  Serotype 33A at Year 1:R | 0.0
  Serotype 33F at Year 1:R: number analyzed (Participants) | 135
  Serotype 33F at Year 1:R | 0.0
  Serotype 34 at Year 1:R: number analyzed (Participants) | 135
  Serotype 34 at Year 1:R | 0.0
  Serotype 35B at Year 1:R: number analyzed (Participants) | 135
  Serotype 35B at Year 1:R | 0.0
  Serotype 35F at Year 1:R: number analyzed (Participants) | 135
  Serotype 35F at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 135
  Serotype 38 at Year 1:R | 0.0
  Serotype clumps at Year 1:R: number analyzed (Participants) | 135
  Serotype clumps at Year 1:R | 0.0
  Serotype Missing/non-viable at Year 1:R: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 111
  Serotype 3 at Year 2:R | 0.0
  Serotype 6C at Year 2:R: number analyzed (Participants) | 111
  Serotype 6C at Year 2:R | 0.0
  Serotype 7C at Year 2:R: number analyzed (Participants) | 111
  Serotype 7C at Year 2:R | 0.0
  Serotype 9N at Year 2:R: number analyzed (Participants) | 111
  Serotype 9N at Year 2:R | 0.0
  Serotype 10 at Year 2:R: number analyzed (Participants) | 111
  Serotype 10 at Year 2:R | 0.0
  Serotype 11 at Year 2:R: number analyzed (Participants) | 111
  Serotype 11 at Year 2:R | 0.9
  Serotype 12 at Year 2:R: number analyzed (Participants) | 111
  Serotype 12 at Year 2:R | 0.0
  Serotype 12F at Year 2:R: number analyzed (Participants) | 111
  Serotype 12F at Year 2:R | 0.0
  Serotype 13 at Year 2:R: number analyzed (Participants) | 111
  Serotype 13 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 111
  Serotype 15A at Year 2:R | 0.9
  Serotype 15B at Year 2:R: number analyzed (Participants) | 111
  Serotype 15B at Year 2:R | 0.0
  Serotype 15C at Year 2:R: number analyzed (Participants) | 111
  Serotype 15C at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 111
  Serotype 15F at Year 2:R | 0.0
  Serotype 16 at Year 2:R: number analyzed (Participants) | 111
  Serotype 16 at Year 2:R | 0.0
  Serotype 17 at Year 2:R: number analyzed (Participants) | 111
  Serotype 17 at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 111
  Serotype 19A at Year 2:R | 6.3
  Serotype 19F at Year 2:R: number analyzed (Participants) | 111
  Serotype 19F at Year 2:R | 0.0
  Serotype 20 at Year 2:R: number analyzed (Participants) | 111
  Serotype 20 at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 111
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 111
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 111
  Serotype 23A at Year 2:R | 0.0
  Serotype 23B at Year 2:R: number analyzed (Participants) | 111
  Serotype 23B at Year 2:R | 0.0
  Serotype 31 at Year 2:R: number analyzed (Participants) | 111
  Serotype 31 at Year 2:R | 0.0
  Serotype 33A at Year 2:R: number analyzed (Participants) | 111
  Serotype 33A at Year 2:R | 0.0
  Serotype 33F at Year 2:R: number analyzed (Participants) | 111
  Serotype 33F at Year 2:R | 0.0
  Serotype 34 at Year 2:R: number analyzed (Participants) | 111
  Serotype 34 at Year 2:R | 0.0
  Serotype 35B at Year 2:R: number analyzed (Participants) | 111
  Serotype 35B at Year 2:R | 0.9
  Serotype 35F at Year 2:R: number analyzed (Participants) | 111
  Serotype 35F at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 111
  Serotype 38 at Year 2:R | 0.0
  Serotype clumps at Year 2:R: number analyzed (Participants) | 111
  Serotype clumps at Year 2:R | 0.0
  Serotype Missing/non-viable at Year 2:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 111
  Serotype 3 at Year 3:R | 0.0
  Serotype 6C at Year 3:R: number analyzed (Participants) | 111
  Serotype 6C at Year 3:R | 0.0
  Serotype 7C at Year 3:R: number analyzed (Participants) | 111
  Serotype 7C at Year 3:R | 0.0
  Serotype 9N at Year 3:R: number analyzed (Participants) | 111
  Serotype 9N at Year 3:R | 0.0
  Serotype 10 at Year 3:R: number analyzed (Participants) | 111
  Serotype 10 at Year 3:R | 0.0
  Serotype 11 at Year 3:R: number analyzed (Participants) | 111
  Serotype 11 at Year 3:R | 0.0
  Serotype 12 at Year 3:R: number analyzed (Participants) | 111
  Serotype 12 at Year 3:R | 0.0
  Serotype 12F at Year 3:R: number analyzed (Participants) | 111
  Serotype 12F at Year 3:R | 0.0
  Serotype 13 at Year 3:R: number analyzed (Participants) | 111
  Serotype 13 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 111
  Serotype 15A at Year 3:R | 0.9
  Serotype 15B at Year 3:R: number analyzed (Participants) | 111
  Serotype 15B at Year 3:R | 0.0
  Serotype 15C at Year 3:R: number analyzed (Participants) | 111
  Serotype 15C at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 111
  Serotype 15F at Year 3:R | 0.0
  Serotype 16 at Year 3:R: number analyzed (Participants) | 111
  Serotype 16 at Year 3:R | 0.0
  Serotype 17 at Year 3:R: number analyzed (Participants) | 111
  Serotype 17 at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 111
  Serotype 19A at Year 3:R | 4.5
  Serotype 19F at Year 3:R: number analyzed (Participants) | 111
  Serotype 19F at Year 3:R | 0.9
  Serotype 20 at Year 3:R: number analyzed (Participants) | 111
  Serotype 20 at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 111
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 111
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 111
  Serotype 23A at Year 3:R | 0.0
  Serotype 23B at Year 3:R: number analyzed (Participants) | 111
  Serotype 23B at Year 3:R | 0.0
  Serotype 31 at Year 3:R: number analyzed (Participants) | 111
  Serotype 31 at Year 3:R | 0.0
  Serotype 33A at Year 3:R: number analyzed (Participants) | 111
  Serotype 33A at Year 3:R | 0.0
  Serotype 33F at Year 3:R: number analyzed (Participants) | 111
  Serotype 33F at Year 3:R | 0.0
  Serotype 34 at Year 3:R: number analyzed (Participants) | 111
  Serotype 34 at Year 3:R | 0.0
  Serotype 35B at Year 3:R: number analyzed (Participants) | 111
  Serotype 35B at Year 3:R | 0.9
  Serotype 35F at Year 3:R: number analyzed (Participants) | 111
  Serotype 35F at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 111
  Serotype 38 at Year 3:R | 0.0
  Serotype clumps at Year 3:R: number analyzed (Participants) | 111
  Serotype clumps at Year 3:R | 0.0
  Serotype Missing/non-viable at Year 3:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:R | 0.0

11. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Erythromycin: Middle Ear Fluid (MEF) Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for erythromycin from MEF samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 19A, 19F, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38, clumps and missing or non-viable, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: as for outcome 8
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 135
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 135
  Serotype 3 at Year 1:S | 5.9
  Serotype 6C at Year 1:S: number analyzed (Participants) | 135
  Serotype 6C at Year 1:S | 4.4
  Serotype 7C at Year 1:S: number analyzed (Participants) | 135
  Serotype 7C at Year 1:S | 1.5
  Serotype 9N at Year 1:S: number analyzed (Participants) | 135
  Serotype 9N at Year 1:S | 2.2
  Serotype 10 at Year 1:S: number analyzed (Participants) | 135
  Serotype 10 at Year 1:S | 3.0
  Serotype 11 at Year 1:S: number analyzed (Participants) | 135
  Serotype 11 at Year 1:S | 3.0
  Serotype 12 at Year 1:S: number analyzed (Participants) | 135
  Serotype 12 at Year 1:S | 0.7
  Serotype 12F at Year 1:S: number analyzed (Participants) | 135
  Serotype 12F at Year 1:S | 0.0
  Serotype 13 at Year 1:S: number analyzed (Participants) | 135
  Serotype 13 at Year 1:S | 0.0
  Serotype 15A at Year 1:S: number analyzed (Participants) | 135
  Serotype 15A at Year 1:S | 1.5
  Serotype 15B at Year 1:S: number analyzed (Participants) | 135
  Serotype 15B at Year 1:S | 3.0
  Serotype 15C at Year 1:S: number analyzed (Participants) | 135
  Serotype 15C at Year 1:S | 1.5
  Serotype 15F at Year 1:S: number analyzed (Participants) | 135
  Serotype 15F at Year 1:S | 0.0
  Serotype 16 at Year 1:S: number analyzed (Participants) | 135
  Serotype 16 at Year 1:S | 1.5
  Serotype 17 at Year 1:S: number analyzed (Participants) | 135
  Serotype 17 at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 135
  Serotype 19A at Year 1:S | 1.5
  Serotype 19F at Year 1:S: number analyzed (Participants) | 135
  Serotype 19F at Year 1:S | 0.7
  Serotype 20 at Year 1:S: number analyzed (Participants) | 135
  Serotype 20 at Year 1:S | 0.0
  Serotype 21 at Year 1:S: number analyzed (Participants) | 135
  Serotype 21 at Year 1:S | 3.0
  Serotype 22F at Year 1:S: number analyzed (Participants) | 135
  Serotype 22F at Year 1:S | 1.5
  Serotype 23A at Year 1:S: number analyzed (Participants) | 135
  Serotype 23A at Year 1:S | 3.0
  Serotype 23B at Year 1:S: number analyzed (Participants) | 135
  Serotype 23B at Year 1:S | 0.7
  Serotype 31 at Year 1:S: number analyzed (Participants) | 135
  Serotype 31 at Year 1:S | 0.7
  Serotype 33A at Year 1:S: number analyzed (Participants) | 135
  Serotype 33A at Year 1:S | 0.0
  Serotype 33F at Year 1:S: number analyzed (Participants) | 135
  Serotype 33F at Year 1:S | 0.7
  Serotype 34 at Year 1:S: number analyzed (Participants) | 135
  Serotype 34 at Year 1:S | 0.0
  Serotype 35B at Year 1:S: number analyzed (Participants) | 135
  Serotype 35B at Year 1:S | 2.2
  Serotype 35F at Year 1:S: number analyzed (Participants) | 135
  Serotype 35F at Year 1:S | 0.0
  Serotype 38 at Year 1:S: number analyzed (Participants) | 135
  Serotype 38 at Year 1:S | 0.7
  Serotype clumps at Year 1:S: number analyzed (Participants) | 135
  Serotype clumps at Year 1:S | 0.7
  Serotype Missing/non-viable at Year 1:S: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:S | 0.7
  Serotype 3 at Year 2:S: number analyzed (Participants) | 111
  Serotype 3 at Year 2:S | 5.4
  Serotype 6C at Year 2:S: number analyzed (Participants) | 111
  Serotype 6C at Year 2:S | 2.7
  Serotype 7C at Year 2:S: number analyzed (Participants) | 111
  Serotype 7C at Year 2:S | 0.0
  Serotype 9N at Year 2:S: number analyzed (Participants) | 111
  Serotype 9N at Year 2:S | 0.0
  Serotype 10 at Year 2:S: number analyzed (Participants) | 111
  Serotype 10 at Year 2:S | 0.0
  Serotype 11 at Year 2:S: number analyzed (Participants) | 111
  Serotype 11 at Year 2:S | 3.6
  Serotype 12 at Year 2:S: number analyzed (Participants) | 111
  Serotype 12 at Year 2:S | 0.0
  Serotype 12F at Year 2:S: number analyzed (Participants) | 111
  Serotype 12F at Year 2:S | 0.9
  Serotype 13 at Year 2:S: number analyzed (Participants) | 111
  Serotype 13 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 111
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 111
  Serotype 15B at Year 2:S | 1.8
  Serotype 15C at Year 2:S: number analyzed (Participants) | 111
  Serotype 15C at Year 2:S | 0.9
  Serotype 15F at Year 2:S: number analyzed (Participants) | 111
  Serotype 15F at Year 2:S | 0.0
  Serotype 16 at Year 2:S: number analyzed (Participants) | 111
  Serotype 16 at Year 2:S | 2.7
  Serotype 17 at Year 2:S: number analyzed (Participants) | 111
  Serotype 17 at Year 2:S | 1.8
  Serotype 19A at Year 2:S: number analyzed (Participants) | 111
  Serotype 19A at Year 2:S | 3.6
  Serotype 19F at Year 2:S: number analyzed (Participants) | 111
  Serotype 19F at Year 2:S | 0.9
  Serotype 20 at Year 2:S: number analyzed (Participants) | 111
  Serotype 20 at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 111
  Serotype 21 at Year 2:S | 9.0
  Serotype 22F at Year 2:S: number analyzed (Participants) | 111
  Serotype 22F at Year 2:S | 0.9
  Serotype 23A at Year 2:S: number analyzed (Participants) | 111
  Serotype 23A at Year 2:S | 3.6
  Serotype 23B at Year 2:S: number analyzed (Participants) | 111
  Serotype 23B at Year 2:S | 5.4
  Serotype 31 at Year 2:S: number analyzed (Participants) | 111
  Serotype 31 at Year 2:S | 1.8
  Serotype 33A at Year 2:S: number analyzed (Participants) | 111
  Serotype 33A at Year 2:S | 0.0
  Serotype 33F at Year 2:S: number analyzed (Participants) | 111
  Serotype 33F at Year 2:S | 0.0
  Serotype 34 at Year 2:S: number analyzed (Participants) | 111
  Serotype 34 at Year 2:S | 0.9
  Serotype 35B at Year 2:S: number analyzed (Participants) | 111
  Serotype 35B at Year 2:S | 3.6
  Serotype 35F at Year 2:S: number analyzed (Participants) | 111
  Serotype 35F at Year 2:S | 0.9
  Serotype 38 at Year 2:S: number analyzed (Participants) | 111
  Serotype 38 at Year 2:S | 0.9
  Serotype clumps at Year 2:S: number analyzed (Participants) | 111
  Serotype clumps at Year 2:S | 0.9
  Serotype Missing/non-viable at Year 2:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:S | 0.9
  Serotype 3 at Year 3:S: number analyzed (Participants) | 111
  Serotype 3 at Year 3:S | 5.4
  Serotype 6C at Year 3:S: number analyzed (Participants) | 111
  Serotype 6C at Year 3:S | 1.8
  Serotype 7C at Year 3:S: number analyzed (Participants) | 111
  Serotype 7C at Year 3:S | 0.0
  Serotype 9N at Year 3:S: number analyzed (Participants) | 111
  Serotype 9N at Year 3:S | 0.9
  Serotype 10 at Year 3:S: number analyzed (Participants) | 111
  Serotype 10 at Year 3:S | 2.7
  Serotype 11 at Year 3:S: number analyzed (Participants) | 111
  Serotype 11 at Year 3:S | 0.9
  Serotype 12 at Year 3:S: number analyzed (Participants) | 111
  Serotype 12 at Year 3:S | 0.0
  Serotype 12F at Year 3:S: number analyzed (Participants) | 111
  Serotype 12F at Year 3:S | 0.0
  Serotype 13 at Year 3:S: number analyzed (Participants) | 111
  Serotype 13 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 111
  Serotype 15A at Year 3:S | 2.7
  Serotype 15B at Year 3:S: number analyzed (Participants) | 111
  Serotype 15B at Year 3:S | 1.8
  Serotype 15C at Year 3:S: number analyzed (Participants) | 111
  Serotype 15C at Year 3:S | 3.6
  Serotype 15F at Year 3:S: number analyzed (Participants) | 111
  Serotype 15F at Year 3:S | 0.0
  Serotype 16 at Year 3:S: number analyzed (Participants) | 111
  Serotype 16 at Year 3:S | 3.6
  Serotype 17 at Year 3:S: number analyzed (Participants) | 111
  Serotype 17 at Year 3:S | 0.9
  Serotype 19A at Year 3:S: number analyzed (Participants) | 111
  Serotype 19A at Year 3:S | 0.9
  Serotype 19F at Year 3:S: number analyzed (Participants) | 111
  Serotype 19F at Year 3:S | 2.7
  Serotype 20 at Year 3:S: number analyzed (Participants) | 111
  Serotype 20 at Year 3:S | 0.9
  Serotype 21 at Year 3:S: number analyzed (Participants) | 111
  Serotype 21 at Year 3:S | 4.5
  Serotype 22F at Year 3:S: number analyzed (Participants) | 111
  Serotype 22F at Year 3:S | 1.8
  Serotype 23A at Year 3:S: number analyzed (Participants) | 111
  Serotype 23A at Year 3:S | 2.7
  Serotype 23B at Year 3:S: number analyzed (Participants) | 111
  Serotype 23B at Year 3:S | 3.6
  Serotype 31 at Year 3:S: number analyzed (Participants) | 111
  Serotype 31 at Year 3:S | 4.5
  Serotype 33A at Year 3:S: number analyzed (Participants) | 111
  Serotype 33A at Year 3:S | 0.0
  Serotype 33F at Year 3:S: number analyzed (Participants) | 111
  Serotype 33F at Year 3:S | 0.0
  Serotype 34 at Year 3:S: number analyzed (Participants) | 111
  Serotype 34 at Year 3:S | 0.9
  Serotype 35B at Year 3:S: number analyzed (Participants) | 111
  Serotype 35B at Year 3:S | 2.7
  Serotype 35F at Year 3:S: number analyzed (Participants) | 111
  Serotype 35F at Year 3:S | 0.9
  Serotype 38 at Year 3:S: number analyzed (Participants) | 111
  Serotype 38 at Year 3:S | 0.9
  Serotype clumps at Year 3:S: number analyzed (Participants) | 111
  Serotype clumps at Year 3:S | 0.0
  Serotype Missing/non-viable at Year 3:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:S | 0.9
  Serotype 3 at Year 1:I: number analyzed (Participants) | 135
  Serotype 3 at Year 1:I | 0.0
  Serotype 6C at Year 1:I: number analyzed (Participants) | 135
  Serotype 6C at Year 1:I | 0.0
  Serotype 7C at Year 1:I: number analyzed (Participants) | 135
  Serotype 7C at Year 1:I | 0.0
  Serotype 9N at Year 1:I: number analyzed (Participants) | 135
  Serotype 9N at Year 1:I | 0.0
  Serotype 10 at Year 1:I: number analyzed (Participants) | 135
  Serotype 10 at Year 1:I | 0.0
  Serotype 11 at Year 1:I: number analyzed (Participants) | 135
  Serotype 11 at Year 1:I | 0.7
  Serotype 12 at Year 1:I: number analyzed (Participants) | 135
  Serotype 12 at Year 1:I | 0.0
  Serotype 12F at Year 1:I: number analyzed (Participants) | 135
  Serotype 12F at Year 1:I | 0.0
  Serotype 13 at Year 1:I: number analyzed (Participants) | 135
  Serotype 13 at Year 1:I | 0.7
  Serotype 15A at Year 1:I: number analyzed (Participants) | 135
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 135
  Serotype 15B at Year 1:I | 0.0
  Serotype 15C at Year 1:I: number analyzed (Participants) | 135
  Serotype 15C at Year 1:I | 0.7
  Serotype 15F at Year 1:I: number analyzed (Participants) | 135
  Serotype 15F at Year 1:I | 0.0
  Serotype 16 at Year 1:I: number analyzed (Participants) | 135
  Serotype 16 at Year 1:I | 0.0
  Serotype 17 at Year 1:I: number analyzed (Participants) | 135
  Serotype 17 at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 135
  Serotype 19A at Year 1:I | 14.1
  Serotype 19F at Year 1:I: number analyzed (Participants) | 135
  Serotype 19F at Year 1:I | 0.7
  Serotype 20 at Year 1:I: number analyzed (Participants) | 135
  Serotype 20 at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 135
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 135
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 135
  Serotype 23A at Year 1:I | 0.0
  Serotype 23B at Year 1:I: number analyzed (Participants) | 135
  Serotype 23B at Year 1:I | 0.0
  Serotype 31 at Year 1:I: number analyzed (Participants) | 135
  Serotype 31 at Year 1:I | 0.7
  Serotype 33A at Year 1:I: number analyzed (Participants) | 135
  Serotype 33A at Year 1:I | 0.0
  Serotype 33F at Year 1:I: number analyzed (Participants) | 135
  Serotype 33F at Year 1:I | 0.0
  Serotype 34 at Year 1:I: number analyzed (Participants) | 135
  Serotype 34 at Year 1:I | 0.0
  Serotype 35B at Year 1:I: number analyzed (Participants) | 135
  Serotype 35B at Year 1:I | 0.0
  Serotype 35F at Year 1:I: number analyzed (Participants) | 135
  Serotype 35F at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 135
  Serotype 38 at Year 1:I | 0.0
  Serotype clumps at Year 1:I: number analyzed (Participants) | 135
  Serotype clumps at Year 1:I | 0.0
  Serotype Missing/non-viable at Year 1:I: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 111
  Serotype 3 at Year 2:I | 0.9
  Serotype 6C at Year 2:I: number analyzed (Participants) | 111
  Serotype 6C at Year 2:I | 0.0
  Serotype 7C at Year 2:I: number analyzed (Participants) | 111
  Serotype 7C at Year 2:I | 0.0
  Serotype 9N at Year 2:I: number analyzed (Participants) | 111
  Serotype 9N at Year 2:I | 0.0
  Serotype 10 at Year 2:I: number analyzed (Participants) | 111
  Serotype 10 at Year 2:I | 0.0
  Serotype 11 at Year 2:I: number analyzed (Participants) | 111
  Serotype 11 at Year 2:I | 0.9
  Serotype 12 at Year 2:I: number analyzed (Participants) | 111
  Serotype 12 at Year 2:I | 0.0
  Serotype 12F at Year 2:I: number analyzed (Participants) | 111
  Serotype 12F at Year 2:I | 0.0
  Serotype 13 at Year 2:I: number analyzed (Participants) | 111
  Serotype 13 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 111
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 111
  Serotype 15B at Year 2:I | 2.7
  Serotype 15C at Year 2:I: number analyzed (Participants) | 111
  Serotype 15C at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 111
  Serotype 15F at Year 2:I | 0.0
  Serotype 16 at Year 2:I: number analyzed (Participants) | 111
  Serotype 16 at Year 2:I | 0.0
  Serotype 17 at Year 2:I: number analyzed (Participants) | 111
  Serotype 17 at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 111
  Serotype 19A at Year 2:I | 12.6
  Serotype 19F at Year 2:I: number analyzed (Participants) | 111
  Serotype 19F at Year 2:I | 0.0
  Serotype 20 at Year 2:I: number analyzed (Participants) | 111
  Serotype 20 at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 111
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 111
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 111
  Serotype 23A at Year 2:I | 0.0
  Serotype 23B at Year 2:I: number analyzed (Participants) | 111
  Serotype 23B at Year 2:I | 0.9
  Serotype 31 at Year 2:I: number analyzed (Participants) | 111
  Serotype 31 at Year 2:I | 0.0
  Serotype 33A at Year 2:I: number analyzed (Participants) | 111
  Serotype 33A at Year 2:I | 0.0
  Serotype 33F at Year 2:I: number analyzed (Participants) | 111
  Serotype 33F at Year 2:I | 0.0
  Serotype 34 at Year 2:I: number analyzed (Participants) | 111
  Serotype 34 at Year 2:I | 0.0
  Serotype 35B at Year 2:I: number analyzed (Participants) | 111
  Serotype 35B at Year 2:I | 0.9
  Serotype 35F at Year 2:I: number analyzed (Participants) | 111
  Serotype 35F at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 111
  Serotype 38 at Year 2:I | 0.0
  Serotype clumps at Year 2:I: number analyzed (Participants) | 111
  Serotype clumps at Year 2:I | 0.0
  Serotype Missing/non-viable at Year 2:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 111
  Serotype 3 at Year 3:I | 1.8
  Serotype 6C at Year 3:I: number analyzed (Participants) | 111
  Serotype 6C at Year 3:I | 0.0
  Serotype 7C at Year 3:I: number analyzed (Participants) | 111
  Serotype 7C at Year 3:I | 0.0
  Serotype 9N at Year 3:I: number analyzed (Participants) | 111
  Serotype 9N at Year 3:I | 0.0
  Serotype 10 at Year 3:I: number analyzed (Participants) | 111
  Serotype 10 at Year 3:I | 0.0
  Serotype 11 at Year 3:I: number analyzed (Participants) | 111
  Serotype 11 at Year 3:I | 0.9
  Serotype 12 at Year 3:I: number analyzed (Participants) | 111
  Serotype 12 at Year 3:I | 0.0
  Serotype 12F at Year 3:I: number analyzed (Participants) | 111
  Serotype 12F at Year 3:I | 0.0
  Serotype 13 at Year 3:I: number analyzed (Participants) | 111
  Serotype 13 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 111
  Serotype 15A at Year 3:I | 2.7
  Serotype 15B at Year 3:I: number analyzed (Participants) | 111
  Serotype 15B at Year 3:I | 0.9
  Serotype 15C at Year 3:I: number analyzed (Participants) | 111
  Serotype 15C at Year 3:I | 0.9
  Serotype 15F at Year 3:I: number analyzed (Participants) | 111
  Serotype 15F at Year 3:I | 0.9
  Serotype 16 at Year 3:I: number analyzed (Participants) | 111
  Serotype 16 at Year 3:I | 0.0
  Serotype 17 at Year 3:I: number analyzed (Participants) | 111
  Serotype 17 at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 111
  Serotype 19A at Year 3:I | 2.7
  Serotype 19F at Year 3:I: number analyzed (Participants) | 111
  Serotype 19F at Year 3:I | 1.8
  Serotype 20 at Year 3:I: number analyzed (Participants) | 111
  Serotype 20 at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 111
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 111
  Serotype 22F at Year 3:I | 0.9
  Serotype 23A at Year 3:I: number analyzed (Participants) | 111
  Serotype 23A at Year 3:I | 0.0
  Serotype 23B at Year 3:I: number analyzed (Participants) | 111
  Serotype 23B at Year 3:I | 1.8
  Serotype 31 at Year 3:I: number analyzed (Participants) | 111
  Serotype 31 at Year 3:I | 0.0
  Serotype 33A at Year 3:I: number analyzed (Participants) | 111
  Serotype 33A at Year 3:I | 0.0
  Serotype 33F at Year 3:I: number analyzed (Participants) | 111
  Serotype 33F at Year 3:I | 0.0
  Serotype 34 at Year 3:I: number analyzed (Participants) | 111
  Serotype 34 at Year 3:I | 0.0
  Serotype 35B at Year 3:I: number analyzed (Participants) | 111
  Serotype 35B at Year 3:I | 2.7
  Serotype 35F at Year 3:I: number analyzed (Participants) | 111
  Serotype 35F at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 111
  Serotype 38 at Year 3:I | 0.0
  Serotype clumps at Year 3:I: number analyzed (Participants) | 111
  Serotype clumps at Year 3:I | 0.0
  Serotype Missing/non-viable at Year 3:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 135
  Serotype 3 at Year 1:R | 0.0
  Serotype 6C at Year 1:R: number analyzed (Participants) | 135
  Serotype 6C at Year 1:R | 2.2
  Serotype 7C at Year 1:R: number analyzed (Participants) | 135
  Serotype 7C at Year 1:R | 0.0
  Serotype 9N at Year 1:R: number analyzed (Participants) | 135
  Serotype 9N at Year 1:R | 0.0
  Serotype 10 at Year 1:R: number analyzed (Participants) | 135
  Serotype 10 at Year 1:R | 0.0
  Serotype 11 at Year 1:R: number analyzed (Participants) | 135
  Serotype 11 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 135
  Serotype 12 at Year 1:R | 0.0
  Serotype 12F at Year 1:R: number analyzed (Participants) | 135
  Serotype 12F at Year 1:R | 0.0
  Serotype 13 at Year 1:R: number analyzed (Participants) | 135
  Serotype 13 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 135
  Serotype 15A at Year 1:R | 1.5
  Serotype 15B at Year 1:R: number analyzed (Participants) | 135
  Serotype 15B at Year 1:R | 0.7
  Serotype 15C at Year 1:R: number analyzed (Participants) | 135
  Serotype 15C at Year 1:R | 1.5
  Serotype 15F at Year 1:R: number analyzed (Participants) | 135
  Serotype 15F at Year 1:R | 0.0
  Serotype 16 at Year 1:R: number analyzed (Participants) | 135
  Serotype 16 at Year 1:R | 0.0
  Serotype 17 at Year 1:R: number analyzed (Participants) | 135
  Serotype 17 at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 135
  Serotype 19A at Year 1:R | 14.8
  Serotype 19F at Year 1:R: number analyzed (Participants) | 135
  Serotype 19F at Year 1:R | 0.7
  Serotype 20 at Year 1:R: number analyzed (Participants) | 135
  Serotype 20 at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 135
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 135
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 135
  Serotype 23A at Year 1:R | 0.0
  Serotype 23B at Year 1:R: number analyzed (Participants) | 135
  Serotype 23B at Year 1:R | 0.0
  Serotype 31 at Year 1:R: number analyzed (Participants) | 135
  Serotype 31 at Year 1:R | 0.7
  Serotype 33A at Year 1:R: number analyzed (Participants) | 135
  Serotype 33A at Year 1:R | 0.7
  Serotype 33F at Year 1:R: number analyzed (Participants) | 135
  Serotype 33F at Year 1:R | 2.2
  Serotype 34 at Year 1:R: number analyzed (Participants) | 135
  Serotype 34 at Year 1:R | 0.0
  Serotype 35B at Year 1:R: number analyzed (Participants) | 135
  Serotype 35B at Year 1:R | 4.4
  Serotype 35F at Year 1:R: number analyzed (Participants) | 135
  Serotype 35F at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 135
  Serotype 38 at Year 1:R | 0.0
  Serotype clumps at Year 1:R: number analyzed (Participants) | 135
  Serotype clumps at Year 1:R | 0.0
  Serotype Missing/non-viable at Year 1:R: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 111
  Serotype 3 at Year 2:R | 0.0
  Serotype 6C at Year 2:R: number analyzed (Participants) | 111
  Serotype 6C at Year 2:R | 0.9
  Serotype 7C at Year 2:R: number analyzed (Participants) | 111
  Serotype 7C at Year 2:R | 0.0
  Serotype 9N at Year 2:R: number analyzed (Participants) | 111
  Serotype 9N at Year 2:R | 0.0
  Serotype 10 at Year 2:R: number analyzed (Participants) | 111
  Serotype 10 at Year 2:R | 0.9
  Serotype 11 at Year 2:R: number analyzed (Participants) | 111
  Serotype 11 at Year 2:R | 2.7
  Serotype 12 at Year 2:R: number analyzed (Participants) | 111
  Serotype 12 at Year 2:R | 0.0
  Serotype 12F at Year 2:R: number analyzed (Participants) | 111
  Serotype 12F at Year 2:R | 0.0
  Serotype 13 at Year 2:R: number analyzed (Participants) | 111
  Serotype 13 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 111
  Serotype 15A at Year 2:R | 0.9
  Serotype 15B at Year 2:R: number analyzed (Participants) | 111
  Serotype 15B at Year 2:R | 0.0
  Serotype 15C at Year 2:R: number analyzed (Participants) | 111
  Serotype 15C at Year 2:R | 1.8
  Serotype 15F at Year 2:R: number analyzed (Participants) | 111
  Serotype 15F at Year 2:R | 0.0
  Serotype 16 at Year 2:R: number analyzed (Participants) | 111
  Serotype 16 at Year 2:R | 0.0
  Serotype 17 at Year 2:R: number analyzed (Participants) | 111
  Serotype 17 at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 111
  Serotype 19A at Year 2:R | 6.3
  Serotype 19F at Year 2:R: number analyzed (Participants) | 111
  Serotype 19F at Year 2:R | 0.0
  Serotype 20 at Year 2:R: number analyzed (Participants) | 111
  Serotype 20 at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 111
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 111
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 111
  Serotype 23A at Year 2:R | 0.9
  Serotype 23B at Year 2:R: number analyzed (Participants) | 111
  Serotype 23B at Year 2:R | 0.9
  Serotype 31 at Year 2:R: number analyzed (Participants) | 111
  Serotype 31 at Year 2:R | 0.0
  Serotype 33A at Year 2:R: number analyzed (Participants) | 111
  Serotype 33A at Year 2:R | 0.0
  Serotype 33F at Year 2:R: number analyzed (Participants) | 111
  Serotype 33F at Year 2:R | 0.0
  Serotype 34 at Year 2:R: number analyzed (Participants) | 111
  Serotype 34 at Year 2:R | 0.0
  Serotype 35B at Year 2:R: number analyzed (Participants) | 111
  Serotype 35B at Year 2:R | 9.0
  Serotype 35F at Year 2:R: number analyzed (Participants) | 111
  Serotype 35F at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 111
  Serotype 38 at Year 2:R | 0.0
  Serotype clumps at Year 2:R: number analyzed (Participants) | 111
  Serotype clumps at Year 2:R | 0.0
  Serotype Missing/non-viable at Year 2:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 111
  Serotype 3 at Year 3:R | 0.0
  Serotype 6C at Year 3:R: number analyzed (Participants) | 111
  Serotype 6C at Year 3:R | 0.0
  Serotype 7C at Year 3:R: number analyzed (Participants) | 111
  Serotype 7C at Year 3:R | 0.0
  Serotype 9N at Year 3:R: number analyzed (Participants) | 111
  Serotype 9N at Year 3:R | 0.0
  Serotype 10 at Year 3:R: number analyzed (Participants) | 111
  Serotype 10 at Year 3:R | 0.0
  Serotype 11 at Year 3:R: number analyzed (Participants) | 111
  Serotype 11 at Year 3:R | 1.8
  Serotype 12 at Year 3:R: number analyzed (Participants) | 111
  Serotype 12 at Year 3:R | 0.0
  Serotype 12F at Year 3:R: number analyzed (Participants) | 111
  Serotype 12F at Year 3:R | 0.0
  Serotype 13 at Year 3:R: number analyzed (Participants) | 111
  Serotype 13 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 111
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 111
  Serotype 15B at Year 3:R | 1.8
  Serotype 15C at Year 3:R: number analyzed (Participants) | 111
  Serotype 15C at Year 3:R | 0.9
  Serotype 15F at Year 3:R: number analyzed (Participants) | 111
  Serotype 15F at Year 3:R | 0.0
  Serotype 16 at Year 3:R: number analyzed (Participants) | 111
  Serotype 16 at Year 3:R | 0.9
  Serotype 17 at Year 3:R: number analyzed (Participants) | 111
  Serotype 17 at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 111
  Serotype 19A at Year 3:R | 6.3
  Serotype 19F at Year 3:R: number analyzed (Participants) | 111
  Serotype 19F at Year 3:R | 0.9
  Serotype 20 at Year 3:R: number analyzed (Participants) | 111
  Serotype 20 at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 111
  Serotype 21 at Year 3:R | 0.9
  Serotype 22F at Year 3:R: number analyzed (Participants) | 111
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 111
  Serotype 23A at Year 3:R | 0.0
  Serotype 23B at Year 3:R: number analyzed (Participants) | 111
  Serotype 23B at Year 3:R | 2.7
  Serotype 31 at Year 3:R: number analyzed (Participants) | 111
  Serotype 31 at Year 3:R | 0.0
  Serotype 33A at Year 3:R: number analyzed (Participants) | 111
  Serotype 33A at Year 3:R | 0.0
  Serotype 33F at Year 3:R: number analyzed (Participants) | 111
  Serotype 33F at Year 3:R | 1.8
  Serotype 34 at Year 3:R: number analyzed (Participants) | 111
  Serotype 34 at Year 3:R | 0.0
  Serotype 35B at Year 3:R: number analyzed (Participants) | 111
  Serotype 35B at Year 3:R | 5.4
  Serotype 35F at Year 3:R: number analyzed (Participants) | 111
  Serotype 35F at Year 3:R | 0.9
  Serotype 38 at Year 3:R: number analyzed (Participants) | 111
  Serotype 38 at Year 3:R | 0.0
  Serotype clumps at Year 3:R: number analyzed (Participants) | 111
  Serotype clumps at Year 3:R | 0.0
  Serotype Missing/non-viable at Year 3:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:R | 0.9

12. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Penicillin: Middle Ear Fluid (MEF) Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for penicillin from MEF samples were summarized by providing the range of MICs for penicillin tested and the percentage of the susceptibility interpretation was categorized as resistant, susceptible or intermediate for each serotype, and for each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 19 A, 19 F, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38, clumps and missing or non-viable, which were to be computed along with exact 2-sided 95 % CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: MEF population included all participants who have at least 1 S pneumoniae isolate from MEF samples, however, actual 'N' for this OM is unknown as these data were not calculated as per planned analysis. number analyzed=number of isolates for the given serotype at specified time point.
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 135
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 135
  Serotype 3 at Year 1:S | 5.2
  Serotype 7C at Year 1:S: number analyzed (Participants) | 135
  Serotype 7C at Year 1:S | 1.5
  Serotype 9N at Year 1:S: number analyzed (Participants) | 135
  Serotype 9N at Year 1:S | 2.2
  Serotype 10 at Year 1:S: number analyzed (Participants) | 135
  Serotype 10 at Year 1:S | 3.0
  Serotype 11 at Year 1:S: number analyzed (Participants) | 135
  Serotype 11 at Year 1:S | 3.7
  Serotype 12 at Year 1:S: number analyzed (Participants) | 135
  Serotype 12 at Year 1:S | 0.0
  Serotype 12F at Year 1:S: number analyzed (Participants) | 135
  Serotype 12F at Year 1:S | 0.0
  Serotype 13 at Year 1:S: number analyzed (Participants) | 135
  Serotype 13 at Year 1:S | 0.0
  Serotype 15A at Year 1:S: number analyzed (Participants) | 135
  Serotype 15A at Year 1:S | 0.7
  Serotype 15B at Year 1:S: number analyzed (Participants) | 135
  Serotype 15B at Year 1:S | 3.7
  Serotype 15C at Year 1:S: number analyzed (Participants) | 135
  Serotype 15C at Year 1:S | 1.5
  Serotype 15F at Year 1:S: number analyzed (Participants) | 135
  Serotype 15F at Year 1:S | 0.0
  Serotype 16 at Year 1:S: number analyzed (Participants) | 135
  Serotype 16 at Year 1:S | 1.5
  Serotype 17 at Year 1:S: number analyzed (Participants) | 135
  Serotype 17 at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 135
  Serotype 19A at Year 1:S | 2.2
  Serotype 19F at Year 1:S: number analyzed (Participants) | 135
  Serotype 19F at Year 1:S | 0.7
  Serotype 20 at Year 1:S: number analyzed (Participants) | 135
  Serotype 20 at Year 1:S | 0.0
  Serotype 21 at Year 1:S: number analyzed (Participants) | 135
  Serotype 21 at Year 1:S | 3.0
  Serotype 22F at Year 1:S: number analyzed (Participants) | 135
  Serotype 22F at Year 1:S | 1.5
  Serotype 23A at Year 1:S: number analyzed (Participants) | 135
  Serotype 23A at Year 1:S | 0.0
  Serotype 23B at Year 1:S: number analyzed (Participants) | 135
  Serotype 23B at Year 1:S | 0.7
  Serotype 31 at Year 1:S: number analyzed (Participants) | 135
  Serotype 31 at Year 1:S | 2.2
  Serotype 33A at Year 1:S: number analyzed (Participants) | 135
  Serotype 33A at Year 1:S | 0.7
  Serotype 33F at Year 1:S: number analyzed (Participants) | 135
  Serotype 33F at Year 1:S | 1.5
  Serotype 34 at Year 1:S: number analyzed (Participants) | 135
  Serotype 34 at Year 1:S | 0.0
  Serotype 35B at Year 1:S: number analyzed (Participants) | 135
  Serotype 35B at Year 1:S | 0.0
  Serotype 35F at Year 1:S: number analyzed (Participants) | 135
  Serotype 35F at Year 1:S | 0.0
  Serotype 38 at Year 1:S: number analyzed (Participants) | 135
  Serotype 38 at Year 1:S | 0.7
  Serotype clumps at Year 1:S: number analyzed (Participants) | 135
  Serotype clumps at Year 1:S | 0.7
  Serotype Missing/non-viable at Year 1:S: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:S | 1.5
  Serotype 3 at Year 2:S: number analyzed (Participants) | 111
  Serotype 3 at Year 2:S | 6.3
  Serotype 6C at Year 2:S: number analyzed (Participants) | 111
  Serotype 6C at Year 2:S | 0.9
  Serotype 7C at Year 2:S: number analyzed (Participants) | 111
  Serotype 7C at Year 2:S | 0.0
  Serotype 9N at Year 2:S: number analyzed (Participants) | 111
  Serotype 9N at Year 2:S | 0.0
  Serotype 10 at Year 2:S: number analyzed (Participants) | 111
  Serotype 10 at Year 2:S | 0.9
  Serotype 11 at Year 2:S: number analyzed (Participants) | 111
  Serotype 11 at Year 2:S | 6.3
  Serotype 12 at Year 2:S: number analyzed (Participants) | 111
  Serotype 12 at Year 2:S | 0.0
  Serotype 12F at Year 2:S: number analyzed (Participants) | 111
  Serotype 12F at Year 2:S | 0.9
  Serotype 13 at Year 2:S: number analyzed (Participants) | 111
  Serotype 13 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 111
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 111
  Serotype 15B at Year 2:S | 1.8
  Serotype 15C at Year 2:S: number analyzed (Participants) | 111
  Serotype 15C at Year 2:S | 1.8
  Serotype 15F at Year 2:S: number analyzed (Participants) | 111
  Serotype 15F at Year 2:S | 0.0
  Serotype 16 at Year 2:S: number analyzed (Participants) | 111
  Serotype 16 at Year 2:S | 1.8
  Serotype 17 at Year 2:S: number analyzed (Participants) | 111
  Serotype 17 at Year 2:S | 0.9
  Serotype 19A at Year 2:S: number analyzed (Participants) | 111
  Serotype 19A at Year 2:S | 1.8
  Serotype 19F at Year 2:S: number analyzed (Participants) | 111
  Serotype 19F at Year 2:S | 0.9
  Serotype 20 at Year 2:S: number analyzed (Participants) | 111
  Serotype 20 at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 111
  Serotype 21 at Year 2:S | 8.1
  Serotype 22F at Year 2:S: number analyzed (Participants) | 111
  Serotype 22F at Year 2:S | 0.9
  Serotype 23A at Year 2:S: number analyzed (Participants) | 111
  Serotype 23A at Year 2:S | 0.0
  Serotype 23B at Year 2:S: number analyzed (Participants) | 111
  Serotype 23B at Year 2:S | 2.7
  Serotype 31 at Year 2:S: number analyzed (Participants) | 111
  Serotype 31 at Year 2:S | 1.8
  Serotype 33A at Year 2:S: number analyzed (Participants) | 111
  Serotype 33A at Year 2:S | 0.0
  Serotype 33F at Year 2:S: number analyzed (Participants) | 111
  Serotype 33F at Year 2:S | 0.0
  Serotype 34 at Year 2:S: number analyzed (Participants) | 111
  Serotype 34 at Year 2:S | 0.9
  Serotype 35B at Year 2:S: number analyzed (Participants) | 111
  Serotype 35B at Year 2:S | 0.9
  Serotype 35F at Year 2:S: number analyzed (Participants) | 111
  Serotype 35F at Year 2:S | 0.9
  Serotype 38 at Year 2:S: number analyzed (Participants) | 111
  Serotype 38 at Year 2:S | 0.9
  Serotype clumps at Year 2:S: number analyzed (Participants) | 111
  Serotype clumps at Year 2:S | 0.9
  Serotype Missing/non-viable at Year 2:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:S | 0.9
  Serotype 3 at Year 3:S: number analyzed (Participants) | 111
  Serotype 3 at Year 3:S | 6.3
  Serotype 6C at Year 3:S: number analyzed (Participants) | 111
  Serotype 6C at Year 3:S | 1.8
  Serotype 7C at Year 3:S: number analyzed (Participants) | 111
  Serotype 7C at Year 3:S | 0.0
  Serotype 9N at Year 3:S: number analyzed (Participants) | 111
  Serotype 9N at Year 3:S | 0.9
  Serotype 10 at Year 3:S: number analyzed (Participants) | 111
  Serotype 10 at Year 3:S | 2.7
  Serotype 11 at Year 3:S: number analyzed (Participants) | 111
  Serotype 11 at Year 3:S | 3.6
  Serotype 12 at Year 3:S: number analyzed (Participants) | 111
  Serotype 12 at Year 3:S | 0.0
  Serotype 12F at Year 3:S: number analyzed (Participants) | 111
  Serotype 12F at Year 3:S | 0.0
  Serotype 13 at Year 3:S: number analyzed (Participants) | 111
  Serotype 13 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 111
  Serotype 15A at Year 3:S | 3.6
  Serotype 15B at Year 3:S: number analyzed (Participants) | 111
  Serotype 15B at Year 3:S | 1.8
  Serotype 15C at Year 3:S: number analyzed (Participants) | 111
  Serotype 15C at Year 3:S | 2.7
  Serotype 15F at Year 3:S: number analyzed (Participants) | 111
  Serotype 15F at Year 3:S | 0.0
  Serotype 16 at Year 3:S: number analyzed (Participants) | 111
  Serotype 16 at Year 3:S | 4.5
  Serotype 17 at Year 3:S: number analyzed (Participants) | 111
  Serotype 17 at Year 3:S | 0.9
  Serotype 19A at Year 3:S: number analyzed (Participants) | 111
  Serotype 19A at Year 3:S | 0.9
  Serotype 19F at Year 3:S: number analyzed (Participants) | 111
  Serotype 19F at Year 3:S | 3.6
  Serotype 20 at Year 3:S: number analyzed (Participants) | 111
  Serotype 20 at Year 3:S | 0.9
  Serotype 21 at Year 3:S: number analyzed (Participants) | 111
  Serotype 21 at Year 3:S | 5.4
  Serotype 22F at Year 3:S: number analyzed (Participants) | 111
  Serotype 22F at Year 3:S | 2.7
  Serotype 23A at Year 3:S: number analyzed (Participants) | 111
  Serotype 23A at Year 3:S | 0.9
  Serotype 23B at Year 3:S: number analyzed (Participants) | 111
  Serotype 23B at Year 3:S | 6.3
  Serotype 31 at Year 3:S: number analyzed (Participants) | 111
  Serotype 31 at Year 3:S | 3.6
  Serotype 33A at Year 3:S: number analyzed (Participants) | 111
  Serotype 33A at Year 3:S | 0.0
  Serotype 33F at Year 3:S: number analyzed (Participants) | 111
  Serotype 33F at Year 3:S | 0.9
  Serotype 34 at Year 3:S: number analyzed (Participants) | 111
  Serotype 34 at Year 3:S | 0.9
  Serotype 35B at Year 3:S: number analyzed (Participants) | 111
  Serotype 35B at Year 3:S | 0.0
  Serotype 35F at Year 3:S: number analyzed (Participants) | 111
  Serotype 35F at Year 3:S | 0.0
  Serotype 38 at Year 3:S: number analyzed (Participants) | 111
  Serotype 38 at Year 3:S | 0.9
  Serotype clumps at Year 3:S: number analyzed (Participants) | 111
  Serotype clumps at Year 3:S | 0.0
  Serotype Missing/non-viable at Year 3:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:S | 0.0
  Serotype 6C at Year 1:S: number analyzed (Participants) | 135
  Serotype 6C at Year 1:S | 2.2
  Serotype 3 at Year 1:I: number analyzed (Participants) | 135
  Serotype 3 at Year 1:I | 0.7
  Serotype 6C at Year 1:I: number analyzed (Participants) | 135
  Serotype 6C at Year 1:I | 3.7
  Serotype 7C at Year 1:I: number analyzed (Participants) | 135
  Serotype 7C at Year 1:I | 0.0
  Serotype 9N at Year 1:I: number analyzed (Participants) | 135
  Serotype 9N at Year 1:I | 0.0
  Serotype 10 at Year 1:I: number analyzed (Participants) | 135
  Serotype 10 at Year 1:I | 0.0
  Serotype 11 at Year 1:I: number analyzed (Participants) | 135
  Serotype 11 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 135
  Serotype 12 at Year 1:I | 0.7
  Serotype 12F at Year 1:I: number analyzed (Participants) | 135
  Serotype 12F at Year 1:I | 0.0
  Serotype 13 at Year 1:I: number analyzed (Participants) | 135
  Serotype 13 at Year 1:I | 0.7
  Serotype 15A at Year 1:I: number analyzed (Participants) | 135
  Serotype 15A at Year 1:I | 3.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 135
  Serotype 15B at Year 1:I | 0.7
  Serotype 15C at Year 1:I: number analyzed (Participants) | 135
  Serotype 15C at Year 1:I | 2.2
  Serotype 15F at Year 1:I: number analyzed (Participants) | 135
  Serotype 15F at Year 1:I | 0.0
  Serotype 16 at Year 1:I: number analyzed (Participants) | 135
  Serotype 16 at Year 1:I | 0.0
  Serotype 17 at Year 1:I: number analyzed (Participants) | 135
  Serotype 17 at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 135
  Serotype 19A at Year 1:I | 2.2
  Serotype 19F at Year 1:I: number analyzed (Participants) | 135
  Serotype 19F at Year 1:I | 0.7
  Serotype 20 at Year 1:I: number analyzed (Participants) | 135
  Serotype 20 at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 135
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 135
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 135
  Serotype 23A at Year 1:I | 3.0
  Serotype 23B at Year 1:I: number analyzed (Participants) | 135
  Serotype 23B at Year 1:I | 0.7
  Serotype 31 at Year 1:I: number analyzed (Participants) | 135
  Serotype 31 at Year 1:I | 0.0
  Serotype 33A at Year 1:I: number analyzed (Participants) | 135
  Serotype 33A at Year 1:I | 0.0
  Serotype 33F at Year 1:I: number analyzed (Participants) | 135
  Serotype 33F at Year 1:I | 1.5
  Serotype 34 at Year 1:I: number analyzed (Participants) | 135
  Serotype 34 at Year 1:I | 0.0
  Serotype 35B at Year 1:I: number analyzed (Participants) | 135
  Serotype 35B at Year 1:I | 5.2
  Serotype 35F at Year 1:I: number analyzed (Participants) | 135
  Serotype 35F at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 135
  Serotype 38 at Year 1:I | 0.0
  Serotype clumps at Year 1:I: number analyzed (Participants) | 135
  Serotype clumps at Year 1:I | 0.0
  Serotype Missing/non-viable at Year 1:I: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 111
  Serotype 3 at Year 2:I | 0.0
  Serotype 6C at Year 2:I: number analyzed (Participants) | 111
  Serotype 6C at Year 2:I | 2.7
  Serotype 7C at Year 2:I: number analyzed (Participants) | 111
  Serotype 7C at Year 2:I | 0.0
  Serotype 9N at Year 2:I: number analyzed (Participants) | 111
  Serotype 9N at Year 2:I | 0.0
  Serotype 10 at Year 2:I: number analyzed (Participants) | 111
  Serotype 10 at Year 2:I | 0.0
  Serotype 11 at Year 2:I: number analyzed (Participants) | 111
  Serotype 11 at Year 2:I | 0.0
  Serotype 12 at Year 2:I: number analyzed (Participants) | 111
  Serotype 12 at Year 2:I | 0.0
  Serotype 12F at Year 2:I: number analyzed (Participants) | 111
  Serotype 12F at Year 2:I | 0.0
  Serotype 13 at Year 2:I: number analyzed (Participants) | 111
  Serotype 13 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 111
  Serotype 15A at Year 2:I | 0.9
  Serotype 15B at Year 2:I: number analyzed (Participants) | 111
  Serotype 15B at Year 2:I | 2.7
  Serotype 15C at Year 2:I: number analyzed (Participants) | 111
  Serotype 15C at Year 2:I | 0.9
  Serotype 15F at Year 2:I: number analyzed (Participants) | 111
  Serotype 15F at Year 2:I | 0.0
  Serotype 16 at Year 2:I: number analyzed (Participants) | 111
  Serotype 16 at Year 2:I | 0.9
  Serotype 17 at Year 2:I: number analyzed (Participants) | 111
  Serotype 17 at Year 2:I | 0.9
  Serotype 19A at Year 2:I: number analyzed (Participants) | 111
  Serotype 19A at Year 2:I | 1.8
  Serotype 19F at Year 2:I: number analyzed (Participants) | 111
  Serotype 19F at Year 2:I | 0.0
  Serotype 20 at Year 2:I: number analyzed (Participants) | 111
  Serotype 20 at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 111
  Serotype 21 at Year 2:I | 0.9
  Serotype 22F at Year 2:I: number analyzed (Participants) | 111
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 111
  Serotype 23A at Year 2:I | 4.5
  Serotype 23B at Year 2:I: number analyzed (Participants) | 111
  Serotype 23B at Year 2:I | 3.6
  Serotype 31 at Year 2:I: number analyzed (Participants) | 111
  Serotype 31 at Year 2:I | 0.0
  Serotype 33A at Year 2:I: number analyzed (Participants) | 111
  Serotype 33A at Year 2:I | 0.0
  Serotype 33F at Year 2:I: number analyzed (Participants) | 111
  Serotype 33F at Year 2:I | 0.0
  Serotype 34 at Year 2:I: number analyzed (Participants) | 111
  Serotype 34 at Year 2:I | 0.0
  Serotype 35B at Year 2:I: number analyzed (Participants) | 111
  Serotype 35B at Year 2:I | 9.9
  Serotype 35F at Year 2:I: number analyzed (Participants) | 111
  Serotype 35F at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 111
  Serotype 38 at Year 2:I | 0.0
  Serotype clumps at Year 2:I: number analyzed (Participants) | 111
  Serotype clumps at Year 2:I | 0.0
  Serotype Missing/non-viable at Year 2:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 111
  Serotype 3 at Year 3:I | 0.0
  Serotype 6C at Year 3:I: number analyzed (Participants) | 111
  Serotype 6C at Year 3:I | 0.0
  Serotype 7C at Year 3:I: number analyzed (Participants) | 111
  Serotype 7C at Year 3:I | 0.0
  Serotype 9N at Year 3:I: number analyzed (Participants) | 111
  Serotype 9N at Year 3:I | 0.0
  Serotype 10 at Year 3:I: number analyzed (Participants) | 111
  Serotype 10 at Year 3:I | 0.0
  Serotype 11 at Year 3:I: number analyzed (Participants) | 111
  Serotype 11 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 111
  Serotype 12 at Year 3:I | 0.0
  Serotype 12F at Year 3:I: number analyzed (Participants) | 111
  Serotype 12F at Year 3:I | 0.0
  Serotype 13 at Year 3:I: number analyzed (Participants) | 111
  Serotype 13 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 111
  Serotype 15A at Year 3:I | 1.8
  Serotype 15B at Year 3:I: number analyzed (Participants) | 111
  Serotype 15B at Year 3:I | 2.7
  Serotype 15C at Year 3:I: number analyzed (Participants) | 111
  Serotype 15C at Year 3:I | 2.7
  Serotype 15F at Year 3:I: number analyzed (Participants) | 111
  Serotype 15F at Year 3:I | 0.9
  Serotype 16 at Year 3:I: number analyzed (Participants) | 111
  Serotype 16 at Year 3:I | 0.0
  Serotype 17 at Year 3:I: number analyzed (Participants) | 111
  Serotype 17 at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 111
  Serotype 19A at Year 3:I | 0.0
  Serotype 19F at Year 3:I: number analyzed (Participants) | 111
  Serotype 19F at Year 3:I | 0.0
  Serotype 20 at Year 3:I: number analyzed (Participants) | 111
  Serotype 20 at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 111
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 111
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 111
  Serotype 23A at Year 3:I | 1.8
  Serotype 23B at Year 3:I: number analyzed (Participants) | 111
  Serotype 23B at Year 3:I | 1.8
  Serotype 31 at Year 3:I: number analyzed (Participants) | 111
  Serotype 31 at Year 3:I | 0.9
  Serotype 33A at Year 3:I: number analyzed (Participants) | 111
  Serotype 33A at Year 3:I | 0.0
  Serotype 33F at Year 3:I: number analyzed (Participants) | 111
  Serotype 33F at Year 3:I | 0.9
  Serotype 34 at Year 3:I: number analyzed (Participants) | 111
  Serotype 34 at Year 3:I | 0.0
  Serotype 35B at Year 3:I: number analyzed (Participants) | 111
  Serotype 35B at Year 3:I | 6.3
  Serotype 35F at Year 3:I: number analyzed (Participants) | 111
  Serotype 35F at Year 3:I | 0.9
  Serotype 38 at Year 3:I: number analyzed (Participants) | 111
  Serotype 38 at Year 3:I | 0.0
  Serotype clumps at Year 3:I: number analyzed (Participants) | 111
  Serotype clumps at Year 3:I | 0.0
  Serotype Missing/non-viable at Year 3:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:I | 1.8
  Serotype 3 at Year 1:R: number analyzed (Participants) | 135
  Serotype 3 at Year 1:R | 0.0
  Serotype 6C at Year 1:R: number analyzed (Participants) | 135
  Serotype 6C at Year 1:R | 0.7
  Serotype 7C at Year 1:R: number analyzed (Participants) | 135
  Serotype 7C at Year 1:R | 0.0
  Serotype 9N at Year 1:R: number analyzed (Participants) | 135
  Serotype 9N at Year 1:R | 0.0
  Serotype 10 at Year 1:R: number analyzed (Participants) | 135
  Serotype 10 at Year 1:R | 0.0
  Serotype 11 at Year 1:R: number analyzed (Participants) | 135
  Serotype 11 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 135
  Serotype 12 at Year 1:R | 0.0
  Serotype 12F at Year 1:R: number analyzed (Participants) | 135
  Serotype 12F at Year 1:R | 0.0
  Serotype 13 at Year 1:R: number analyzed (Participants) | 135
  Serotype 13 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 135
  Serotype 15A at Year 1:R | 0.0
  Serotype 15B at Year 1:R: number analyzed (Participants) | 135
  Serotype 15B at Year 1:R | 0.0
  Serotype 15C at Year 1:R: number analyzed (Participants) | 135
  Serotype 15C at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 135
  Serotype 15F at Year 1:R | 0.0
  Serotype 16 at Year 1:R: number analyzed (Participants) | 135
  Serotype 16 at Year 1:R | 0.0
  Serotype 17 at Year 1:R: number analyzed (Participants) | 135
  Serotype 17 at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 135
  Serotype 19A at Year 1:R | 25.9
  Serotype 19F at Year 1:R: number analyzed (Participants) | 135
  Serotype 19F at Year 1:R | 0.7
  Serotype 20 at Year 1:R: number analyzed (Participants) | 135
  Serotype 20 at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 135
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 135
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 135
  Serotype 23A at Year 1:R | 0.0
  Serotype 23B at Year 1:R: number analyzed (Participants) | 135
  Serotype 23B at Year 1:R | 0.0
  Serotype 31 at Year 1:R: number analyzed (Participants) | 135
  Serotype 31 at Year 1:R | 0.0
  Serotype 33A at Year 1:R: number analyzed (Participants) | 135
  Serotype 33A at Year 1:R | 0.0
  Serotype 33F at Year 1:R: number analyzed (Participants) | 135
  Serotype 33F at Year 1:R | 0.0
  Serotype 34 at Year 1:R: number analyzed (Participants) | 135
  Serotype 34 at Year 1:R | 0.0
  Serotype 35B at Year 1:R: number analyzed (Participants) | 135
  Serotype 35B at Year 1:R | 1.5
  Serotype 35F at Year 1:R: number analyzed (Participants) | 135
  Serotype 35F at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 135
  Serotype 38 at Year 1:R | 0.0
  Serotype clumps at Year 1:R: number analyzed (Participants) | 135
  Serotype clumps at Year 1:R | 0.7
  Serotype Missing/non-viable at Year 1:R: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 111
  Serotype 3 at Year 2:R | 0.0
  Serotype 6C at Year 2:R: number analyzed (Participants) | 111
  Serotype 6C at Year 2:R | 0.0
  Serotype 7C at Year 2:R: number analyzed (Participants) | 111
  Serotype 7C at Year 2:R | 0.0
  Serotype 9N at Year 2:R: number analyzed (Participants) | 111
  Serotype 9N at Year 2:R | 0.0
  Serotype 10 at Year 2:R: number analyzed (Participants) | 111
  Serotype 10 at Year 2:R | 0.0
  Serotype 11 at Year 2:R: number analyzed (Participants) | 111
  Serotype 11 at Year 2:R | 0.9
  Serotype 12 at Year 2:R: number analyzed (Participants) | 111
  Serotype 12 at Year 2:R | 0.0
  Serotype 12F at Year 2:R: number analyzed (Participants) | 111
  Serotype 12F at Year 2:R | 0.0
  Serotype 13 at Year 2:R: number analyzed (Participants) | 111
  Serotype 13 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 111
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 111
  Serotype 15B at Year 2:R | 0.0
  Serotype 15C at Year 2:R: number analyzed (Participants) | 111
  Serotype 15C at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 111
  Serotype 15F at Year 2:R | 0.0
  Serotype 16 at Year 2:R: number analyzed (Participants) | 111
  Serotype 16 at Year 2:R | 0.0
  Serotype 17 at Year 2:R: number analyzed (Participants) | 111
  Serotype 17 at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 111
  Serotype 19A at Year 2:R | 18.9
  Serotype 19F at Year 2:R: number analyzed (Participants) | 111
  Serotype 19F at Year 2:R | 0.0
  Serotype 20 at Year 2:R: number analyzed (Participants) | 111
  Serotype 20 at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 111
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 111
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 111
  Serotype 23A at Year 2:R | 0.0
  Serotype 23B at Year 2:R: number analyzed (Participants) | 111
  Serotype 23B at Year 2:R | 0.9
  Serotype 31 at Year 2:R: number analyzed (Participants) | 111
  Serotype 31 at Year 2:R | 0.0
  Serotype 33A at Year 2:R: number analyzed (Participants) | 111
  Serotype 33A at Year 2:R | 0.0
  Serotype 33F at Year 2:R: number analyzed (Participants) | 111
  Serotype 33F at Year 2:R | 0.0
  Serotype 34 at Year 2:R: number analyzed (Participants) | 111
  Serotype 34 at Year 2:R | 0.0
  Serotype 35B at Year 2:R: number analyzed (Participants) | 111
  Serotype 35B at Year 2:R | 1.8
  Serotype 35F at Year 2:R: number analyzed (Participants) | 111
  Serotype 35F at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 111
  Serotype 38 at Year 2:R | 0.0
  Serotype clumps at Year 2:R: number analyzed (Participants) | 111
  Serotype clumps at Year 2:R | 0.0
  Serotype Missing/non-viable at Year 2:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 111
  Serotype 3 at Year 3:R | 0.9
  Serotype 6C at Year 3:R: number analyzed (Participants) | 111
  Serotype 6C at Year 3:R | 0.0
  Serotype 7C at Year 3:R: number analyzed (Participants) | 111
  Serotype 7C at Year 3:R | 0.0
  Serotype 9N at Year 3:R: number analyzed (Participants) | 111
  Serotype 9N at Year 3:R | 0.0
  Serotype 10 at Year 3:R: number analyzed (Participants) | 111
  Serotype 10 at Year 3:R | 0.0
  Serotype 11 at Year 3:R: number analyzed (Participants) | 111
  Serotype 11 at Year 3:R | 0.0
  Serotype 12 at Year 3:R: number analyzed (Participants) | 111
  Serotype 12 at Year 3:R | 0.0
  Serotype 12F at Year 3:R: number analyzed (Participants) | 111
  Serotype 12F at Year 3:R | 0.0
  Serotype 13 at Year 3:R: number analyzed (Participants) | 111
  Serotype 13 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 111
  Serotype 15A at Year 3:R | 0.9
  Serotype 15B at Year 3:R: number analyzed (Participants) | 111
  Serotype 15B at Year 3:R | 0.0
  Serotype 15C at Year 3:R: number analyzed (Participants) | 111
  Serotype 15C at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 111
  Serotype 15F at Year 3:R | 0.0
  Serotype 16 at Year 3:R: number analyzed (Participants) | 111
  Serotype 16 at Year 3:R | 0.0
  Serotype 17 at Year 3:R: number analyzed (Participants) | 111
  Serotype 17 at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 111
  Serotype 19A at Year 3:R | 9.0
  Serotype 19F at Year 3:R: number analyzed (Participants) | 111
  Serotype 19F at Year 3:R | 1.8
  Serotype 20 at Year 3:R: number analyzed (Participants) | 111
  Serotype 20 at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 111
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 111
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 111
  Serotype 23A at Year 3:R | 0.0
  Serotype 23B at Year 3:R: number analyzed (Participants) | 111
  Serotype 23B at Year 3:R | 0.0
  Serotype 31 at Year 3:R: number analyzed (Participants) | 111
  Serotype 31 at Year 3:R | 0.0
  Serotype 33A at Year 3:R: number analyzed (Participants) | 111
  Serotype 33A at Year 3:R | 0.0
  Serotype 33F at Year 3:R: number analyzed (Participants) | 111
  Serotype 33F at Year 3:R | 0.0
  Serotype 34 at Year 3:R: number analyzed (Participants) | 111
  Serotype 34 at Year 3:R | 0.0
  Serotype 35B at Year 3:R: number analyzed (Participants) | 111
  Serotype 35B at Year 3:R | 2.7
  Serotype 35F at Year 3:R: number analyzed (Participants) | 111
  Serotype 35F at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 111
  Serotype 38 at Year 3:R | 0.0
  Serotype clumps at Year 3:R: number analyzed (Participants) | 111
  Serotype clumps at Year 3:R | 0.0
  Serotype Missing/non-viable at Year 3:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:R | 0.0

13. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Trimethoprim/Sulfamethoxazole (TMP/S): Middle Ear Fluid (MEF) Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for TMP/S from MEF samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 6C, 7C, 9N, 10, 11, 12, 12F, 13, 15A, 15B, 15C, 15F, 16, 17, 19A, 19F, 20, 21, 22F, 23A, 23B, 31, 33A, 33F, 34, 35B, 35F, 38, clumps and missing or non-viable, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. Missing or non-viable included isolates that were either not sent from an external laboratory, were non-viable or lost on culture prior to sending, or were non-viable on receipt in the central laboratory.'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: as for outcome 8
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | MEF Population
Number analyzed (Participants) | 357
Number analyzed (Isolates) | 135
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 135
  Serotype 3 at Year 1:S | 3.0
  Serotype 6C at Year 1:S: number analyzed (Participants) | 135
  Serotype 6C at Year 1:S | 0.7
  Serotype 7C at Year 1:S: number analyzed (Participants) | 135
  Serotype 7C at Year 1:S | 1.5
  Serotype 9N at Year 1:S: number analyzed (Participants) | 135
  Serotype 9N at Year 1:S | 1.5
  Serotype 10 at Year 1:S: number analyzed (Participants) | 135
  Serotype 10 at Year 1:S | 0.7
  Serotype 11 at Year 1:S: number analyzed (Participants) | 135
  Serotype 11 at Year 1:S | 2.2
  Serotype 12 at Year 1:S: number analyzed (Participants) | 135
  Serotype 12 at Year 1:S | 0.0
  Serotype 12F at Year 1:S: number analyzed (Participants) | 135
  Serotype 12F at Year 1:S | 0.0
  Serotype 13 at Year 1:S: number analyzed (Participants) | 135
  Serotype 13 at Year 1:S | 0.7
  Serotype 15A at Year 1:S: number analyzed (Participants) | 135
  Serotype 15A at Year 1:S | 0.0
  Serotype 15B at Year 1:S: number analyzed (Participants) | 135
  Serotype 15B at Year 1:S | 1.5
  Serotype 15C at Year 1:S: number analyzed (Participants) | 135
  Serotype 15C at Year 1:S | 0.0
  Serotype 15F at Year 1:S: number analyzed (Participants) | 135
  Serotype 15F at Year 1:S | 0.0
  Serotype 16 at Year 1:S: number analyzed (Participants) | 135
  Serotype 16 at Year 1:S | 1.5
  Serotype 17 at Year 1:S: number analyzed (Participants) | 135
  Serotype 17 at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 135
  Serotype 19A at Year 1:S | 0.7
  Serotype 19F at Year 1:S: number analyzed (Participants) | 135
  Serotype 19F at Year 1:S | 0.7
  Serotype 20 at Year 1:S: number analyzed (Participants) | 135
  Serotype 20 at Year 1:S | 0.0
  Serotype 21 at Year 1:S: number analyzed (Participants) | 135
  Serotype 21 at Year 1:S | 1.5
  Serotype 22F at Year 1:S: number analyzed (Participants) | 135
  Serotype 22F at Year 1:S | 0.7
  Serotype 23A at Year 1:S: number analyzed (Participants) | 135
  Serotype 23A at Year 1:S | 0.7
  Serotype 23B at Year 1:S: number analyzed (Participants) | 135
  Serotype 23B at Year 1:S | 0.0
  Serotype 31 at Year 1:S: number analyzed (Participants) | 135
  Serotype 31 at Year 1:S | 0.7
  Serotype 33A at Year 1:S: number analyzed (Participants) | 135
  Serotype 33A at Year 1:S | 0.0
  Serotype 33F at Year 1:S: number analyzed (Participants) | 135
  Serotype 33F at Year 1:S | 0.7
  Serotype 34 at Year 1:S: number analyzed (Participants) | 135
  Serotype 34 at Year 1:S | 0.0
  Serotype 35B at Year 1:S: number analyzed (Participants) | 135
  Serotype 35B at Year 1:S | 0.7
  Serotype 35F at Year 1:S: number analyzed (Participants) | 135
  Serotype 35F at Year 1:S | 0.0
  Serotype 38 at Year 1:S: number analyzed (Participants) | 135
  Serotype 38 at Year 1:S | 0.7
  Serotype clumps at Year 1:S: number analyzed (Participants) | 135
  Serotype clumps at Year 1:S | 0.7
  Serotype Missing/non-viable at Year 1:S: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:S | 0.7
  Serotype 3 at Year 2:S: number analyzed (Participants) | 111
  Serotype 3 at Year 2:S | 1.8
  Serotype 6C at Year 2:S: number analyzed (Participants) | 111
  Serotype 6C at Year 2:S | 0.9
  Serotype 7C at Year 2:S: number analyzed (Participants) | 111
  Serotype 7C at Year 2:S | 0.0
  Serotype 9N at Year 2:S: number analyzed (Participants) | 111
  Serotype 9N at Year 2:S | 0.0
  Serotype 10 at Year 2:S: number analyzed (Participants) | 111
  Serotype 10 at Year 2:S | 0.0
  Serotype 11 at Year 2:S: number analyzed (Participants) | 111
  Serotype 11 at Year 2:S | 3.6
  Serotype 12 at Year 2:S: number analyzed (Participants) | 111
  Serotype 12 at Year 2:S | 0.0
  Serotype 12F at Year 2:S: number analyzed (Participants) | 111
  Serotype 12F at Year 2:S | 0.0
  Serotype 13 at Year 2:S: number analyzed (Participants) | 111
  Serotype 13 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 111
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 111
  Serotype 15B at Year 2:S | 1.8
  Serotype 15C at Year 2:S: number analyzed (Participants) | 111
  Serotype 15C at Year 2:S | 0.0
  Serotype 15F at Year 2:S: number analyzed (Participants) | 111
  Serotype 15F at Year 2:S | 0.0
  Serotype 16 at Year 2:S: number analyzed (Participants) | 111
  Serotype 16 at Year 2:S | 0.9
  Serotype 17 at Year 2:S: number analyzed (Participants) | 111
  Serotype 17 at Year 2:S | 0.0
  Serotype 19A at Year 2:S: number analyzed (Participants) | 111
  Serotype 19A at Year 2:S | 1.8
  Serotype 19F at Year 2:S: number analyzed (Participants) | 111
  Serotype 19F at Year 2:S | 0.0
  Serotype 20 at Year 2:S: number analyzed (Participants) | 111
  Serotype 20 at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 111
  Serotype 21 at Year 2:S | 3.6
  Serotype 22F at Year 2:S: number analyzed (Participants) | 111
  Serotype 22F at Year 2:S | 0.9
  Serotype 23A at Year 2:S: number analyzed (Participants) | 111
  Serotype 23A at Year 2:S | 0.9
  Serotype 23B at Year 2:S: number analyzed (Participants) | 111
  Serotype 23B at Year 2:S | 0.9
  Serotype 31 at Year 2:S: number analyzed (Participants) | 111
  Serotype 31 at Year 2:S | 0.0
  Serotype 33A at Year 2:S: number analyzed (Participants) | 111
  Serotype 33A at Year 2:S | 0.0
  Serotype 33F at Year 2:S: number analyzed (Participants) | 111
  Serotype 33F at Year 2:S | 0.0
  Serotype 34 at Year 2:S: number analyzed (Participants) | 111
  Serotype 34 at Year 2:S | 0.0
  Serotype 35B at Year 2:S: number analyzed (Participants) | 111
  Serotype 35B at Year 2:S | 2.7
  Serotype 35F at Year 2:S: number analyzed (Participants) | 111
  Serotype 35F at Year 2:S | 0.0
  Serotype 38 at Year 2:S: number analyzed (Participants) | 111
  Serotype 38 at Year 2:S | 0.0
  Serotype clumps at Year 2:S: number analyzed (Participants) | 111
  Serotype clumps at Year 2:S | 0.9
  Serotype Missing/non-viable at Year 2:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:S | 0.0
  Serotype 3 at Year 3:S: number analyzed (Participants) | 111
  Serotype 3 at Year 3:S | 2.7
  Serotype 6C at Year 3:S: number analyzed (Participants) | 111
  Serotype 6C at Year 3:S | 1.8
  Serotype 7C at Year 3:S: number analyzed (Participants) | 111
  Serotype 7C at Year 3:S | 0.0
  Serotype 9N at Year 3:S: number analyzed (Participants) | 111
  Serotype 9N at Year 3:S | 0.0
  Serotype 10 at Year 3:S: number analyzed (Participants) | 111
  Serotype 10 at Year 3:S | 0.0
  Serotype 11 at Year 3:S: number analyzed (Participants) | 111
  Serotype 11 at Year 3:S | 0.9
  Serotype 12 at Year 3:S: number analyzed (Participants) | 111
  Serotype 12 at Year 3:S | 0.0
  Serotype 12F at Year 3:S: number analyzed (Participants) | 111
  Serotype 12F at Year 3:S | 0.0
  Serotype 13 at Year 3:S: number analyzed (Participants) | 111
  Serotype 13 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 111
  Serotype 15A at Year 3:S | 1.8
  Serotype 15B at Year 3:S: number analyzed (Participants) | 111
  Serotype 15B at Year 3:S | 0.0
  Serotype 15C at Year 3:S: number analyzed (Participants) | 111
  Serotype 15C at Year 3:S | 2.7
  Serotype 15F at Year 3:S: number analyzed (Participants) | 111
  Serotype 15F at Year 3:S | 0.0
  Serotype 16 at Year 3:S: number analyzed (Participants) | 111
  Serotype 16 at Year 3:S | 0.9
  Serotype 17 at Year 3:S: number analyzed (Participants) | 111
  Serotype 17 at Year 3:S | 0.0
  Serotype 19A at Year 3:S: number analyzed (Participants) | 111
  Serotype 19A at Year 3:S | 0.9
  Serotype 19F at Year 3:S: number analyzed (Participants) | 111
  Serotype 19F at Year 3:S | 0.9
  Serotype 20 at Year 3:S: number analyzed (Participants) | 111
  Serotype 20 at Year 3:S | 0.0
  Serotype 21 at Year 3:S: number analyzed (Participants) | 111
  Serotype 21 at Year 3:S | 3.6
  Serotype 22F at Year 3:S: number analyzed (Participants) | 111
  Serotype 22F at Year 3:S | 2.7
  Serotype 23A at Year 3:S: number analyzed (Participants) | 111
  Serotype 23A at Year 3:S | 0.0
  Serotype 23B at Year 3:S: number analyzed (Participants) | 111
  Serotype 23B at Year 3:S | 1.8
  Serotype 31 at Year 3:S: number analyzed (Participants) | 111
  Serotype 31 at Year 3:S | 1.8
  Serotype 33A at Year 3:S: number analyzed (Participants) | 111
  Serotype 33A at Year 3:S | 0.0
  Serotype 33F at Year 3:S: number analyzed (Participants) | 111
  Serotype 33F at Year 3:S | 0.0
  Serotype 34 at Year 3:S: number analyzed (Participants) | 111
  Serotype 34 at Year 3:S | 0.0
  Serotype 35B at Year 3:S: number analyzed (Participants) | 111
  Serotype 35B at Year 3:S | 0.9
  Serotype 35F at Year 3:S: number analyzed (Participants) | 111
  Serotype 35F at Year 3:S | 0.9
  Serotype 38 at Year 3:S: number analyzed (Participants) | 111
  Serotype 38 at Year 3:S | 0.0
  Serotype clumps at Year 3:S: number analyzed (Participants) | 111
  Serotype clumps at Year 3:S | 0.0
  Serotype Missing/non-viable at Year 3:S: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:S | 0.0
  Serotype 3 at Year 1:I: number analyzed (Participants) | 135
  Serotype 3 at Year 1:I | 0.0
  Serotype 6C at Year 1:I: number analyzed (Participants) | 135
  Serotype 6C at Year 1:I | 1.5
  Serotype 7C at Year 1:I: number analyzed (Participants) | 135
  Serotype 7C at Year 1:I | 0.0
  Serotype 9N at Year 1:I: number analyzed (Participants) | 135
  Serotype 9N at Year 1:I | 0.0
  Serotype 10 at Year 1:I: number analyzed (Participants) | 135
  Serotype 10 at Year 1:I | 0.0
  Serotype 11 at Year 1:I: number analyzed (Participants) | 135
  Serotype 11 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 135
  Serotype 12 at Year 1:I | 0.0
  Serotype 12F at Year 1:I: number analyzed (Participants) | 135
  Serotype 12F at Year 1:I | 0.0
  Serotype 13 at Year 1:I: number analyzed (Participants) | 135
  Serotype 13 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 135
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 135
  Serotype 15B at Year 1:I | 0.0
  Serotype 15C at Year 1:I: number analyzed (Participants) | 135
  Serotype 15C at Year 1:I | 0.7
  Serotype 15F at Year 1:I: number analyzed (Participants) | 135
  Serotype 15F at Year 1:I | 0.0
  Serotype 16 at Year 1:I: number analyzed (Participants) | 135
  Serotype 16 at Year 1:I | 0.0
  Serotype 17 at Year 1:I: number analyzed (Participants) | 135
  Serotype 17 at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 135
  Serotype 19A at Year 1:I | 14.1
  Serotype 19F at Year 1:I: number analyzed (Participants) | 135
  Serotype 19F at Year 1:I | 0.7
  Serotype 20 at Year 1:I: number analyzed (Participants) | 135
  Serotype 20 at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 135
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 135
  Serotype 22F at Year 1:I | 0.7
  Serotype 23A at Year 1:I: number analyzed (Participants) | 135
  Serotype 23A at Year 1:I | 0.0
  Serotype 23B at Year 1:I: number analyzed (Participants) | 135
  Serotype 23B at Year 1:I | 0.0
  Serotype 31 at Year 1:I: number analyzed (Participants) | 135
  Serotype 31 at Year 1:I | 0.0
  Serotype 33A at Year 1:I: number analyzed (Participants) | 135
  Serotype 33A at Year 1:I | 0.0
  Serotype 33F at Year 1:I: number analyzed (Participants) | 135
  Serotype 33F at Year 1:I | 0.0
  Serotype 34 at Year 1:I: number analyzed (Participants) | 135
  Serotype 34 at Year 1:I | 0.0
  Serotype 35B at Year 1:I: number analyzed (Participants) | 135
  Serotype 35B at Year 1:I | 0.0
  Serotype 35F at Year 1:I: number analyzed (Participants) | 135
  Serotype 35F at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 135
  Serotype 38 at Year 1:I | 0.0
  Serotype clumps at Year 1:I: number analyzed (Participants) | 135
  Serotype clumps at Year 1:I | 0.0
  Serotype Missing/non-viable at Year 1:I: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 111
  Serotype 3 at Year 2:I | 0.0
  Serotype 6C at Year 2:I: number analyzed (Participants) | 111
  Serotype 6C at Year 2:I | 0.0
  Serotype 7C at Year 2:I: number analyzed (Participants) | 111
  Serotype 7C at Year 2:I | 0.0
  Serotype 9N at Year 2:I: number analyzed (Participants) | 111
  Serotype 9N at Year 2:I | 0.0
  Serotype 10 at Year 2:I: number analyzed (Participants) | 111
  Serotype 10 at Year 2:I | 0.0
  Serotype 11 at Year 2:I: number analyzed (Participants) | 111
  Serotype 11 at Year 2:I | 0.9
  Serotype 12 at Year 2:I: number analyzed (Participants) | 111
  Serotype 12 at Year 2:I | 0.0
  Serotype 12F at Year 2:I: number analyzed (Participants) | 111
  Serotype 12F at Year 2:I | 0.0
  Serotype 13 at Year 2:I: number analyzed (Participants) | 111
  Serotype 13 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 111
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 111
  Serotype 15B at Year 2:I | 1.8
  Serotype 15C at Year 2:I: number analyzed (Participants) | 111
  Serotype 15C at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 111
  Serotype 15F at Year 2:I | 0.0
  Serotype 16 at Year 2:I: number analyzed (Participants) | 111
  Serotype 16 at Year 2:I | 0.0
  Serotype 17 at Year 2:I: number analyzed (Participants) | 111
  Serotype 17 at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 111
  Serotype 19A at Year 2:I | 12.6
  Serotype 19F at Year 2:I: number analyzed (Participants) | 111
  Serotype 19F at Year 2:I | 0.0
  Serotype 20 at Year 2:I: number analyzed (Participants) | 111
  Serotype 20 at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 111
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 111
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 111
  Serotype 23A at Year 2:I | 0.0
  Serotype 23B at Year 2:I: number analyzed (Participants) | 111
  Serotype 23B at Year 2:I | 0.9
  Serotype 31 at Year 2:I: number analyzed (Participants) | 111
  Serotype 31 at Year 2:I | 0.0
  Serotype 33A at Year 2:I: number analyzed (Participants) | 111
  Serotype 33A at Year 2:I | 0.0
  Serotype 33F at Year 2:I: number analyzed (Participants) | 111
  Serotype 33F at Year 2:I | 0.0
  Serotype 34 at Year 2:I: number analyzed (Participants) | 111
  Serotype 34 at Year 2:I | 0.0
  Serotype 35B at Year 2:I: number analyzed (Participants) | 111
  Serotype 35B at Year 2:I | 0.0
  Serotype 35F at Year 2:I: number analyzed (Participants) | 111
  Serotype 35F at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 111
  Serotype 38 at Year 2:I | 0.0
  Serotype clumps at Year 2:I: number analyzed (Participants) | 111
  Serotype clumps at Year 2:I | 0.0
  Serotype Missing/non-viable at Year 2:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 111
  Serotype 3 at Year 3:I | 0.9
  Serotype 6C at Year 3:I: number analyzed (Participants) | 111
  Serotype 6C at Year 3:I | 0.0
  Serotype 7C at Year 3:I: number analyzed (Participants) | 111
  Serotype 7C at Year 3:I | 0.0
  Serotype 9N at Year 3:I: number analyzed (Participants) | 111
  Serotype 9N at Year 3:I | 0.0
  Serotype 10 at Year 3:I: number analyzed (Participants) | 111
  Serotype 10 at Year 3:I | 0.0
  Serotype 11 at Year 3:I: number analyzed (Participants) | 111
  Serotype 11 at Year 3:I | 0.9
  Serotype 12 at Year 3:I: number analyzed (Participants) | 111
  Serotype 12 at Year 3:I | 0.0
  Serotype 12F at Year 3:I: number analyzed (Participants) | 111
  Serotype 12F at Year 3:I | 0.0
  Serotype 13 at Year 3:I: number analyzed (Participants) | 111
  Serotype 13 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 111
  Serotype 15A at Year 3:I | 1.8
  Serotype 15B at Year 3:I: number analyzed (Participants) | 111
  Serotype 15B at Year 3:I | 0.9
  Serotype 15C at Year 3:I: number analyzed (Participants) | 111
  Serotype 15C at Year 3:I | 0.9
  Serotype 15F at Year 3:I: number analyzed (Participants) | 111
  Serotype 15F at Year 3:I | 0.9
  Serotype 16 at Year 3:I: number analyzed (Participants) | 111
  Serotype 16 at Year 3:I | 0.0
  Serotype 17 at Year 3:I: number analyzed (Participants) | 111
  Serotype 17 at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 111
  Serotype 19A at Year 3:I | 2.7
  Serotype 19F at Year 3:I: number analyzed (Participants) | 111
  Serotype 19F at Year 3:I | 2.7
  Serotype 20 at Year 3:I: number analyzed (Participants) | 111
  Serotype 20 at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 111
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 111
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 111
  Serotype 23A at Year 3:I | 0.0
  Serotype 23B at Year 3:I: number analyzed (Participants) | 111
  Serotype 23B at Year 3:I | 0.0
  Serotype 31 at Year 3:I: number analyzed (Participants) | 111
  Serotype 31 at Year 3:I | 0.0
  Serotype 33A at Year 3:I: number analyzed (Participants) | 111
  Serotype 33A at Year 3:I | 0.0
  Serotype 33F at Year 3:I: number analyzed (Participants) | 111
  Serotype 33F at Year 3:I | 0.0
  Serotype 34 at Year 3:I: number analyzed (Participants) | 111
  Serotype 34 at Year 3:I | 0.9
  Serotype 35B at Year 3:I: number analyzed (Participants) | 111
  Serotype 35B at Year 3:I | 0.9
  Serotype 35F at Year 3:I: number analyzed (Participants) | 111
  Serotype 35F at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 111
  Serotype 38 at Year 3:I | 0.0
  Serotype clumps at Year 3:I: number analyzed (Participants) | 111
  Serotype clumps at Year 3:I | 0.0
  Serotype Missing/non-viable at Year 3:I: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 135
  Serotype 3 at Year 1:R | 3.0
  Serotype 6C at Year 1:R: number analyzed (Participants) | 135
  Serotype 6C at Year 1:R | 4.4
  Serotype 7C at Year 1:R: number analyzed (Participants) | 135
  Serotype 7C at Year 1:R | 0.0
  Serotype 9N at Year 1:R: number analyzed (Participants) | 135
  Serotype 9N at Year 1:R | 0.7
  Serotype 10 at Year 1:R: number analyzed (Participants) | 135
  Serotype 10 at Year 1:R | 1.5
  Serotype 11 at Year 1:R: number analyzed (Participants) | 135
  Serotype 11 at Year 1:R | 1.5
  Serotype 12 at Year 1:R: number analyzed (Participants) | 135
  Serotype 12 at Year 1:R | 0.7
  Serotype 12F at Year 1:R: number analyzed (Participants) | 135
  Serotype 12F at Year 1:R | 0.0
  Serotype 13 at Year 1:R: number analyzed (Participants) | 135
  Serotype 13 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 135
  Serotype 15A at Year 1:R | 3.7
  Serotype 15B at Year 1:R: number analyzed (Participants) | 135
  Serotype 15B at Year 1:R | 2.2
  Serotype 15C at Year 1:R: number analyzed (Participants) | 135
  Serotype 15C at Year 1:R | 3.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 135
  Serotype 15F at Year 1:R | 0.0
  Serotype 16 at Year 1:R: number analyzed (Participants) | 135
  Serotype 16 at Year 1:R | 0.0
  Serotype 17 at Year 1:R: number analyzed (Participants) | 135
  Serotype 17 at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 135
  Serotype 19A at Year 1:R | 15.6
  Serotype 19F at Year 1:R: number analyzed (Participants) | 135
  Serotype 19F at Year 1:R | 0.7
  Serotype 20 at Year 1:R: number analyzed (Participants) | 135
  Serotype 20 at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 135
  Serotype 21 at Year 1:R | 1.5
  Serotype 22F at Year 1:R: number analyzed (Participants) | 135
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 135
  Serotype 23A at Year 1:R | 2.2
  Serotype 23B at Year 1:R: number analyzed (Participants) | 135
  Serotype 23B at Year 1:R | 0.7
  Serotype 31 at Year 1:R: number analyzed (Participants) | 135
  Serotype 31 at Year 1:R | 1.5
  Serotype 33A at Year 1:R: number analyzed (Participants) | 135
  Serotype 33A at Year 1:R | 0.7
  Serotype 33F at Year 1:R: number analyzed (Participants) | 135
  Serotype 33F at Year 1:R | 2.2
  Serotype 34 at Year 1:R: number analyzed (Participants) | 135
  Serotype 34 at Year 1:R | 0.0
  Serotype 35B at Year 1:R: number analyzed (Participants) | 135
  Serotype 35B at Year 1:R | 5.9
  Serotype 35F at Year 1:R: number analyzed (Participants) | 135
  Serotype 35F at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 135
  Serotype 38 at Year 1:R | 0.0
  Serotype clumps at Year 1:R: number analyzed (Participants) | 135
  Serotype clumps at Year 1:R | 0.0
  Serotype Missing/non-viable at Year 1:R: number analyzed (Participants) | 135
  Serotype Missing/non-viable at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 111
  Serotype 3 at Year 2:R | 4.5
  Serotype 6C at Year 2:R: number analyzed (Participants) | 111
  Serotype 6C at Year 2:R | 2.7
  Serotype 7C at Year 2:R: number analyzed (Participants) | 111
  Serotype 7C at Year 2:R | 0.0
  Serotype 9N at Year 2:R: number analyzed (Participants) | 111
  Serotype 9N at Year 2:R | 0.0
  Serotype 10 at Year 2:R: number analyzed (Participants) | 111
  Serotype 10 at Year 2:R | 0.9
  Serotype 11 at Year 2:R: number analyzed (Participants) | 111
  Serotype 11 at Year 2:R | 2.7
  Serotype 12 at Year 2:R: number analyzed (Participants) | 111
  Serotype 12 at Year 2:R | 0.0
  Serotype 12F at Year 2:R: number analyzed (Participants) | 111
  Serotype 12F at Year 2:R | 0.9
  Serotype 13 at Year 2:R: number analyzed (Participants) | 111
  Serotype 13 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 111
  Serotype 15A at Year 2:R | 0.9
  Serotype 15B at Year 2:R: number analyzed (Participants) | 111
  Serotype 15B at Year 2:R | 0.9
  Serotype 15C at Year 2:R: number analyzed (Participants) | 111
  Serotype 15C at Year 2:R | 2.7
  Serotype 15F at Year 2:R: number analyzed (Participants) | 111
  Serotype 15F at Year 2:R | 0.0
  Serotype 16 at Year 2:R: number analyzed (Participants) | 111
  Serotype 16 at Year 2:R | 1.8
  Serotype 17 at Year 2:R: number analyzed (Participants) | 111
  Serotype 17 at Year 2:R | 1.8
  Serotype 19A at Year 2:R: number analyzed (Participants) | 111
  Serotype 19A at Year 2:R | 8.1
  Serotype 19F at Year 2:R: number analyzed (Participants) | 111
  Serotype 19F at Year 2:R | 0.9
  Serotype 20 at Year 2:R: number analyzed (Participants) | 111
  Serotype 20 at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 111
  Serotype 21 at Year 2:R | 4.5
  Serotype 22F at Year 2:R: number analyzed (Participants) | 111
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 111
  Serotype 23A at Year 2:R | 3.6
  Serotype 23B at Year 2:R: number analyzed (Participants) | 111
  Serotype 23B at Year 2:R | 5.4
  Serotype 31 at Year 2:R: number analyzed (Participants) | 111
  Serotype 31 at Year 2:R | 1.8
  Serotype 33A at Year 2:R: number analyzed (Participants) | 111
  Serotype 33A at Year 2:R | 0.0
  Serotype 33F at Year 2:R: number analyzed (Participants) | 111
  Serotype 33F at Year 2:R | 0.0
  Serotype 34 at Year 2:R: number analyzed (Participants) | 111
  Serotype 34 at Year 2:R | 0.9
  Serotype 35B at Year 2:R: number analyzed (Participants) | 111
  Serotype 35B at Year 2:R | 9.9
  Serotype 35F at Year 2:R: number analyzed (Participants) | 111
  Serotype 35F at Year 2:R | 0.9
  Serotype 38 at Year 2:R: number analyzed (Participants) | 111
  Serotype 38 at Year 2:R | 0.9
  Serotype clumps at Year 2:R: number analyzed (Participants) | 111
  Serotype clumps at Year 2:R | 0.0
  Serotype Missing/non-viable at Year 2:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 2:R | 0.9
  Serotype 3 at Year 3:R: number analyzed (Participants) | 111
  Serotype 3 at Year 3:R | 3.6
  Serotype 6C at Year 3:R: number analyzed (Participants) | 111
  Serotype 6C at Year 3:R | 0.0
  Serotype 7C at Year 3:R: number analyzed (Participants) | 111
  Serotype 7C at Year 3:R | 0.0
  Serotype 9N at Year 3:R: number analyzed (Participants) | 111
  Serotype 9N at Year 3:R | 0.9
  Serotype 10 at Year 3:R: number analyzed (Participants) | 111
  Serotype 10 at Year 3:R | 2.7
  Serotype 11 at Year 3:R: number analyzed (Participants) | 111
  Serotype 11 at Year 3:R | 1.8
  Serotype 12 at Year 3:R: number analyzed (Participants) | 111
  Serotype 12 at Year 3:R | 0.0
  Serotype 12F at Year 3:R: number analyzed (Participants) | 111
  Serotype 12F at Year 3:R | 0.0
  Serotype 13 at Year 3:R: number analyzed (Participants) | 111
  Serotype 13 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 111
  Serotype 15A at Year 3:R | 2.7
  Serotype 15B at Year 3:R: number analyzed (Participants) | 111
  Serotype 15B at Year 3:R | 3.6
  Serotype 15C at Year 3:R: number analyzed (Participants) | 111
  Serotype 15C at Year 3:R | 1.8
  Serotype 15F at Year 3:R: number analyzed (Participants) | 111
  Serotype 15F at Year 3:R | 0.0
  Serotype 16 at Year 3:R: number analyzed (Participants) | 111
  Serotype 16 at Year 3:R | 3.6
  Serotype 17 at Year 3:R: number analyzed (Participants) | 111
  Serotype 17 at Year 3:R | 0.9
  Serotype 19A at Year 3:R: number analyzed (Participants) | 111
  Serotype 19A at Year 3:R | 6.3
  Serotype 19F at Year 3:R: number analyzed (Participants) | 111
  Serotype 19F at Year 3:R | 1.8
  Serotype 20 at Year 3:R: number analyzed (Participants) | 111
  Serotype 20 at Year 3:R | 0.9
  Serotype 21 at Year 3:R: number analyzed (Participants) | 111
  Serotype 21 at Year 3:R | 1.8
  Serotype 22F at Year 3:R: number analyzed (Participants) | 111
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 111
  Serotype 23A at Year 3:R | 2.7
  Serotype 23B at Year 3:R: number analyzed (Participants) | 111
  Serotype 23B at Year 3:R | 6.3
  Serotype 31 at Year 3:R: number analyzed (Participants) | 111
  Serotype 31 at Year 3:R | 2.7
  Serotype 33A at Year 3:R: number analyzed (Participants) | 111
  Serotype 33A at Year 3:R | 0.0
  Serotype 33F at Year 3:R: number analyzed (Participants) | 111
  Serotype 33F at Year 3:R | 1.8
  Serotype 34 at Year 3:R: number analyzed (Participants) | 111
  Serotype 34 at Year 3:R | 0.0
  Serotype 35B at Year 3:R: number analyzed (Participants) | 111
  Serotype 35B at Year 3:R | 9.0
  Serotype 35F at Year 3:R: number analyzed (Participants) | 111
  Serotype 35F at Year 3:R | 0.9
  Serotype 38 at Year 3:R: number analyzed (Participants) | 111
  Serotype 38 at Year 3:R | 0.9
  Serotype clumps at Year 3:R: number analyzed (Participants) | 111
  Serotype clumps at Year 3:R | 0.0
  Serotype Missing/non-viable at Year 3:R: number analyzed (Participants) | 111
  Serotype Missing/non-viable at Year 3:R | 1.8

14. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Ceftriaxone: Mastoid Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for ceftriaxone from mastoid samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 12, 15A, 15B, 15F, 19A, 19F, 21, 22F, 23A, 38, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. 'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: Mastoid population. N (number of participants analyzed) includes total number of participants in mastoid population, however actual 'N' for this OM is unknown as this data were not calculated as per planned analysis and number analyzed=number of isolates for the given serotype at specified time point.
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
Number analyzed (Isolates) | 29
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 18
  Serotype 3 at Year 1:S | 0.0
  Serotype 12 at Year 1:S: number analyzed (Participants) | 18
  Serotype 12 at Year 1:S | 5.6
  Serotype 15A at Year 1:S: number analyzed (Participants) | 18
  Serotype 15A at Year 1:S | 5.6
  Serotype 15B at Year 1:S: number analyzed (Participants) | 18
  Serotype 15B at Year 1:S | 5.6
  Serotype 15F at Year 1:S: number analyzed (Participants) | 18
  Serotype 15F at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 18
  Serotype 19A at Year 1:S | 27.8
  Serotype 19F at Year 1:S: number analyzed (Participants) | 18
  Serotype 19F at Year 1:S | 11.1
  Serotype 21 at Year 1:S: number analyzed (Participants) | 18
  Serotype 21 at Year 1:S | 0.0
  Serotype 22F at Year 1:S: number analyzed (Participants) | 18
  Serotype 22F at Year 1:S | 11.1
  Serotype 23A at Year 1:S: number analyzed (Participants) | 18
  Serotype 23A at Year 1:S | 5.6
  Serotype 38 at Year 1:S: number analyzed (Participants) | 18
  Serotype 38 at Year 1:S | 5.6
  Serotype 3 at Year 2:S: number analyzed (Participants) | 7
  Serotype 3 at Year 2:S | 28.6
  Serotype 12 at Year 2:S: number analyzed (Participants) | 7
  Serotype 12 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 7
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 7
  Serotype 15B at Year 2:S | 0.0
  Serotype 15F at Year 2:S: number analyzed (Participants) | 7
  Serotype 15F at Year 2:S | 0.0
  Serotype 19A at Year 2:S: number analyzed (Participants) | 7
  Serotype 19A at Year 2:S | 57.1
  Serotype 19F at Year 2:S: number analyzed (Participants) | 7
  Serotype 19F at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 7
  Serotype 21 at Year 2:S | 0.0
  Serotype 22F at Year 2:S: number analyzed (Participants) | 7
  Serotype 22F at Year 2:S | 0.0
  Serotype 23A at Year 2:S: number analyzed (Participants) | 7
  Serotype 23A at Year 2:S | 0.0
  Serotype 38 at Year 2:S: number analyzed (Participants) | 7
  Serotype 38 at Year 2:S | 0.0
  Serotype 3 at Year 3:S: number analyzed (Participants) | 9
  Serotype 3 at Year 3:S | 44.4
  Serotype 12 at Year 3:S: number analyzed (Participants) | 9
  Serotype 12 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 9
  Serotype 15A at Year 3:S | 0.0
  Serotype 15B at Year 3:S: number analyzed (Participants) | 9
  Serotype 15B at Year 3:S | 0.0
  Serotype 15F at Year 3:S: number analyzed (Participants) | 9
  Serotype 15F at Year 3:S | 0.0
  Serotype 19A at Year 3:S: number analyzed (Participants) | 9
  Serotype 19A at Year 3:S | 0.0
  Serotype 19F at Year 3:S: number analyzed (Participants) | 9
  Serotype 19F at Year 3:S | 11.1
  Serotype 21 at Year 3:S: number analyzed (Participants) | 9
  Serotype 21 at Year 3:S | 0.0
  Serotype 22F at Year 3:S: number analyzed (Participants) | 9
  Serotype 22F at Year 3:S | 0.0
  Serotype 23A at Year 3:S: number analyzed (Participants) | 9
  Serotype 23A at Year 3:S | 0.0
  Serotype 38 at Year 3:S: number analyzed (Participants) | 9
  Serotype 38 at Year 3:S | 0.0
  Serotype 3 at Year 1:I: number analyzed (Participants) | 18
  Serotype 3 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 18
  Serotype 12 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 18
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 18
  Serotype 15B at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 18
  Serotype 15F at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 18
  Serotype 19A at Year 1:I | 0.0
  Serotype 19F at Year 1:I: number analyzed (Participants) | 18
  Serotype 19F at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 18
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 18
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 18
  Serotype 23A at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 18
  Serotype 38 at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 7
  Serotype 3 at Year 2:I | 0.0
  Serotype 12 at Year 2:I: number analyzed (Participants) | 7
  Serotype 12 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 7
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 7
  Serotype 15B at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 7
  Serotype 15F at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 7
  Serotype 19A at Year 2:I | 0.0
  Serotype 19F at Year 2:I: number analyzed (Participants) | 7
  Serotype 19F at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 7
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 7
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 7
  Serotype 23A at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 7
  Serotype 38 at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 9
  Serotype 3 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 9
  Serotype 12 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 9
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 9
  Serotype 15B at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 9
  Serotype 15F at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 9
  Serotype 19A at Year 3:I | 0.0
  Serotype 19F at Year 3:I: number analyzed (Participants) | 9
  Serotype 19F at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 9
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 9
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 9
  Serotype 23A at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 9
  Serotype 38 at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 18
  Serotype 3 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 18
  Serotype 12 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 18
  Serotype 15A at Year 1:R | 0.0
  Serotype 15B at Year 1:R: number analyzed (Participants) | 18
  Serotype 15B at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 18
  Serotype 15F at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 18
  Serotype 19A at Year 1:R | 5.6
  Serotype 19F at Year 1:R: number analyzed (Participants) | 18
  Serotype 19F at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 18
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 18
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 18
  Serotype 23A at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 18
  Serotype 38 at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 7
  Serotype 3 at Year 2:R | 0.0
  Serotype 12 at Year 2:R: number analyzed (Participants) | 7
  Serotype 12 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 7
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 7
  Serotype 15B at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 7
  Serotype 15F at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 7
  Serotype 19A at Year 2:R | 0.0
  Serotype 19F at Year 2:R: number analyzed (Participants) | 7
  Serotype 19F at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 7
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 7
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 7
  Serotype 23A at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 7
  Serotype 38 at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 9
  Serotype 3 at Year 3:R | 0.0
  Serotype 12 at Year 3:R: number analyzed (Participants) | 9
  Serotype 12 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 9
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 9
  Serotype 15B at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 9
  Serotype 15F at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 9
  Serotype 19A at Year 3:R | 11.1
  Serotype 19F at Year 3:R: number analyzed (Participants) | 9
  Serotype 19F at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 9
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 9
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 9
  Serotype 23A at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 9
  Serotype 38 at Year 3:R | 0.0

15. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Clindamycin: Mastoid Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for clindamycin from mastoid samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 12, 15A, 15B, 15F, 19A, 19F, 21, 22F, 23A, 38, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. 'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: as for outcome 14
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
Number analyzed (Isolates) | 29
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 18
  Serotype 3 at Year 1:S | 0.0
  Serotype 15F at Year 1:S: number analyzed (Participants) | 18
  Serotype 15F at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 18
  Serotype 19A at Year 1:S | 5.6
  Serotype 19F at Year 1:S: number analyzed (Participants) | 18
  Serotype 19F at Year 1:S | 0.0
  Serotype 21 at Year 1:S: number analyzed (Participants) | 18
  Serotype 21 at Year 1:S | 0.0
  Serotype 22F at Year 1:S: number analyzed (Participants) | 18
  Serotype 22F at Year 1:S | 5.6
  Serotype 23A at Year 1:S: number analyzed (Participants) | 18
  Serotype 23A at Year 1:S | 5.6
  Serotype 38 at Year 1:S: number analyzed (Participants) | 18
  Serotype 38 at Year 1:S | 5.6
  Serotype 3 at Year 2:S: number analyzed (Participants) | 7
  Serotype 3 at Year 2:S | 28.6
  Serotype 12 at Year 2:S: number analyzed (Participants) | 7
  Serotype 12 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 7
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 7
  Serotype 15B at Year 2:S | 0.0
  Serotype 15F at Year 2:S: number analyzed (Participants) | 7
  Serotype 15F at Year 2:S | 0.0
  Serotype 19A at Year 2:S: number analyzed (Participants) | 7
  Serotype 19A at Year 2:S | 28.6
  Serotype 19F at Year 2:S: number analyzed (Participants) | 7
  Serotype 19F at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 7
  Serotype 21 at Year 2:S | 0.0
  Serotype 22F at Year 2:S: number analyzed (Participants) | 7
  Serotype 22F at Year 2:S | 0.0
  Serotype 23A at Year 2:S: number analyzed (Participants) | 7
  Serotype 23A at Year 2:S | 0.0
  Serotype 38 at Year 2:S: number analyzed (Participants) | 7
  Serotype 38 at Year 2:S | 0.0
  Serotype 3 at Year 3:S: number analyzed (Participants) | 9
  Serotype 3 at Year 3:S | 22.2
  Serotype 12 at Year 3:S: number analyzed (Participants) | 9
  Serotype 12 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 9
  Serotype 15A at Year 3:S | 0.0
  Serotype 15B at Year 3:S: number analyzed (Participants) | 9
  Serotype 15B at Year 3:S | 0.0
  Serotype 15F at Year 3:S: number analyzed (Participants) | 9
  Serotype 15F at Year 3:S | 0.0
  Serotype 19A at Year 3:S: number analyzed (Participants) | 9
  Serotype 19A at Year 3:S | 0.0
  Serotype 19F at Year 3:S: number analyzed (Participants) | 9
  Serotype 19F at Year 3:S | 11.1
  Serotype 21 at Year 3:S: number analyzed (Participants) | 9
  Serotype 21 at Year 3:S | 0.0
  Serotype 22F at Year 3:S: number analyzed (Participants) | 9
  Serotype 22F at Year 3:S | 0.0
  Serotype 23A at Year 3:S: number analyzed (Participants) | 9
  Serotype 23A at Year 3:S | 0.0
  Serotype 38 at Year 3:S: number analyzed (Participants) | 9
  Serotype 38 at Year 3:S | 0.0
  Serotype 3 at Year 1:I: number analyzed (Participants) | 18
  Serotype 3 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 18
  Serotype 12 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 18
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 18
  Serotype 15B at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 18
  Serotype 15F at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 18
  Serotype 19A at Year 1:I | 5.6
  Serotype 19F at Year 1:I: number analyzed (Participants) | 18
  Serotype 19F at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 18
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 18
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 18
  Serotype 23A at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 18
  Serotype 38 at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 7
  Serotype 3 at Year 2:I | 0.0
  Serotype 12 at Year 2:I: number analyzed (Participants) | 7
  Serotype 12 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 7
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 7
  Serotype 15B at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 7
  Serotype 15F at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 7
  Serotype 19A at Year 2:I | 14.3
  Serotype 19F at Year 2:I: number analyzed (Participants) | 7
  Serotype 19F at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 7
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 7
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 7
  Serotype 23A at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 7
  Serotype 38 at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 9
  Serotype 3 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 9
  Serotype 12 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 9
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 9
  Serotype 15B at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 9
  Serotype 15F at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 9
  Serotype 19A at Year 3:I | 0.0
  Serotype 19F at Year 3:I: number analyzed (Participants) | 9
  Serotype 19F at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 9
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 9
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 9
  Serotype 23A at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 9
  Serotype 38 at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 18
  Serotype 3 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 18
  Serotype 12 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 18
  Serotype 15A at Year 1:R | 5.6
  Serotype 15B at Year 1:R: number analyzed (Participants) | 18
  Serotype 15B at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 18
  Serotype 15F at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 18
  Serotype 19A at Year 1:R | 22.2
  Serotype 19F at Year 1:R: number analyzed (Participants) | 18
  Serotype 19F at Year 1:R | 5.6
  Serotype 21 at Year 1:R: number analyzed (Participants) | 18
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 18
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 18
  Serotype 23A at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 18
  Serotype 38 at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 7
  Serotype 3 at Year 2:R | 0.0
  Serotype 12 at Year 2:R: number analyzed (Participants) | 7
  Serotype 12 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 7
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 7
  Serotype 15B at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 7
  Serotype 15F at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 7
  Serotype 19A at Year 2:R | 28.6
  Serotype 19F at Year 2:R: number analyzed (Participants) | 7
  Serotype 19F at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 7
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 7
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 7
  Serotype 23A at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 7
  Serotype 38 at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 9
  Serotype 3 at Year 3:R | 11.1
  Serotype 12 at Year 3:R: number analyzed (Participants) | 9
  Serotype 12 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 9
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 9
  Serotype 15B at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 9
  Serotype 15F at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 9
  Serotype 19A at Year 3:R | 11.1
  Serotype 19F at Year 3:R: number analyzed (Participants) | 9
  Serotype 19F at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 9
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 9
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 9
  Serotype 23A at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 9
  Serotype 38 at Year 3:R | 0.0
  Serotype 12 at Year 1:S: number analyzed (Participants) | 18
  Serotype 12 at Year 1:S | 5.6
  Serotype 15A at Year 1:S: number analyzed (Participants) | 18
  Serotype 15A at Year 1:S | 0.0
  Serotype 15B at Year 1:S: number analyzed (Participants) | 18
  Serotype 15B at Year 1:S | 5.6

16. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Erythromycin: Mastoid Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for erythromycin from mastoid samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 12, 15A, 15B, 15F, 19A, 19F, 21, 22F, 23A, 38, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. 'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: as for outcome 14
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
Number analyzed (Isolates) | 29
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 18
  Serotype 3 at Year 1:S | 0.0
  Serotype 12 at Year 1:S: number analyzed (Participants) | 18
  Serotype 12 at Year 1:S | 5.6
  Serotype 15A at Year 1:S: number analyzed (Participants) | 18
  Serotype 15A at Year 1:S | 0.0
  Serotype 15B at Year 1:S: number analyzed (Participants) | 18
  Serotype 15B at Year 1:S | 5.6
  Serotype 15F at Year 1:S: number analyzed (Participants) | 18
  Serotype 15F at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 18
  Serotype 19A at Year 1:S | 5.6
  Serotype 19F at Year 1:S: number analyzed (Participants) | 18
  Serotype 19F at Year 1:S | 5.6
  Serotype 21 at Year 1:S: number analyzed (Participants) | 18
  Serotype 21 at Year 1:S | 0.0
  Serotype 22F at Year 1:S: number analyzed (Participants) | 18
  Serotype 22F at Year 1:S | 11.1
  Serotype 23A at Year 1:S: number analyzed (Participants) | 18
  Serotype 23A at Year 1:S | 5.6
  Serotype 38 at Year 1:S: number analyzed (Participants) | 18
  Serotype 38 at Year 1:S | 5.6
  Serotype 3 at Year 2:S: number analyzed (Participants) | 7
  Serotype 3 at Year 2:S | 28.6
  Serotype 12 at Year 2:S: number analyzed (Participants) | 7
  Serotype 12 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 7
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 7
  Serotype 15B at Year 2:S | 0.0
  Serotype 15F at Year 2:S: number analyzed (Participants) | 7
  Serotype 15F at Year 2:S | 0.0
  Serotype 19A at Year 2:S: number analyzed (Participants) | 7
  Serotype 19A at Year 2:S | 28.6
  Serotype 19F at Year 2:S: number analyzed (Participants) | 7
  Serotype 19F at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 7
  Serotype 21 at Year 2:S | 0.0
  Serotype 22F at Year 2:S: number analyzed (Participants) | 7
  Serotype 22F at Year 2:S | 0.0
  Serotype 23A at Year 2:S: number analyzed (Participants) | 7
  Serotype 23A at Year 2:S | 0.0
  Serotype 38 at Year 2:S: number analyzed (Participants) | 7
  Serotype 38 at Year 2:S | 0.0
  Serotype 3 at Year 3:S: number analyzed (Participants) | 9
  Serotype 3 at Year 3:S | 33.3
  Serotype 12 at Year 3:S: number analyzed (Participants) | 9
  Serotype 12 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 9
  Serotype 15A at Year 3:S | 0.0
  Serotype 15B at Year 3:S: number analyzed (Participants) | 9
  Serotype 15B at Year 3:S | 0.0
  Serotype 15F at Year 3:S: number analyzed (Participants) | 9
  Serotype 15F at Year 3:S | 0.0
  Serotype 19A at Year 3:S: number analyzed (Participants) | 9
  Serotype 19A at Year 3:S | 0.0
  Serotype 19F at Year 3:S: number analyzed (Participants) | 9
  Serotype 19F at Year 3:S | 0.0
  Serotype 21 at Year 3:S: number analyzed (Participants) | 9
  Serotype 21 at Year 3:S | 0.0
  Serotype 22F at Year 3:S: number analyzed (Participants) | 9
  Serotype 22F at Year 3:S | 0.0
  Serotype 23A at Year 3:S: number analyzed (Participants) | 9
  Serotype 23A at Year 3:S | 0.0
  Serotype 38 at Year 3:S: number analyzed (Participants) | 9
  Serotype 38 at Year 3:S | 0.0
  Serotype 3 at Year 1:I: number analyzed (Participants) | 18
  Serotype 3 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 18
  Serotype 12 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 18
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 18
  Serotype 15B at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 18
  Serotype 15F at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 18
  Serotype 19A at Year 1:I | 5.6
  Serotype 19F at Year 1:I: number analyzed (Participants) | 18
  Serotype 19F at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 18
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 18
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 18
  Serotype 23A at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 18
  Serotype 38 at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 7
  Serotype 3 at Year 2:I | 0.0
  Serotype 12 at Year 2:I: number analyzed (Participants) | 7
  Serotype 12 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 7
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 7
  Serotype 15B at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 7
  Serotype 15F at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 7
  Serotype 19A at Year 2:I | 14.3
  Serotype 19F at Year 2:I: number analyzed (Participants) | 7
  Serotype 19F at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 7
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 7
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 7
  Serotype 23A at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 7
  Serotype 38 at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 9
  Serotype 3 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 9
  Serotype 12 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 9
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 9
  Serotype 15B at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 9
  Serotype 15F at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 9
  Serotype 19A at Year 3:I | 0.0
  Serotype 19F at Year 3:I: number analyzed (Participants) | 9
  Serotype 19F at Year 3:I | 11.1
  Serotype 21 at Year 3:I: number analyzed (Participants) | 9
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 9
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 9
  Serotype 23A at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 9
  Serotype 38 at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 18
  Serotype 3 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 18
  Serotype 12 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 18
  Serotype 15A at Year 1:R | 5.6
  Serotype 15B at Year 1:R: number analyzed (Participants) | 18
  Serotype 15B at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 18
  Serotype 15F at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 18
  Serotype 19A at Year 1:R | 22.2
  Serotype 19F at Year 1:R: number analyzed (Participants) | 18
  Serotype 19F at Year 1:R | 0.0
  Serotype 21 at Year 1:R: number analyzed (Participants) | 18
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 18
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 18
  Serotype 23A at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 18
  Serotype 38 at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 7
  Serotype 3 at Year 2:R | 0.0
  Serotype 12 at Year 2:R: number analyzed (Participants) | 7
  Serotype 12 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 7
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 7
  Serotype 15B at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 7
  Serotype 15F at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 7
  Serotype 19A at Year 2:R | 28.6
  Serotype 19F at Year 2:R: number analyzed (Participants) | 7
  Serotype 19F at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 7
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 7
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 7
  Serotype 23A at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 7
  Serotype 38 at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 9
  Serotype 3 at Year 3:R | 11.1
  Serotype 12 at Year 3:R: number analyzed (Participants) | 9
  Serotype 12 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 9
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 9
  Serotype 15B at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 9
  Serotype 15F at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 9
  Serotype 19A at Year 3:R | 11.1
  Serotype 19F at Year 3:R: number analyzed (Participants) | 9
  Serotype 19F at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 9
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 9
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 9
  Serotype 23A at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 9
  Serotype 38 at Year 3:R | 0.0

17. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Penicillin: Mastoid Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for penicillin from mastoid samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 12, 15A, 15B, 15F, 19A, 19F, 21, 22F, 23A, 38, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. 'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: as for outcome 14
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
Number analyzed (Isolates) | 29
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 18
  Serotype 3 at Year 1:S | 0.0
  Serotype 12 at Year 1:S: number analyzed (Participants) | 18
  Serotype 12 at Year 1:S | 5.6
  Serotype 15A at Year 1:S: number analyzed (Participants) | 18
  Serotype 15A at Year 1:S | 0.0
  Serotype 15B at Year 1:S: number analyzed (Participants) | 18
  Serotype 15B at Year 1:S | 5.6
  Serotype 15F at Year 1:S: number analyzed (Participants) | 18
  Serotype 15F at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 18
  Serotype 19A at Year 1:S | 5.6
  Serotype 19F at Year 1:S: number analyzed (Participants) | 18
  Serotype 19F at Year 1:S | 5.6
  Serotype 21 at Year 1:S: number analyzed (Participants) | 18
  Serotype 21 at Year 1:S | 0.0
  Serotype 22F at Year 1:S: number analyzed (Participants) | 18
  Serotype 22F at Year 1:S | 11.1
  Serotype 23A at Year 1:S: number analyzed (Participants) | 18
  Serotype 23A at Year 1:S | 5.6
  Serotype 38 at Year 1:S: number analyzed (Participants) | 18
  Serotype 38 at Year 1:S | 5.6
  Serotype 3 at Year 2:S: number analyzed (Participants) | 7
  Serotype 3 at Year 2:S | 28.6
  Serotype 12 at Year 2:S: number analyzed (Participants) | 7
  Serotype 12 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 7
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 7
  Serotype 15B at Year 2:S | 0.0
  Serotype 15F at Year 2:S: number analyzed (Participants) | 7
  Serotype 15F at Year 2:S | 0.0
  Serotype 19A at Year 2:S: number analyzed (Participants) | 7
  Serotype 19A at Year 2:S | 14.3
  Serotype 19F at Year 2:S: number analyzed (Participants) | 7
  Serotype 19F at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 7
  Serotype 21 at Year 2:S | 0.0
  Serotype 22F at Year 2:S: number analyzed (Participants) | 7
  Serotype 22F at Year 2:S | 0.0
  Serotype 23A at Year 2:S: number analyzed (Participants) | 7
  Serotype 23A at Year 2:S | 0.0
  Serotype 38 at Year 2:S: number analyzed (Participants) | 7
  Serotype 38 at Year 2:S | 0.0
  Serotype 3 at Year 3:S: number analyzed (Participants) | 9
  Serotype 3 at Year 3:S | 44.4
  Serotype 12 at Year 3:S: number analyzed (Participants) | 9
  Serotype 12 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 9
  Serotype 15A at Year 3:S | 0.0
  Serotype 15B at Year 3:S: number analyzed (Participants) | 9
  Serotype 15B at Year 3:S | 0.0
  Serotype 15F at Year 3:S: number analyzed (Participants) | 9
  Serotype 15F at Year 3:S | 0.0
  Serotype 19A at Year 3:S: number analyzed (Participants) | 9
  Serotype 19A at Year 3:S | 0.0
  Serotype 19F at Year 3:S: number analyzed (Participants) | 9
  Serotype 19F at Year 3:S | 0.0
  Serotype 21 at Year 3:S: number analyzed (Participants) | 9
  Serotype 21 at Year 3:S | 0.0
  Serotype 22F at Year 3:S: number analyzed (Participants) | 9
  Serotype 22F at Year 3:S | 11.1
  Serotype 23A at Year 3:S: number analyzed (Participants) | 9
  Serotype 23A at Year 3:S | 0.0
  Serotype 38 at Year 3:S: number analyzed (Participants) | 9
  Serotype 38 at Year 3:S | 0.0
  Serotype 3 at Year 1:I: number analyzed (Participants) | 18
  Serotype 3 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 18
  Serotype 12 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 18
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 18
  Serotype 15B at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 18
  Serotype 15F at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 18
  Serotype 19A at Year 1:I | 0.0
  Serotype 19F at Year 1:I: number analyzed (Participants) | 18
  Serotype 19F at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 18
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 18
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 18
  Serotype 23A at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 18
  Serotype 38 at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 7
  Serotype 3 at Year 2:I | 0.0
  Serotype 12 at Year 2:I: number analyzed (Participants) | 7
  Serotype 12 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 7
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 7
  Serotype 15B at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 7
  Serotype 15F at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 7
  Serotype 19A at Year 2:I | 0.0
  Serotype 19F at Year 2:I: number analyzed (Participants) | 7
  Serotype 19F at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 7
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 7
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 7
  Serotype 23A at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 7
  Serotype 38 at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 9
  Serotype 3 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 9
  Serotype 12 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 9
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 9
  Serotype 15B at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 9
  Serotype 15F at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 9
  Serotype 19A at Year 3:I | 0.0
  Serotype 19F at Year 3:I: number analyzed (Participants) | 9
  Serotype 19F at Year 3:I | 0.0
  Serotype 21 at Year 3:I: number analyzed (Participants) | 9
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 9
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 9
  Serotype 23A at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 9
  Serotype 38 at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 18
  Serotype 3 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 18
  Serotype 12 at Year 1:R | 0.0
  Serotype 15A at Year 1:R: number analyzed (Participants) | 18
  Serotype 15A at Year 1:R | 5.6
  Serotype 15B at Year 1:R: number analyzed (Participants) | 18
  Serotype 15B at Year 1:R | 0.0
  Serotype 15F at Year 1:R: number analyzed (Participants) | 18
  Serotype 15F at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 18
  Serotype 19A at Year 1:R | 33.3
  Serotype 19F at Year 1:R: number analyzed (Participants) | 18
  Serotype 19F at Year 1:R | 5.6
  Serotype 21 at Year 1:R: number analyzed (Participants) | 18
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 18
  Serotype 22F at Year 1:R | 0.0
  Serotype 23A at Year 1:R: number analyzed (Participants) | 18
  Serotype 23A at Year 1:R | 0.0
  Serotype 38 at Year 1:R: number analyzed (Participants) | 18
  Serotype 38 at Year 1:R | 0.0
  Serotype 3 at Year 2:R: number analyzed (Participants) | 7
  Serotype 3 at Year 2:R | 0.0
  Serotype 12 at Year 2:R: number analyzed (Participants) | 7
  Serotype 12 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 7
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 7
  Serotype 15B at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 7
  Serotype 15F at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 7
  Serotype 19A at Year 2:R | 57.1
  Serotype 19F at Year 2:R: number analyzed (Participants) | 7
  Serotype 19F at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 7
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 7
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 7
  Serotype 23A at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 7
  Serotype 38 at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 9
  Serotype 3 at Year 3:R | 0.0
  Serotype 12 at Year 3:R: number analyzed (Participants) | 9
  Serotype 12 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 9
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 9
  Serotype 15B at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 9
  Serotype 15F at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 9
  Serotype 19A at Year 3:R | 11.1
  Serotype 19F at Year 3:R: number analyzed (Participants) | 9
  Serotype 19F at Year 3:R | 11.1
  Serotype 21 at Year 3:R: number analyzed (Participants) | 9
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 9
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 9
  Serotype 23A at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 9
  Serotype 38 at Year 3:R | 0.0

18. Secondary Outcome: Antimicrobial Susceptibility of Streptococcus Pneumoniae Isolates for Trimethoprim/Sulfamethoxazole (TMP/S): Mastoid Population
Description: Antimicrobial susceptibility of S pneumoniae isolates for TMP/S from mastoid samples was categorized as resistant, susceptible or intermediate based on MIC for each serotype at each year of the whole surveillance period. The percentage of S pneumoniae serotypes included 3, 12, 15A, 15B, 15F, 19A, 19F, 21, 22F, 23A, 38, which were to be computed along with exact 2-sided 95% CI based on the observed proportion of isolates. 'Number of isolates analyzed' signifies total number of isolates that were evaluable for this OM.
Time Frame: Surveillance Year 1, 2, 3
Population: as for outcome 14
Measure: Number; unit: percentage of isolates
Units Other Than Participants: Isolates
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
Number analyzed (Isolates) | 29
percentage of isolates
  Serotype 3 at Year 1:S: number analyzed (Participants) | 18
  Serotype 3 at Year 1:S | 0.0
  Serotype 12 at Year 1:S: number analyzed (Participants) | 18
  Serotype 12 at Year 1:S | 0.0
  Serotype 15A at Year 1:S: number analyzed (Participants) | 18
  Serotype 15A at Year 1:S | 0.0
  Serotype 15B at Year 1:S: number analyzed (Participants) | 18
  Serotype 15B at Year 1:S | 0.0
  Serotype 15F at Year 1:S: number analyzed (Participants) | 18
  Serotype 15F at Year 1:S | 0.0
  Serotype 19A at Year 1:S: number analyzed (Participants) | 18
  Serotype 19A at Year 1:S | 0.0
  Serotype 19F at Year 1:S: number analyzed (Participants) | 18
  Serotype 19F at Year 1:S | 5.6
  Serotype 21 at Year 1:S: number analyzed (Participants) | 18
  Serotype 21 at Year 1:S | 0.0
  Serotype 22F at Year 1:S: number analyzed (Participants) | 18
  Serotype 22F at Year 1:S | 5.6
  Serotype 23A at Year 1:S: number analyzed (Participants) | 18
  Serotype 23A at Year 1:S | 0.0
  Serotype 38 at Year 1:S: number analyzed (Participants) | 18
  Serotype 38 at Year 1:S | 0.0
  Serotype 3 at Year 2:S: number analyzed (Participants) | 7
  Serotype 3 at Year 2:S | 0.0
  Serotype 12 at Year 2:S: number analyzed (Participants) | 7
  Serotype 12 at Year 2:S | 0.0
  Serotype 15A at Year 2:S: number analyzed (Participants) | 7
  Serotype 15A at Year 2:S | 0.0
  Serotype 15B at Year 2:S: number analyzed (Participants) | 7
  Serotype 15B at Year 2:S | 0.0
  Serotype 15F at Year 2:S: number analyzed (Participants) | 7
  Serotype 15F at Year 2:S | 0.0
  Serotype 19A at Year 2:S: number analyzed (Participants) | 7
  Serotype 19A at Year 2:S | 0.0
  Serotype 19F at Year 2:S: number analyzed (Participants) | 7
  Serotype 19F at Year 2:S | 0.0
  Serotype 21 at Year 2:S: number analyzed (Participants) | 7
  Serotype 21 at Year 2:S | 0.0
  Serotype 22F at Year 2:S: number analyzed (Participants) | 7
  Serotype 22F at Year 2:S | 0.0
  Serotype 23A at Year 2:S: number analyzed (Participants) | 7
  Serotype 23A at Year 2:S | 0.0
  Serotype 38 at Year 2:S: number analyzed (Participants) | 7
  Serotype 38 at Year 2:S | 0.0
  Serotype 3 at Year 3:S: number analyzed (Participants) | 9
  Serotype 3 at Year 3:S | 33.3
  Serotype 12 at Year 3:S: number analyzed (Participants) | 9
  Serotype 12 at Year 3:S | 0.0
  Serotype 15A at Year 3:S: number analyzed (Participants) | 9
  Serotype 15A at Year 3:S | 0.0
  Serotype 15B at Year 3:S: number analyzed (Participants) | 9
  Serotype 15B at Year 3:S | 0.0
  Serotype 15F at Year 3:S: number analyzed (Participants) | 9
  Serotype 15F at Year 3:S | 0.0
  Serotype 19A at Year 3:S: number analyzed (Participants) | 9
  Serotype 19A at Year 3:S | 0.0
  Serotype 19F at Year 3:S: number analyzed (Participants) | 9
  Serotype 19F at Year 3:S | 0.0
  Serotype 21 at Year 3:S: number analyzed (Participants) | 9
  Serotype 21 at Year 3:S | 0.0
  Serotype 22F at Year 3:S: number analyzed (Participants) | 9
  Serotype 22F at Year 3:S | 0.0
  Serotype 23A at Year 3:S: number analyzed (Participants) | 9
  Serotype 23A at Year 3:S | 0.0
  Serotype 38 at Year 3:S: number analyzed (Participants) | 9
  Serotype 38 at Year 3:S | 0.0
  Serotype 3 at Year 1:I: number analyzed (Participants) | 18
  Serotype 3 at Year 1:I | 0.0
  Serotype 12 at Year 1:I: number analyzed (Participants) | 18
  Serotype 12 at Year 1:I | 0.0
  Serotype 15A at Year 1:I: number analyzed (Participants) | 18
  Serotype 15A at Year 1:I | 0.0
  Serotype 15B at Year 1:I: number analyzed (Participants) | 18
  Serotype 15B at Year 1:I | 0.0
  Serotype 15F at Year 1:I: number analyzed (Participants) | 18
  Serotype 15F at Year 1:I | 0.0
  Serotype 19A at Year 1:I: number analyzed (Participants) | 18
  Serotype 19A at Year 1:I | 5.6
  Serotype 19F at Year 1:I: number analyzed (Participants) | 18
  Serotype 19F at Year 1:I | 0.0
  Serotype 21 at Year 1:I: number analyzed (Participants) | 18
  Serotype 21 at Year 1:I | 0.0
  Serotype 22F at Year 1:I: number analyzed (Participants) | 18
  Serotype 22F at Year 1:I | 0.0
  Serotype 23A at Year 1:I: number analyzed (Participants) | 18
  Serotype 23A at Year 1:I | 0.0
  Serotype 38 at Year 1:I: number analyzed (Participants) | 18
  Serotype 38 at Year 1:I | 0.0
  Serotype 3 at Year 2:I: number analyzed (Participants) | 7
  Serotype 3 at Year 2:I | 0.0
  Serotype 12 at Year 2:I: number analyzed (Participants) | 7
  Serotype 12 at Year 2:I | 0.0
  Serotype 15A at Year 2:I: number analyzed (Participants) | 7
  Serotype 15A at Year 2:I | 0.0
  Serotype 15B at Year 2:I: number analyzed (Participants) | 7
  Serotype 15B at Year 2:I | 0.0
  Serotype 15F at Year 2:I: number analyzed (Participants) | 7
  Serotype 15F at Year 2:I | 0.0
  Serotype 19A at Year 2:I: number analyzed (Participants) | 7
  Serotype 19A at Year 2:I | 28.6
  Serotype 19F at Year 2:I: number analyzed (Participants) | 7
  Serotype 19F at Year 2:I | 0.0
  Serotype 21 at Year 2:I: number analyzed (Participants) | 7
  Serotype 21 at Year 2:I | 0.0
  Serotype 22F at Year 2:I: number analyzed (Participants) | 7
  Serotype 22F at Year 2:I | 0.0
  Serotype 23A at Year 2:I: number analyzed (Participants) | 7
  Serotype 23A at Year 2:I | 0.0
  Serotype 38 at Year 2:I: number analyzed (Participants) | 7
  Serotype 38 at Year 2:I | 0.0
  Serotype 3 at Year 3:I: number analyzed (Participants) | 9
  Serotype 3 at Year 3:I | 0.0
  Serotype 12 at Year 3:I: number analyzed (Participants) | 9
  Serotype 12 at Year 3:I | 0.0
  Serotype 15A at Year 3:I: number analyzed (Participants) | 9
  Serotype 15A at Year 3:I | 0.0
  Serotype 15B at Year 3:I: number analyzed (Participants) | 9
  Serotype 15B at Year 3:I | 0.0
  Serotype 15F at Year 3:I: number analyzed (Participants) | 9
  Serotype 15F at Year 3:I | 0.0
  Serotype 19A at Year 3:I: number analyzed (Participants) | 9
  Serotype 19A at Year 3:I | 0.0
  Serotype 19F at Year 3:I: number analyzed (Participants) | 9
  Serotype 19F at Year 3:I | 11.1
  Serotype 21 at Year 3:I: number analyzed (Participants) | 9
  Serotype 21 at Year 3:I | 0.0
  Serotype 22F at Year 3:I: number analyzed (Participants) | 9
  Serotype 22F at Year 3:I | 0.0
  Serotype 23A at Year 3:I: number analyzed (Participants) | 9
  Serotype 23A at Year 3:I | 0.0
  Serotype 38 at Year 3:I: number analyzed (Participants) | 9
  Serotype 38 at Year 3:I | 0.0
  Serotype 3 at Year 1:R: number analyzed (Participants) | 18
  Serotype 3 at Year 1:R | 0.0
  Serotype 12 at Year 1:R: number analyzed (Participants) | 18
  Serotype 12 at Year 1:R | 5.6
  Serotype 15A at Year 1:R: number analyzed (Participants) | 18
  Serotype 15A at Year 1:R | 0.0
  Serotype 15B at Year 1:R: number analyzed (Participants) | 18
  Serotype 15B at Year 1:R | 5.6
  Serotype 15F at Year 1:R: number analyzed (Participants) | 18
  Serotype 15F at Year 1:R | 0.0
  Serotype 19A at Year 1:R: number analyzed (Participants) | 18
  Serotype 19A at Year 1:R | 22.2
  Serotype 19F at Year 1:R: number analyzed (Participants) | 18
  Serotype 19F at Year 1:R | 5.6
  Serotype 21 at Year 1:R: number analyzed (Participants) | 18
  Serotype 21 at Year 1:R | 0.0
  Serotype 22F at Year 1:R: number analyzed (Participants) | 18
  Serotype 22F at Year 1:R | 5.6
  Serotype 23A at Year 1:R: number analyzed (Participants) | 18
  Serotype 23A at Year 1:R | 5.6
  Serotype 38 at Year 1:R: number analyzed (Participants) | 18
  Serotype 38 at Year 1:R | 5.6
  Serotype 3 at Year 2:R: number analyzed (Participants) | 7
  Serotype 3 at Year 2:R | 28.6
  Serotype 12 at Year 2:R: number analyzed (Participants) | 7
  Serotype 12 at Year 2:R | 0.0
  Serotype 15A at Year 2:R: number analyzed (Participants) | 7
  Serotype 15A at Year 2:R | 0.0
  Serotype 15B at Year 2:R: number analyzed (Participants) | 7
  Serotype 15B at Year 2:R | 0.0
  Serotype 15F at Year 2:R: number analyzed (Participants) | 7
  Serotype 15F at Year 2:R | 0.0
  Serotype 19A at Year 2:R: number analyzed (Participants) | 7
  Serotype 19A at Year 2:R | 42.9
  Serotype 19F at Year 2:R: number analyzed (Participants) | 7
  Serotype 19F at Year 2:R | 0.0
  Serotype 21 at Year 2:R: number analyzed (Participants) | 7
  Serotype 21 at Year 2:R | 0.0
  Serotype 22F at Year 2:R: number analyzed (Participants) | 7
  Serotype 22F at Year 2:R | 0.0
  Serotype 23A at Year 2:R: number analyzed (Participants) | 7
  Serotype 23A at Year 2:R | 0.0
  Serotype 38 at Year 2:R: number analyzed (Participants) | 7
  Serotype 38 at Year 2:R | 0.0
  Serotype 3 at Year 3:R: number analyzed (Participants) | 9
  Serotype 3 at Year 3:R | 11.1
  Serotype 12 at Year 3:R: number analyzed (Participants) | 9
  Serotype 12 at Year 3:R | 0.0
  Serotype 15A at Year 3:R: number analyzed (Participants) | 9
  Serotype 15A at Year 3:R | 0.0
  Serotype 15B at Year 3:R: number analyzed (Participants) | 9
  Serotype 15B at Year 3:R | 0.0
  Serotype 15F at Year 3:R: number analyzed (Participants) | 9
  Serotype 15F at Year 3:R | 0.0
  Serotype 19A at Year 3:R: number analyzed (Participants) | 9
  Serotype 19A at Year 3:R | 11.1
  Serotype 19F at Year 3:R: number analyzed (Participants) | 9
  Serotype 19F at Year 3:R | 0.0
  Serotype 21 at Year 3:R: number analyzed (Participants) | 9
  Serotype 21 at Year 3:R | 0.0
  Serotype 22F at Year 3:R: number analyzed (Participants) | 9
  Serotype 22F at Year 3:R | 0.0
  Serotype 23A at Year 3:R: number analyzed (Participants) | 9
  Serotype 23A at Year 3:R | 0.0
  Serotype 38 at Year 3:R: number analyzed (Participants) | 9
  Serotype 38 at Year 3:R | 0.0

19. Secondary Outcome: Percentage of Participants With Primary Clinical Diagnosis of Otitis Media
Description: Percentage of participants with primary diagnosis of otitis media was computed along with exact 2-sided 95% CI based on the observed proportion of participants for each of the 3 surveillance year. Results for baseline period were analyzed for participants who received routinely recommended vaccination of 13vPnC. The cases of otitis media reported during the baseline period were captured by the Texas Children's Hospital, which was the only site that collected this information during the baseline period. Percentage of participants was calculated by dividing number of participants with at least 1 MEF sample for the specified year by total number of participants with at least 1 MEF sample for the 3 year surveillance period.
Time Frame: Baseline Year 1, 2, 3; Surveillance Year 1, 2, 3
Population: MEF population included all participants who have at least 1 S pneumoniae isolate from MEF samples during baseline (2007-2009) and surveillance (2011-2013) period.N(number of participants analyzed) includes total number of participants in MEF population and n=number of participants for the specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MEF Population
Number analyzed (Participants) | 357
percentage of participants
  Baseline Year 1: 2007: number analyzed (Participants) | 75
  Baseline Year 1: 2007 | 24.0 [14.9 to 35.3]
  Baseline Year 2: 2008: number analyzed (Participants) | 75
  Baseline Year 2: 2008 | 45.3 [33.8 to 57.3]
  Baseline Year 3: 2009: number analyzed (Participants) | 75
  Baseline Year 3: 2009 | 30.7 [20.5 to 42.4]
  Surveillance Year 1: 2011 | 37.8 [32.8 to 43.1]
  Surveillance Year 2: 2012 | 31.1 [26.3 to 36.2]
  Surveillance Year 3: 2013 | 31.1 [26.3 to 36.2]

20. Secondary Outcome: Percentage of Participants With Primary Clinical Diagnosis of Mastoiditis
Description: Percentage of participants with primary diagnosis of mastoiditis was computed along with exact 2-sided 95% CI based on the observed proportion of participants for each of the 3 surveillance year. Percentage of participants was calculated by dividing number of participants with at least 1 mastoid sample for the specified year by total number of participants with at least 1 mastoid sample for the 3 year surveillance period.
Time Frame: Surveillance Year 1, 2, 3
Population: Mastoid population included all participants who have at least 1 S pneumoniae isolate from mastoid samples surveillance period. N(number of participants analyzed) includes total number of participants in mastoid population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mastoid Population
Number analyzed (Participants) | 34
percentage of participants
  Surveillance Year 1 | 52.9 [35.1 to 70.2]
  Surveillance Year 2 | 20.6 [8.7 to 37.9]
  Surveillance Year 3 | 26.5 [12.9 to 44.4]

ADVERSE EVENTS:
Description: Due to observational nature of study , individual adverse events (AEs) were not planned to be collected and reported.
Arm/Group | MEF Population | Mastoid Population
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.